

# Statistical Analysis Plan

Study Title: A Phase 2, Open-Label, Multi-Center Trial of Mavorixafor

in Patients with WHIM Syndrome

Phase: 2

**Protocol Number:** X4P-001-MKKA

**Sponsor:** X4 Pharmaceuticals, Inc.

61 North Beacon Street, 4<sup>th</sup> Floor

Boston, MA 02134

**Protocol Number:** X4P-001-MKKA (21 December 2020, Version 5.0)

**Document Version:** Version 3.0, 16<sup>th</sup> February 2022

# **Approvals**



# **Document History**

| Version | Date | Author | Description |
|---|---|---|---|
| 1.0 | 01Jun 2016 | | Initial Draft: Submitted to FDA (Initial IND 129092, 10 June 2016 |
| 2.0 | 21 Feb 2018 | | Updated based on protocol amendments, increase total daily dose to 400mg, specify exploratory analyses and other various administrative updates |
| 3.0 | 18 Sep 2020 | | Updated based on protocol amendment 4.6 (added objectives for the extension phase, added an updated schedule of events), Infection rate calculation has been added in section 6.1.2 |
| | | | • Added Figure 1 and Box plot analysis in section 6.1.4 |
| | | | • Time above threshold analysis added as section 6.1.5 |
| | | | • Re-enrollment due to COVID-19 added as section 6.1.6 |
| | | | Local lab analysis and Cerba Research lab corrections added in section 9.2 |
| | | | • Added derivations for infection rate & infection score for 6 month time intervals in section 6.1.2 |
| 3.0 | 22 Feb 2021 | | Add ITT population |
| | | | Add handling of partial dates for infection events |
| | | | • Updated based on protocol amendment 5.0 |

| 3.0 | 29 July 2021 | <ul> <li>Updated infection rate calculations and corresponding TLFs</li> <li>Added in 6 month time interval for infection rate</li> </ul> |
|---|---|---|
| 3.0 | 16 February<br>2022 | <ul> <li>Updated TLF shells</li> <li>Updated section 2.2.3 to note that local lab was used to analyze whole blood samples due to COVID-19</li> <li>Added in DRC meeting timelines for extension phase to sections 3 and 4.3.</li> <li>Updated laboratory baseline derivation</li> <li>Updated medical history text to reference 12 months prior to study start instead of 6 months</li> <li>Updated protocol deviations classification to be important/non-important instead of major/minor</li> <li>Updated per protocol population definition to reference important protocol violations instead of major protocol violations.</li> </ul> |

### **Table of Contents** Approvals 1 List of Figures 10 Abbreviations 10 1. Overview 12 2.1. 2.2. 3.1. 3.2. 3.3. Treatments Administered 16 3.4. 3.5. 3.6. 4. Statistical Analysis and Reporting 23 4.1. 4.2. Statistical Hypothesis 23 4.3. 5. 6. 6.1. 6.1.2. Derived Variables 25 7. 7.1.

| | 7.2. | Protocol Violations and Deviations | 29 |
|---|---|---|---|
| | 7.3. | Demographics and Other Baseline Characteristics | 29 |
| | 7.4. | Medical History | 29 |
| 8. | Ef | ficacy Analysis | 29 |
| | 8.1. | Primary Efficacy Analysis | 29 |
| | 8.2. | Exploratory Efficacy Analysis | |
| | 8.3. | Subgroup Analysis | |
| 9. | Sa | fety and Tolerability Analysis | |
| | 9.1. | Adverse Events | |
| | 9.1.1. | Adverse Events Leading to Withdrawal | 31 |
| | 9.1.2. | _ | |
| | 9.1.3. | Treatment Limiting Toxicities | 31 |
| | 9.2. | Clinical Laboratory Evaluations | |
| | 9.3. | Vital Signs | |
| | 9.4. | Electrocardiograms | 34 |
| | 9.5. | Concomitant Medication. | |
| | 9.6. | Exposure and Compliance | 34 |
| 10 | Cl | nanges from Planned Analysis | |
| 11. | Ot | ther Planned Analysis | 35 |
| | 11.1. | Pharmacokinetic and Pharmacodynamic (PK/PD) Analysis | 35 |
| | 11.2. | Biomarker Analysis | 35 |
| 12 | Re | eferences | 36 |
| 13. | Ta | bles, Listings, and Figures | 37 |
| | 13.1. | Planned Table Descriptions | |
| | 13.2. | Demographic Data | 37 |
| | 13.3. | Efficacy Data | 37 |
| | 13.4. | Safety Data | 38 |
| | 13.5. | Pharmacokinetic Data | 39 |
| | 13.6. | Planned Listing Descriptions | 39 |
| | 13.7. | Planned Figure Descriptions | 40 |
| 14 | Ta | bles, Listings, and Figure Shells | 42 |
| | 14.1. | Standard Layout for all Tables, Listings, and Figures | 42 |
| | 14.2. | Planned Table Shells | 42 |
| | Table | 14.1.1 Subject Disposition Informed Consent Signed | 43 |
| | Table | 14.1.2 Summary of Protocol Deviations Safety Population | 44 |
| | Table | 14.1.3 Demographics and Baseline Characteristics Safety Population | 46 |
| | Table | 14.1.4 Summary of Study Drug Exposure Safety Population | 48 |
| | Table | 14.1.5 Summary of Medical History Safety Population | 49 |

| Table 14.2.1.1 Summary of AUCs and Mean of AUCs for ANC by Dose Level - $AUC_{ANC} \ge 600/\mu L$ Threshold Safety Population | 50 |
|---|---|
| Table 14.2.1.1.1 Summary of AUCs and Mean of AUCs for ANC by Dose Level - | 50 |
| AUC $_{\rm ANC} \ge 500/\mu L$ Threshold Safety Population | 52 |
| Table 14.2.1.2 Summary of AUCs and Mean of AUCs for ALC by Dose Level Safety | 52 |
| Population | 53 |
| Table 14.2.2.3 Summary of Highest Grade Infections Safety Population | |
| Table 14.2.2.4 Summary of Infection Scores Safety Population | |
| Table 14.2.3.1 Summary of Non-Genital Warts Safety Population | |
| Table 14.2.3.2 Summary of Non-Genital Warts by location Safety Population | |
| Table 14.2.4.1 Summary of Genital Warts Safety Population | |
| Table 14.2.5 Summary of Antibody Levels following Revaccination Safety Population | |
| Table 14.2.6 Summary of Rescue Medications Safety Population | |
| Table 14.2.7 Summary of Hospitalizations Safety Population | |
| Table 14.2.8 Summary of Ig and Specified Antibodies Safety Population | |
| Table 14.2.9 Time above Threshold (Hours) for ANC by Dose Level Safety | |
| Population | 70 |
| Table 14.2.9.1 Time above Threshold (Hours) for ANC by Dose Level – Sensitivity | |
| Analysis Safety Population | 70 |
| Table 14.2.10 Time above Threshold (Hours) for ALC by Dose Level Safety | 70 |
| Population | /0 |
| Table 14.2.10.1 Time above Threshold (Hours) for ALC by Dose Level – Sensitivity Analysis Safety Population | 71 |
| Table 14.2.11 Time above Threshold (Hours) for AMC by Dose Level Safety | / 1 |
| Population | 71 |
| Table 14.3.1.1 Overall Summary of Treatment-Emergent Adverse Events Safety | |
| Population | 72 |
| Table 14.3.1.2 Summary of Treatment-Emergent Adverse Events by System Organ | |
| Class and Preferred Term Safety Population | 74 |
| Table 14.3.1.3 Summary of Treatment-Emergent Adverse Events Related to Study | |
| Treatment by System Organ Class and Preferred Term Safety Population | 76 |
| Table 14.3.2.1 Summary of Serious Adverse Events by System Organ Class and Preferred Term Safety Population | 78 |
| Table 14.3.2.2 Summary of Serious Adverse Events Related to Study Treatment by | |
| System Organ Class and Preferred Term Safety Population | 80 |
| Table 14.3.2.3 Summary of Treatment-Limiting Toxicities by System Organ Class and Preferred Term Safety Population | 82 |
| Table 14.3.2.4 Summary of Grade 3 or Higher Treatment-Emergent Adverse Events by | |
| System Organ Class and Preferred Term Safety Population | 83 |
| Table 14.3.2.5 Rate of Treatment Emergent Adverse Events by System Organ Class | |
| and Preferred Term Safety Population | 84 |

| Table 14.3.2.6.1 Summary of Yearly Infection Rate for Subjects on 300mg and 400mg Dose Levels by 6 Month Intervals Safety Population |
|---|
| Table 14.3.2.6.2 Summary of Yearly Infection Score for Subjects on 300mg and |
| 400mg Dose Levels by 6 Month Intervals Safety Population |
| Table 14.3.2.7.1 Summary of Yearly Infection Rate by Dose Level – Method 1 Safety Population |
| Table 14.3.2.7.2 Summary of Yearly Infection Rate by Dose Level – Method 2 Safety Population |
| Table 14.3.3.1 Listing of Serious Adverse Events Safety Population |
| Table 14.3.3.2 Listing of Treatment Emergent Adverse Events Leading to Discontinuation Safety Population |
| Table 14.3.4.1 Listing of Out of Reference Range Laboratory Values Safety Population 91 |
| Table 14.3.5.1.1 Summary of Actual and Change from Baseline in Hematology Results Safety Population 92 |
| Table 14.3.5.1.2 Shift from Baseline in Hematology Results Safety Population94 |
| Table 14.3.5.2.1 Summary of Actual and Change from Baseline in Serum Chemistry Results Safety Population |
| Table 14.3.5.2.2 Shift from Baseline in Serum Chemistry Results Safety Population 95 |
| Table 14.3.5.3.1 Summary of Actual and Change from Baseline in Coagulation Results Safety Population |
| Table 14.3.5.3.2 Shift from Baseline in Coagulation Results Safety Population |
| Table 14.3.5.4.1 Summary of Actual and Change from Baseline in Cytometry Results Safety Population 95 |
| Table 14.3.6.1.1 Summary of Actual and Change from Baseline in Vital Signs Safety Population |
| Table 14.3.6.2.1 Summary of Actual and Change from Baseline of 12-Lead Electrocardiogram (ECG) Parameters Safety Population |
| Table 14.3.6.3.1 Summary of Ophthalmologic Examination Results (Local Reader) Safety Populaion 98 |
| Table 14.3.6.3.2 Summary of Ophthalmologic Examination Results (Central Retinal Findings) Safety Populaion |
| Table 14.3.6.4 Summary of Concomitant Medications Safety Population |
| Table 14.3.6.5.1 Summary of Use of Antibiotics, G-CSF, Immunoglobulins, and Imiquamod – Concomitant Medications Safety Population |
| Table 14.3.6.5.2 Summary of Use of Antibiotics, G-CSF, Immunoglobulins, and Imiquamod – Prior Medications Safety Population |
| Table 14.3.6.6 Summary of Actual and Change from Baseline in SF-36 QOL Scores Safety Population |
| Table 14.3.6.6 Summary of Actual and Change from Baseline in HPV Impact Profile (HIP) Questionnaire - Domain Scores Safety Population |

| Table 14.4.1 Summary of Plasma X4P-001 Concentrations by Dose Level Safety Population | . 103 |
|---|---|
| Table 14.4.2 Summary of Plasma X4P-001 Pharmacokinetic Parameters by Dose Level Safety Population | |
| 14.3. Planned Figure Shells | |
| Figure 14.4.1.1 WBC over Time by Patient Safety Population | |
| Figure 14.4.1.2a ANC over Time by Patient Safety Population | |
| Figure 14.4.1.2b ANC over Time by Dose Level Safety Population | |
| Figure 14.4.1.3a ALC over Time by Patient Safety Population | |
| Figure 14.4.1.3b ALC over Time by Dose Level Safety Population | . 106 |
| Figure 14.4.1.4a Monocytes over Time by Patient Safety Population | . 106 |
| Figure 14.4.1.4b Monocytes over Time by Dose Level Safety Population | . 108 |
| Figure 14.4.1.5 Mean (+/– SE) Plasma Concentration - Time Profile of X4P-001 by Dose Level Safety Population | . 109 |
| Figure 14.4.1.6 Mean Dose Response of ANC - Time Profile Safety Population | . 110 |
| Figure 14.4.1.7 Mean Dose Response of ALC - Time Profile Safety Population | . 111 |
| Figure 14.4.1.8 Mean Dose Response of Monocytes - Time Profile Safety Population | . 111 |
| Figure 14.4.1.9 Box plots of WBC change from baseline ratio at 300mg and 400mg by Dose Level Safety Population | . 112 |
| Figure 14.4.1.10 Box plots of AUC for ANC by Dose Level Safety Population | . 113 |
| Figure 14.4.1.11 Scatter Plot of Time above Threshold values for ANC versus AUC for ANC Safety Population | . 114 |
| Figure 14.4.1.12 Scatter Plot of Time above Threshold values for ALC versus AUC for ALC Safety Population | . 114 |
| Figure 14.4.1.13.1 Plot of Yearly Infection Rate by Dose Level Safety Population | . 115 |
| Figure 14.4.1.13.2 Plot of Yearly Infection Score by Dose Level Safety Population | . 116 |
| Figure 14.4.1.14.1 Plot of Yearly Infection Rate for Subjects on 300mg and 400 mg Dose Levels by 6 Month Intervals Safety Population | . 117 |
| Figure 14.4.1.14.2 Plot of Yearly Infection Score for Subjects on 300 mg and 400 mg Dose Levels by 6 Month Intervals Safety Population | . 118 |
| Figure 14.4.2.1 Scatter Plot of Plasma Drug Level and ANC Safety Population | . 119 |
| Figure 14.4.2.2 Scatter Plot of Plasma Drug Level and ALC Safety Population | . 119 |
| Figure 14.4.3.1 Mean Plasma Concentrations of X4P-001 vs Nominal Time (Dense Sampling Visits) by Dose Level - Linear Scale Safety Population | . 119 |
| Figure 14.4.3.2 Mean Plasma Concentrations of X4P-001 vs Nominal Time (Dense Sampling Visits) by Dose Level - Semi-Logarithmic Scale Safety Population | . 119 |
| Figure 14.4.4.1 Subject Plasma Concentrations of X4P-001 vs Nominal Time (Dense Sampling Visits) by Dose Level - Linear Scale Safety Population | . 120 |
| Figure 14.4.4.2 Subject Plasma Concentrations of X4P-001 vs Nominal Time (Dense Sampling Visits) by Dose Level - Semi-Logarithmic Scale Safety Population | . 120 |

| 14.4. Planned Listing Shells | 121 |
|---|---|
| Listing 16.2.1 Subject Disposition All Enrolled Patients | 122 |
| Listing 16.2.2.1 Eligibility Criteria Not Met All Enrolled Patients | 123 |
| Listing 16.2.2.2 Protocol Deviations Safety Population | 124 |
| Listing 16.2.3 Analysis Populations All Enrolled Patients | 125 |
| Listing 16.2.4.1 Demographics and Baseline Characteristics Safety Population | 126 |
| Listing 16.2.4.2 Medical History Safety Population | 127 |
| Listing 16.2.4.3.1 History of WHIM Syndrome - Hospitalizations Safety Population | 128 |
| Listing 16.2.4.3.2 History of WHIM Syndrome - Infections Managed as Out-Patient Safety Population | 129 |
| Listing 16.2.4.3.3 History of WHIM Syndrome - Prior Treatments for WHIM syndrome Safety Population | 130 |
| Listing 16.2.4.3.4 WHIM Syndrome Genotyping Safety Population | 131 |
| Listing 16.2.4.4.1 Study Drug Administration Safety Population | 132 |
| Listing 16.2.4.4.2 Study Drug Exposure Safety Population | 133 |
| Listing 16.2.4.5 Assessment of Warts Safety Population | 134 |
| Listing 16.2.4.6 Revaccination Safety Population | 135 |
| Listing 16.2.4.7 Bone Marrow Aspirate Safety Population | 136 |
| Listing 16.2.5.1 Pharmacokinetic Blood Collection and Concentrations Safety Population | 137 |
| Listing 16.2.5.2 Calculated Pharmacokinetic Parameters Safety Population | 138 |
| Listing 16.2.6.1 ANC/ALC Sample Collection Safety Population | 139 |
| Listing 16.2.6.2.1 Threshold Adjusted AUC values for ANC Safety Population | 140 |
| Listing 16.2.6.2.2 Threshold Adjusted AUC values for ALC Safety Population | 141 |
| Listing 16.2.6.2.3 Time Above Threshold by Dose Level - Assessment of ANC/ALC/AMC Safety Population | 142 |
| Listing 16.2.6.2.4 Time Above Threshold - Assessment of ANC/ALC/AMC with Time | |
| Crossed Safety Population | 144 |
| Listing 16.2.7.1 Treatment Emergent Adverse Events Safety Population | 145 |
| Listing 16.2.7.2 Adverse Events that occur during Screening and ended before Exposure to study Drug Safety Population | 146 |
| Listing 16.2.7.3 Infections Reported as Adverse Events Safety Population | 147 |
| Listing 16.2.7.4 Deaths All Enrolled Patients. | 149 |
| Listing 16.2.7.5 Treatment Limiting Toxicities Safety Population | 150 |
| Listing 16.2.7.6 Infections in Subjects Treated on 300mg or 400 mg Dose by Time Period Safety Population | 151 |
| Listing 16.2.7.7 Infections by Dose Level Safety Population | |
| Listing 16.2.7.8 Infections by Subject Safety Population | 153 |
| Listing 16.2.8.1 Clinical Laboratory Data: Serum Chemistry Safety Population | |
| Listing 16.2.8.2 Clinical Laboratory Data: Hematology Safety Population | 156 |

| Listing 16.2.8.3 S | erology and Other Laboratory Test Results Safety Population | 156 |
|---|---|---|
| Listing 16.2.8.4 S | erum Ig and Specific Antibody Laboratory Test Results Safety | |
| | 1 | 157 |
| Listing 16.2.8.5 P | regnancy Test Safety Population | 158 |
| | oagulation Laboratory Test Results Safety Population | |
| | rinalysis Laboratory Test Results Safety Population | |
| | ytometryTest Results Safety Population | |
| | rior or Concomitant Medications Safety Population | |
| <del>-</del> | Tital Signs Measurements Safety Population | |
| | 2-Lead Electrocardiograms Safety Population | |
| <del>-</del> | hysical Examinations Safety Population | |
| | ophthalmologic Examination (Site Assessment) Safety Population | |
| <del>-</del> | Ophthalmologic Examination (Central Readings) Safety Population | |
| | escue Medications Safety Population | |
| <del>-</del> | F-36 QOL Safety Population | |
| Listing 16.2.9.9.1 | HPV Impact Profile (HIP) Questionnaire Safety Population | 171 |
| Listing 16.2.9.9.2 | HPV Impact Profile (HIP) Questionnaire - Domain Scores Safety | |
| Population | 1 | 172 |
| List of Tables | | |
| | Events – Initial Treatment Period | |
| | Events – Extension Phase | |
| Table 3: Overview of | Conversion Factors | 33 |
| List of Figures | | |
| List of Figures | | |
| Figure 1: Calculation | of 24-hr AUC for a Hypothetical Set of ALC Data | 27 |
| Abbreviations | | |
| ABBREVIATION | DEFINITION OR DESCRIPTION | |
| AE | Adverse event | |
| ALC | Absolute lymphocyte count | |
| AMC | Absolute monocyte count | |
| ANC | Absolute neutrophil count | |
| ATC | Anatomical Therapeutic Chemical classification | |
| AUC | Area under the plasma concentration curve | |
| AUC <sub>ALC</sub> | Area under the plasma concentration curve for absolute lymphocyt count | e |
| AUC <sub>ANC</sub> | Area under the plasma concentration curve for absolute neutrophil | count |

Below the limit of quantification

Body mass index

BLQ

BMI

| BOCF | Baseline-observation-carried-forward |
|---|---|
| C <sub>max</sub> | Maximum concentration |
| CRF | Case report form |
| CSR | Clinical study report |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CXCR4 | Chemokine receptor type 4 |
| DRC | Data review committee |
| ECG | Electrocardiogram |
| eCRF | Electronic Case report form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FACS | Fluorescence activated cell sorting |
| G-CSF | Granulocyte-colony stimulating factor |
| HIP | HPV Impact Profile |
| ICH | International Council for Harmonisation |
| iCSR | Interim Clinical Study Report |
| Ig | Immunoglobulin |
| LOCF | Last-observation-carried-forward |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NCI | National Cancer Institute |
| PBMC | Peripheral blood mononuclear cells |
| PD | Pharmacodynamic |
| PK | Pharmacokinetic |
| QD | Once Daily |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SOC | System organ class |
| TEAE | Treatment-emergent adverse event |
| T <sub>max</sub> | Time to maximum concentration |
| WBC | White blood cell |
| WHIM | Warts, Hypogammaglobulinemia, Infections, and Myelokathexis |
| WHO-DD | World Health Organization Drug Dictionary |

#### 1. Overview

This Statistical Analysis Plan (SAP) describes the planned analyses and data presentation for the Phase 2 component of the Phase 2 Study X4P-001-MKKA, titled "A Phase 2, Open-Label, Multi-Center Trial of Mavorixafor in Patients with WHIM Syndrome".

The development of this SAP is based on Protocol Version 5.0, dated 21<sup>st</sup> December 2020. The structure and content of this SAP provides sufficient detail to meet the requirements identified by the Food and Drug Administration (FDA), European Medicines Agency (EMA), and International Council for Harmonisation (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use: Guidance on Statistical Principles in Clinical Trials. All work planned and reported in this SAP will follow internationally accepted guidelines, published by the American Statistical Association and the Royal Statistical Society, for statistical practice.

The analyses described in this SAP will be used to support the clinical study reports (CSRs), regulatory submissions, or future manuscripts. Post-hoc exploratory analyses not identified in this SAP may be performed to further examine study data. Any post-hoc analyses will be clearly identified as such in the CSR.

# 2. Study Objectives and Endpoints

# 2.1. Study Objectives

#### 2.1.1. Primary Objectives

The objectives of the initial treatment period are:

- To evaluate safety and tolerability of mavorixafor (X4P-001) in patients with WHIM syndrome.
- To assess the dose required to achieve a consistent increase in circulating neutrophils and lymphocytes in patients with WHIM syndrome.

The objectives of the extension phase are:

- To evaluate the safety of long-term treatment with mavorixafor.
- To evaluate the efficacy of long-term mavorixafor treatment on infection rate, cutaneous warts, vaccine titers, and neutrophil and lymphocyte counts.

#### 2.2. Study Endpoints

# 2.2.1. Primary Endpoints

The primary endpoints of the study are:

- To determine the safety and tolerability of X4P-001; and
- To evaluate the mean area under the curve (AUC) of the absolute neutrophil count (ANC) AUC<sub>ANC</sub> and/or AUC<sub>ALC</sub> (absolute lymphocyte count) collected over 24-hour period

above clinically meaningful thresholds during the initial treatment phase of the study (first 6 month).

# 2.2.1.1. Safety and Tolerability

Safety and tolerability will be evaluated by the following:

- Treatment-emergent adverse events (TEAEs)
- Adverse events (AEs) assessed as related, possibly, or probably related to treatment by grade (all grades and grade  $\geq 3$ )
- Serious adverse events (SAEs)
- Deaths
- Discontinuations due to AEs

С

- Vital signs
- Clinical laboratory test results
  - o Hematology
  - o Serum chemistry
  - Pregnancy test (as applicable)
- Physical examination findings
- 12-lead ECG results
- Ophthalmology (local and central)

#### 2.2.1.2. 24-Hour AUCANC and/or AUCALC

The primary efficacy endpoint is the mean 24-hour AUC<sub>ANC</sub> and/or AUC<sub>ALC</sub> above the clinically meaningful thresholds. The clinically meaningful threshold for ANC is  $\geq 600/\mu L$  and for ALC is  $\geq 1000/\mu L$ .

# 2.2.2. Exploratory Endpoints

- Time above threshold values for ANC, AMC, and ALC, as applicable, will be calculated using the ANC and ALC assessments collected during the 24-hour collection times and analyzed as percentage of time (from initial to final value obtained during each of these visits) above the clinically meaningful thresholds of 500/µL and 1000/µL Time (hours)>ANC Threshold<sub>500</sub>, Time (hours)>ALC Threshold<sub>1000</sub>), respectively. These parameters will be compared between dose levels to determine if there is a dosedependent change in the respective Time (hours)>Time Above Thresholds.
- Frequency and severity of infections (severity assessed as Grade 1 to 5 (protocol only mention Grade 1 to 4) using National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 or higher).
- **Number of Cutaneous warts** applicable only to patients with cutaneous warts at baseline, and comparing number at baseline to number at end of Treatment Period.
- Severity of genital warts applicable only to patients with genital warts, and comparing number of lesions, size of largest lesion, and patient-reported morbidity at baseline to end of Treatment Period.

- Antibody levels following revaccination applicable only to patients who were (a) previously administered approved vaccines, (b) found at baseline to have predefined subprotective levels of antibody, and (c) agree to repeat administration of the vaccine after 12 weeks of treatment.
- Frequency of events requiring rescue therapy (granulocyte-colony stimulating factor [G-CSF] and/or intravenous immunoglobulins [Ig]).
- Rate of hospitalization events will be evaluated based on the information collected in the 12 months prior to start of participation in Study X4P-001-MKKA through end of Phase 2 Treatment Period and end of the study or data cutoff for the interim and final Clinical Study Report (CSR).
- Circulating white blood cells (WBCs) Absolute and fold change from baseline in total WBC counts, and in absolute numbers of lymphocytes, neutrophils, monocytes, and lymphocyte subpopulations cells.
  - o Correlation of ANC and ALC levels with plasma drug levels

# • Ig and specific antibodies

- Changes from baseline in levels of total IgG, IgG subclasses, IgA, IgD, IgE and IgM.
- Bone marrow aspirates Optional (analyzed centrally by a blinded reviewer) Change from baseline in cellularity. Change from baseline in frequency of apoptotic cells.
- **Quality of Life** as assessed by SF-36 short form survey, Life Quality Index (LQI) and Human papillomavirus (HPV) Impact Profile (HIP).

#### 2.2.3. Pharmacokinetic and Pharmacodynamic (PK/PD) Endpoints

For all patients receiving study drug, dense PK samples will be obtained during the 24-hour periods in-residence at the following time points:

• Time 0 (-15 min), 30, 60, 90 min (each  $\pm$ 5 min) and 2, 3, 4, 8, 12, 16, 24 hr (each  $\pm$ 15 min).

Additional time point 0 samples (trough) will be collected at Day 1 and Weeks 9, 17 and 25. Blood samples for plasma levels of X4P-001 will be analyzed for X4P-001 concentration using reversed-phase high performance liquid chromatography with tandem mass spectrometry detection. The PK parameters include AUC, maximum concentration ( $C_{max}$ ) and time to maximum concentration ( $T_{max}$ ). X4P-001 concentration and PK parameters will be analyzed by treated patients and dosage regimen over the preceding week.

The in-residence stay will be rescheduled in the event of recent infection, administration of antibiotics, or of rescue therapy with G-CSF or intravenous Ig. Whole blood samples could be analyzed in local laboratories instead of a central laboratory due to COVID-19 restrictions, ANC and ALC were determined by standard methods. ANC and/or ALC will be calculated over time by patient and by dose. A full PK analysis plan will be developed separately from this document.

# 2.2.4. Biomarker Endpoints

Biomarker samples will be collected concurrent with time point 0 PK samples. Assessments may include samples analyzed by flow cytometry for subpopulations of peripheral blood mononuclear cells (PBMC). Candidate subsets are naïve T cells, memory T cells, B cells, transitional B cells, NK cells, and monocytes.

### 3. Overall Study Design and Plan

Patients will be scheduled for several 24-hour visits to permit collection of serial samples over 24 hours for determination of ANC/ALC and plasma drug levels. This will be calculated as the mean AUC over the 24-week Treatment Phase and Extension Phase, as data are available.

During the initial Treatment Phase, all available safety data will be reviewed approximately every 12 weeks by a Phase 2 Data Review Committee (DRC). The DRC will include participating Investigator(s), an independent physician with relevant experience in clinical research and/or immune deficiency diseases, the Medical Monitor, and a representative of the Sponsor. During the Extension Phase, the DRC will review data approximately every 6 months.

During the scheduled treatment period, patients will attend monthly office visits and will be monitored daily using an automated telephone- or web-based reporting system for temperature, activities of daily living, antibiotic usage, and unscheduled healthcare visits. Patients may receive standard of care antibiotics in the event of infection, but may not receive routine G-CSF or immunoglobulin therapy as a prophylactic treatment. In the event of an episode consistent with acute, severe bacterial infection, the investigator may add rescue therapy consisting of a course of G-CSF and/or immunoglobulin therapy if applicable (see Section 7.4.4.2 of the Protocol).

Participation in the initial Treatment Phase of the study is considered complete after 24 weeks of treatment with X4P-001 or until development of a TLT. For the definition of a treatment limiting toxicity, please see Section 5.7 of the Protocol. Thereafter, patients may continue participation in an open-label Phase 2 Extension Phase of the protocol where dose escalation and/or additional in-residence stays may be permitted.

#### **Phase 2 Extension Phase**

With the agreement of the Investigator, patients may enter the Extension Phase of the study and receive study drug until it becomes available via an alternative mechanism (e.g., drug is commercially available, an expanded access program, etc.). At the discretion of the Sponsor and with agreement from the investigator, patients may have their dose escalated and have additional in-residence or dense-sampling visits conducted during the Extension Phase.

Patients from the Phase 2 study receiving less than the selected Phase 3 dose may choose to receive the recommended Phase 3 dose once determined. The patient's participation in the Extension Phase will be complete when study treatment is discontinued, and all Extension Phase visits are complete. The procedures during the extension phase are described in Section 7.3.1 of the Protocol in detail.

# 3.1. Sample Size and Power

Given the rarity of the disease under study as well as the known PK and PD profile of mavorixafor, albeit in populations other than WHIM syndrome, a traditional 3+3 dose escalation design was not selected. Alternatively, a small number of adult subjects (N= up to 15) will be treated with mavorixafor on an open-label basis. A sample size of up to 15 patients is considered adequate for the study objectives of assessing safety, tolerability, and preliminary efficacy for planning Phase 3.

# 3.2. Study Population

The target patient population is adult patients with a confirmed diagnosis of WHIM syndrome to be eligible for the study.

### 3.3. Treatments Administered

The investigational drug is X4P-001, which is administered orally once daily not to exceed 400 mg daily dose. Patients either received a 25 mg capsule strength or a 100 mg capsule strength. Patients who received lower doses (50 mg to 200 mg QD) received 25 mg capsules until it was determined that higher doses would be necessary (i.e., total daily dose not to exceed 400 mg). Therefore, after September 2017 patients either switched to or started initial dosing at a larger capsule strength (100 mg) when it was determined by the Investigator and Sponsor that higher daily doses (300 mg and 400 mg) would be appropriate.

# 3.4. Method of Assigning Patients to Treatment Groups

All patients will be treated with X4P-001 open-label. The decision for dose-escalation, if necessary, will be based on ANC and ALC analyzed as AUCs relative to pre-specified clinically meaning thresholds of  $600/\mu L$  and  $1000/\mu L$ , respectively. The 24-hour AUC will be calculated using the trapezoidal method with area above threshold being positive, and area below threshold, negative (see Section 10.4.2 of the protocol). Patients with AUC<sub>ANC</sub> <2000 cell•hr/ $\mu L$  or AUC<sub>ALC</sub> <5000 cell•hr/ $\mu L$  at the Week 5 or Week 13 evaluations will have mavorixafor daily dose increased to a maximum daily dose of 400 mg as indicated below:

- Planned doses: 100 mg QD, 200 mg QD, 300 mg QD, 400 mg QD.
- Based on the emerging safety, PK, and pharmacodynamic (PD) data, the planned dose may be omitted, an intermediate dose may be used to substitute the planned dose, or a BID dosing regimen may be explored. However, the maximum daily dose will be ≤400 mg.

Subsequent dose-escalations may be conducted in both treatment periods after prior approval from the Data Monitoring Committee, based on  $AUC_{ANC/ALC}$  values, safety data, and review of clinical efficacy, up to a maximum dose of 400 mg daily. Dose-escalation may occur to determine the Phase 3 dose that will provide the most consistent increase in circulating neutrophils and lymphocytes in the most number of patients. Patients who experience  $a \ge Grade 3$  treatment-related SAE will not be escalated.

#### 3.5. Blinding and Unblinding

Not applicable.

# 3.6. Schedule of Events

For a detailed schedule of events, please see Table 1.

**Table 1: Schedule of Events – Initial Treatment Period** 

| Table 1: Schedule of | L vents – | iniviai 1 | - catillell | . I CIIUU | | Study Per | riod / Visit | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | T <sub>1</sub> | nitial Treati | | 1 | | | | EOS <sup>5 6</sup> |
| Procedure | Screen-<br>ing <sup>2</sup> | Day 1 | Week 2 <sup>3</sup> (± 3D) | Week 3 <sup>3</sup> (± 3D) | Week 4 <sup>3</sup> (± 3D) | Week 5 <sup>4</sup><br>(-7D/<br>+14D) | Week 9 <sup>3</sup> (± 7D) | Week 13 <sup>4</sup> (± 14D) | Week 17 <sup>3</sup> (± 7D) | Week 21 <sup>4</sup> (± 14D) | Week 25<br>(EOT)<br>(± 7D) | |
| Informed consent | X | | | | | | | | | | X <sup>6</sup> | $X^6$ |
| General medical history | X | | | | | | | | | | | |
| History of WHIM syndrome | X | | | | | | | | | | | |
| Inclusion / exclusion criteria | X | | | | | | | | | | | |
| Genotyping for eligibility | X | | | | | | | | | | | |
| ANC and ALC for eligibility | X | | | | | | | | | | | |
| Serology | X | | | | | | | | | | | |
| Height | X | X | | | | X | | X | | | X | X |
| Body weight | X | X | | | | X | | X | | | X | X |
| Physical examination | X | X | | | | X | | X | | | X | X |
| Vital signs <sup>7</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| Safety laboratory tests <sup>8</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| 12-lead ECG <sup>9</sup> | X | X | | | | X | | X | | X | | |
| Ophthalmologic examination <sup>10</sup> | X | | | | | | | X | | | X | |
| Pregnancy test <sup>11</sup> | X | X <sup>12</sup> | | | | X | X | X | X | X | X | X |
| Serial WBC, AMC, ANC and ALC sampling (for time above threshold and AUC) <sup>13</sup> | | | | | | X <sup>14</sup> | | X | | X | | |
| Assessment of warts <sup>15</sup> | X | X | | | | X | | $X^{16}$ | | X | | |

| | Study Period / Visit | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Initial Treatment Period <sup>1</sup> | | | | | | | | | | |
| Procedure | Screen-ing <sup>2</sup> | Day 1 | Week 2 <sup>3</sup> (± 3D) | Week 3 <sup>3</sup> (± 3D) | Week 4 <sup>3</sup> (± 3D) | Week 5 <sup>4</sup><br>(-7D/<br>+14D) | Week 9 <sup>3</sup> (± 7D) | Week 13 <sup>4</sup> (± 14D) | Week 17 <sup>3</sup> (± 7D) | Week 21 <sup>4</sup> (± 14D) | Week 25<br>(EOT)<br>(± 7D) | EOS <sup>5 6</sup> |
| Serum Ig and specific antibodies | | X | | | | | X | | X | | X | |
| Revaccination | | | | | | | | X | | | | |
| Quality of life questionnaires | | X | | X | | X | X | X | X | X | Х | |
| PK and Biomarker Time 0 sample <sup>17</sup> | | X | | | | | X | | X | | X | |
| PK dense sampling <sup>17</sup> | | | | | | X | | X | | X | | |
| Bone marrow aspirate <i>(optional)</i> <sup>18</sup> | X | | | | | | | | | | X | |
| Study drug administration | | | | | | X (D | aily) | | | | | |
| Diary completion <sup>19</sup> | | X (Daily) | | | | | | | | | | |
| Concomitant medication monitoring | | Continuous from Screening to EOS | | | | | | | | | | |
| Adverse event monitoring | | | | | Continuo | us from Info | rmed Conse | nt to EOS | | | | |

Abbreviations: ALC=Absolute lymphocyte count; AMC=Absolute monocyte count; ANC=Absolute neutrophil count; AUC=Area under the curve; ECG=electrocardiogram; EOS=End-of-Study; EOT=End-of-Treatment; HR=heart rate; Ig=immunoglobulin; PK=pharmacokinetics; WBC=white blood cell count; Note: Home-health visits are authorized if there are extenuating circumstances that would impede patients from coming to the study site for a scheduled visit. Requests for home health visits will be reviewed and approved by X4 on a case-by-case basis. Home health visits will be an option applicable for all study visits, including screening and baseline.

<sup>&</sup>lt;sup>1</sup> The schedule is presented relative to Study Week and Time of Dosing. The calendar day of the first administration of study drug is designated Day 1. All weeks are relative to Week 1, defined as Day 1 through Day 7, inclusive. Pre-and post-dose intervals are relative to the time of oral administration, designated 0 hr.

<sup>2</sup> Screening Visit and Day 1 may be done during the same visit.

<sup>&</sup>lt;sup>3</sup> Depending upon patient situation the Week 2, 3, 4, 9 and 17 vital signs and blood draws could be done at either the study site or by a visiting research nurse in the patient's home.

<sup>&</sup>lt;sup>4</sup> In-residence visits are conducted at Week 5 + 14 days and Weeks 13 and 21 ±14 days. If a patient cannot return to the study site for an in-residence visit, a dense-sampling visit may be conducted by visiting research nurse or by the patient's primary care physician; however, in-residence visits at the study site are preferred. If a patient has their dose escalated during the Extension Phase, additional in-residence or dense-sampling visits may be conducted after the patient has received the escalated dose for at least 2 weeks. Additional in-resident or dense-sampling visits may also be conducted in the absence of dose escalation in order to collect

additional data regarding a specific dose. Patients will have all of the same assessments conducted at the Weeks 5, 13 and 21 visits repeated at these additional inresidence or dense-sampling visit intervals.

<sup>&</sup>lt;sup>5</sup> The EOS visit is scheduled for 30 days  $\pm$  5 days after the last dose of study drug.

<sup>&</sup>lt;sup>6</sup> Patients may be considered eligible for the Extension Phase after the EOT or EOS visit; informed consent will be completed before entry into the Extension Phase.

<sup>&</sup>lt;sup>7</sup> Vital signs comprise heart rate, blood pressure, and temperature. For patients dosed in clinic for PK dense sampling, vital signs will be performed and safety laboratory tests collected pre-dose.

<sup>&</sup>lt;sup>8</sup> Safety laboratory tests – hematology and chemistry; see Section 7.2.1.1 of the Protocol for details. Safety laboratory tests may be conducted by a central or local laboratory

<sup>&</sup>lt;sup>9</sup> 12-lead ECG to be done pre-dose on Day 1 and at 2 hours post-dose during each in-residence dense PK sampling.

<sup>&</sup>lt;sup>10</sup> Ophthalmologic examination – see Section 7.1.1.8 of the Protocol for details.

<sup>&</sup>lt;sup>11</sup> Women of childbearing potential only.

<sup>&</sup>lt;sup>12</sup> Women of childbearing potential (see Section 7.4.1.1 of the Protocol for definition) will have a urine or serum pregnancy test done at the site on Day 1 and the results obtained prior to dosing.

<sup>&</sup>lt;sup>13</sup> Samples to be collected during an in-residence stay. See Section 7.1.4.1 of the Protocol for details of times for serial WBC, ANC, ALC and AMC blood samples.

<sup>&</sup>lt;sup>14</sup> WBC, ANC, ALC and AMC performed by a Central Laboratory determined by the Sponsor.

<sup>&</sup>lt;sup>15</sup> Wart assessment details are further described in Section 7.1.1.7 of the Protocol.

<sup>&</sup>lt;sup>16</sup> After consultation with the medical monitor, treatment with imiquimod to a sub-set of warts.

<sup>&</sup>lt;sup>17</sup> See Section 7.1.2 and Section 7.1.3 of the Protocol for details of times and permitted variances for collection of PK and biomarker blood samples at time 0 and during dense sampling.

<sup>&</sup>lt;sup>18</sup> Bone marrow aspirates are considered optional for this study (see Section 7.1.1.3 of the Protocol).

<sup>&</sup>lt;sup>19</sup> Daily diary for study drug administration, temperature, activities of daily living, antibiotic usage, and unscheduled healthcare visits for infection.

**Table 2: Schedule of Events – Extension Phase** 

| Procedure | Office Visits:<br>Every 6 Months<br>(±30 days) | Office Visits:<br>Every 12 Months<br>(±30 days) | End of Study<br>(30 days ±5 days) |
|---|---|---|---|
| Body weight | | X | X |
| Physical examination | | X | X |
| Vital signs (HR, BP, temp) | X | X | X |
| Safety laboratory tests (Section 7.2.1.1 of the Protocol) | X | X | X |
| Pregnancy test (WOCBP only) | X | X | X |
| Ophthalmological examination (Section 7.1.1.8 of the Protocol) | X | | |
| Mavorixafor metabolite assessment <sup>1</sup> | | X <sup>1</sup> | |
| Trough WBC, ANC, ALC, AMC, and PK sampling | | X | |
| ANC, ALC, and AMC sampling for time above threshold and AUC (optional) (Section 7.1.4.1 of the Protocol) | | X | |
| PK dense sampling (optional) (Section 7.1.2 of the Protocol) | | X | |
| Assessments of warts | | X | |
| Serum Ig and specific antibodies | | X | |
| Revaccination (optional) (Section 7.1.1.4 of the Protocol) | | X | |
| Biomarker Time 0 sample (Section 7.1.3 of the Protocol) | | X | |
| Study drug administration | Con | tinuous | |
| Diary completion <sup>2</sup> | Con | tinuous | |
| Concomitant medication monitoring | Con | tinuous | |
| Adverse event monitoring | | Continuous | |
| Quality of life questionnaires | | X | |
| Pharmacogenetic sampling (optional) <sup>3</sup> | | $X^3$ | |
| Qualitative patient interview conducted by a third party (optional) (Section 7.1.5.3) <sup>4</sup> | | $X^4$ | |
| Research blood (optional) | X | X | |

Abbreviations: ALC=Absolute lymphocyte count; AMC=Absolute monocyte count; ANC=Absolute neutrophil count; AUC=Area under the curve; BP=Blood pressure; HR=Heart rate; Ig=Immunoglobulin; PK=Pharmacokinetic; WBC=White blood cell count; WOCBP=Woman of childbearing potential.

**Note**: Home-health visits are authorized if there are extenuating circumstances that would impede patients from coming to the study site for a scheduled visit. Requests for home health visits will be reviewed and approved by X4 on a case-by-case basis. Home health visits will be an option applicable for all study visits, including screening and baseline.

<sup>&</sup>lt;sup>1</sup> A single sample will be obtained for evaluation of mavorixafor metabolites at the yearly visit (e.g., Month 12, 24, etc.), whichever occurs earliest for each patient after implementation of the v5.0 protocol amendment.

<sup>&</sup>lt;sup>2</sup> Daily diary for study drug administration, temperature, activities of daily living, antibiotic usage, and unscheduled healthcare visits for infection.

<sup>&</sup>lt;sup>3</sup> Optional assessment that may occur one time during the course of the study.

<sup>&</sup>lt;sup>4</sup> The qualitative patient interview can be performed by telephone at any time during the Extension Phase. For additional details see Section 7.1.5.3 of the Protocol.

# 4. Statistical Analysis and Reporting

After at least 4 patients have completed treatment during the Phase 2 treatment period, the DRC will review all available data and make a recommendation regarding the recommended Phase 3 dose (RP3D). At that point, the iCSR was generated summarizing all planned analyses identified in the protocol and in this SAP for the Phase 2 treatment and extension portion of the study.

A final clinical study report (CSR) summarizing all planned analyses identified in the study protocol and in this analysis plan will be generated after the last patient has completed his/her last visit and the database has been locked. Any post-hoc analysis not identified in this SAP but completed will be documented and reported in the CSR.

# 4.1. Introduction Of Statistical and Reproting Section

Descriptive statistics will be provided for all safety, exploratory and PK endpoints. The analyses results will be presented by dose levels.

For continuous variables, the number of patients (n) with non-missing values, the mean, standard deviation, median, and ranges will be provided. The minimum and maximum will be reported with the same degree of precision (i.e., the same number of decimal places) as the observed data. Measures of location (mean and median) will be reported to 1 degree of precision more than the observed data and measures of spread (standard deviation [SD]) will be reported to 2 degrees of precision more than the observed data.

For categorical variables, summaries will include the frequency and percentage of patients who are in the particular category. In general, the denominator for the percentage calculation will be based upon the total number of patients in the study population, unless otherwise specified. Percentages will be presented to 1 decimal place, unless otherwise specified.

#### 4.2. Statistical Hypothesis

Statistical hypothesis testing will be performed in order to evaluate the Phase 2 primary and exploratory objectives. All statistical analyses will be descriptive. Statistical evaluation for the primary endpoint of increase in ALC and/or ANC will be based on demonstration of a significant increase in these parameters as threshold-corrected AUC relative to clinically meaningful values, as described in protocol Section 10.4.2. The null hypothesis test is defined as an AUC  $\leq$ 0, with an alternative that the respective parameter (ALC or ANC) is  $\geq$ 0.

#### 4.3. Interim Analysis and Data Monitoring

No formal interim analyses are planned for this study; however, safety data will be reviewed by a Phase 2 DRC that includes all participating investigator(s), an independent physician with relevant experience in clinical research and/or immune deficiency diseases, the medical monitor, and a representative of the Sponsor. During the initial Treatment Phase, all available safety data will be reviewed approximately every 12 weeks by a Phase 2 DRC. During the Extension Phase, the DRC will review data approximately every 6 months. Detailed information regarding the DRC is described in the DRC Charter.

After at least 4 patients have completed 12 weeks of treatment, the DRC will review all available safety data and make recommendations regarding the course of the study. The expected outcomes of the DRC review include:

• Continuation of the Phase 2 component with further observation.

In addition, based on the experience in Phase 2 with both safety and efficacy data, a recommended dose regimen for Phase 3 will be selected by the Sponsor with input from the DRC. A subset of analyses will be performed for meetings with the scientific community (e.g., American Society for Hematology).

Once the recommended Phase 3 dose has been determined, an iCSR will be generated to summarize the open label, Phase 2 findings prior to proceeding to the Phase 3 portion of the study.

# 5. Analysis Populations

The analysis populations for this study are as follows:

- Intent to Treat (ITT): The ITT Population includes all patients who received at least one dose of the study medication(mavorixafor).
- Safety Population (SP): The Safety Population includes all patients who received at least one dose of the study medication (mavorixafor). Safety and ITT populations are identical.
- **Per Protocol (PP) Population:** All patients in the ITT population without any important protocol violations (as defined in the SAP) and at least one efficacy evaluation. Active infections during efficacy evaluation and/or missing samples may be excluded.

#### 6. General Issues for Statistical Analysis

# 6.1. General Statistical Methodology

All data will be presented in data listings. Descriptive summaries will be provided where appropriate for each of the safety and exploratory endpoints. Baseline characteristics and safety data will be summarized using the safety population unless otherwise specified.

Data processing, statistical analyses and graphical representations will be performed primarily using SAS® (version 9.4 or higher). All PK parameter estimations will be performed using Phoenix WinNonlin® software (Version 6.4 or higher; Pharsight, Cary, NC).

Unless otherwise indicated, all statistical tests will be 2-sided and tested at a significance level of p-value=0.05. All tests performed for secondary or for exploratory endpoints (specified in Section 8.1) will be exploratory in nature.

#### 6.1.1. Handling of Missing Data

For the mean of AUC<sub>ANC</sub> and/or AUC<sub>ALC</sub> during 24-hour sampling, last-observation-carried-forward (LOCF) method will be used to impute missing AUC values. Each AUC will be

calculated based on 11 samples collected over a 24-hour period. There will be no imputation for intermediate missing values within any AUC calculations during 24-hour sampling. If the last sample (the sample for 24-hour) is missing, the baseline-observation-carried-forward (BOCF) method will be used to impute the missing value. For patients who are missing all AUC assessments, the mean AUC value will be set to missing.

A sensitivity analysis will be performed in which there are no modifications made for missing data. For the Phase 2 analysis, comparisons of the results with and without imputations will be reviewed and analyzed in order to determine appropriate data handling methods to be used in a future Phase 3 trial.

The following rules will be applied to the programming logic to handle missing or partial concomitant medication dates.

For prior infection events with partial dates (day and/or month missing), the following rules will be applied to identify events occurring approximately a year before first study treatment administration and to include them as occurring 12 months prior to treatment initiation in infection reporting outputs:

- If infection onset year is the same as year of first study treatment administration, or
- If infection onset year is one less than year of first study treatment administration and initial treatment was administered in January, or
- If infection onset year is one less than year of first study treatment administration and infection onset month is on or after the month of initial treatment administration.

If the prior infection onset date is complete, then the event will be classed as taking place 12 months prior to first study treatment administration if it falls within 365 days prior to first study treatment dose.

#### **6.1.2.** Derived Variables

- Day 1 is defined as the day that first study dose is administered.
- If the assessment is prior to Day 1, then Study day = Assessment date date of Day 1; otherwise Study Day = Assessment date date of Day 1 + 1.
- Baseline = Last non-missing observation immediately prior to the first dose of study medication. For the laboratory data, if an infection event occurred ± 1 day of the baseline observation or the baseline value is 2x higher than the inclusion criteria value then the screening value will be assigned as the baseline value. If a patient had a Splenectomy prior to screening then the values can be 2x higher than the inclusion criteria.
- Change from Baseline = post baseline value value at Baseline.
- Fold-change = Value ÷ Baseline.
- Infection Rate = Number of infection events ÷ duration of treatment exposure (in years).
- Summary of dose level infection rate: 1. total number of infection events for all patients within each dose level ÷ total duration of exposure (in years) for all patient within each dose level; 2. For each patient calculate the infection rate for each dose level, then calculate the average for all patients for each dose level.
- Infection Score = (Number of infection events  $\times$  severity)  $\div$  exposure (in years).

- Summary of dose level infection score: For each patient calculate the infection score for each dose level, then calculate the average for all patients for each dose level.
- For each 6 month time interval:
  - o Infection Rate of 6 month time interval = Number of infection events occurred in 6 month time interval  $\div$  0.5.
  - o Infection Score 6 month time interval = (Number of infection events occurred in 6 month time interval  $\times$  severity)  $\div$  0.5.

#### **6.1.3. Data Conventions**

All collected data will be presented in listings. Data not subject to analysis according to this plan will not appear in any tables or figures but will be included in listings. Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) (Version 19.0 or higher). A treatment related AE is any AE with a relationship to the study drug (i.e., possibly, probably or related).

- Missing severity of an AE will be imputed to the maximum severity (In case the severity is graded and the maximum grade corresponds to death, the grade immediately below the maximum grade should be used).
- Missing relationship to study drug of an AE will be imputed to the strongest possible relationship.
- Any TEAE will be summarized under the dose level of onset.
- If the start date and the dose of onset is missing, the TEAE will be summarized in the lowest possible dose level the patient received.

#### 6.1.4. Calculation of the AUC<sub>ANC</sub> and/or AUC<sub>ALC</sub>

The ANC and ALC sampling will be performed during the in-residence stays. The area under curve (AUC) for each parameter ANC and ALC will be calculated and analyzed relative to pre-specified clinically meaningful thresholds of AUC<sub>ANC</sub>  $\geq 600/\mu L$  and AUC<sub>ALC</sub>  $\geq 1000/\mu L$ , respectively. A separate table for AUC for ANC by dose level will be presented where the threshold of AUC<sub>ANC</sub>  $\geq 500/\mu L$ .

Patients are scheduled for 24-hour measurements of ANC and ALC via blood samples collected as follows:

• Time 0 (-15 min), 30, 60, 90 min (each  $\pm$  5 min) and 2, 3, 4, 8, 12, 16, 24 hr (each  $\pm$ 15 min)

Additional visits may occur at the discretion of the Sponsor and with the agreement of the Investigator both during the 24-week treatment period and/or the Extension Phase. For patients receiving study drug, time 0 represents time of oral dosing that morning (typically between 7 and 8 am) and the sample will be drawn pre-dose. The 24-hour AUC will be calculated using the trapezoidal rule with area above threshold being positive, and area below threshold, negative. The results are referred to as threshold-adjusted AUC.

Patients with AUC<sub>ANC</sub> <2000 cell•hr/ $\mu$ L or AUC<sub>ALC</sub> <5000 cell•hr/ $\mu$ L after an in-residence stay will have X4P-001 daily dose increased in 100 mg increments up to a maximum daily dose of 400 mg QD.



Figure 1: Calculation of 24-hr AUC for a Hypothetical Set of ALC Data.

Abbreviations: ALC=Absolute lymphocyte count; AUC=Area under the curve. Note: 24-hr AUC is the net sum of the interval areas.

To calculate the AUC above the clinically meaningful threshold for each in-residence stay, the area below the clinically meaningful threshold will be subtracted from the total AUC. Figure 1 illustrates the calculation of the AUC for ALC, where the red shaded area represents the area below the clinically meaningful threshold of  $1000/\mu L$ , and the vertical blue lines represent the data collection time points.

Patients with fewer than the required 3 AUC calculations for ANC or ALC, as appropriate, will have the last available AUC carried forward for calculation of the mean of 3 AUC values post-treatment.

Box-plots of AUC for ANC at doses up to 400 mg doses will be generated. The mean ANC, ALC and absolute monocyte count (AMC) values will be plotted from 0-24 hours at all the dose levels.

#### 6.1.5. Time above threshold analysis

Patients are scheduled for 24-hour measurements of ANC and ALC via blood samples collected at the following scheduled timepoints: Time 0 (-15 min), 30, 60, 90 min (each  $\pm$  5 min) and 2, 3,

4, 8, 12, 16, 24 hr (each  $\pm 15$  min). During these time points, the time above thereshold is the total time a patients ANC and ALC values were above a pre-defined threshold. The threshold is defined as 500/uL for ANC and as 1000/uL for ALC. For example, if a patients ANC value is 600 at 30 mins and 700 at 60 mins, then the patients ANC values was above the threshold for 30 mins (60 mins -30 mins). If the ANC value was 800 at 4 hours and 400 at 8 hours then the patients ANC value was above the threshold from 4 hours until the time between 4 and 8 hours when the ANC value went below the pre-defined threshold of 500. This time is estimated using linear interpolation.

The time above threshold will be calculated for AMC based on the age and gender specific threshold as described in the following table:

| Age (year) | Gender Threshold (/uL) | |
|------------|------------------------|-----|
| >=18 | F | 250 |
| | M | 290 |

A scatter plot showing the correlation of time above threshold for ANC, ALC vs AUC for ANC and ALC will be generated.

The dense samples collected on 9<sup>th</sup> to 10<sup>th</sup> October 2017 (Extension visit 1, 300mg dose) for patient the dense samples collected on 12<sup>th</sup> to 13<sup>th</sup> February 2018 (Extension visit 3, 400mg dose) for patient the dense samples collected on 21<sup>st</sup> February 2018 (Week 21, 400mg dose) for patient the occurred during an infection event. These values will be excluded from the summary tables of absolute WBC, ANC, ALC, AMC; and TAT and AUC of ANC, ALC, and AMC. Dense sample data for subject the will be excluded from the TAT summary tables and figures since the WBC, ANC, ALC, and AMC levels were normal at screening.

As a sensitivity <u>analysis</u>, separate summary tables of TAT will be presented including the dense sample data for ...

#### 6.1.6. Re-enrollment due to COVID-19

The re-enrollment visit for the two patients ( , ) who dropped out the study due to study fatigue for about 6 months (400mg dose), and were re-enrolled on the study due to the fear of infection during the covid pandemic, will be mapped as Extension Visit 6 (re-enroll). All data will be presented in the listings. Data within the drop-out period will be excluded from the summary tables for infection, warts and other safety data analyses.

#### 7. Study Patients and Demographics

#### 7.1. Disposition of Patients and Withdrawals

The patient disposition table will include the number and percentage of patients who completed the initiation phase of the study, the number and percentage of patients entered into the extension phase, the number and percentage of patients who discontinue from the study along with the reasons for discontinuation, and number and percentage of patients analysis population The percentage in this table will be based on all patients enrolled in the Phase 2 study.

#### 7.2. Protocol Violations and Deviations

Protocol deviations will be identified and classified as non-important or important and if COVID-19-related, and reviewed when preparing the Phase 2 analysis prior to the final database lock. Protocol deviations will be summarized by catogory using the Safety population.

# 7.3. Demographics and Other Baseline Characteristics

Descriptive summaries of demographics and other baseline conditions will include age, gender, race, ethnicity, height, weight, body mass index (BMI) and will be presented by dose levels and capsule strength received.

#### 7.4. Medical History

The number and percent of patients reporting medical histories, grouped by MedDRA system organ class (SOC) and preferred term (PT) (coded using MedDRA Version 19.0 or higher), will be presented by dose level and a listing will be provided. Similarly, the history of WHIM syndrome manifestations (i.e., date of diagnosis, mutational status, and the following history in the 12 months prior to study entry: hospitalizations for infection, number and type of infections managed as an out-patient, any prior medical treatments for WHIM disease) will be summarized and presented by dose level and a listing will be provided. The Safety population will be used to perform these analyses.

# 8. Efficacy Analysis

#### 8.1. Primary Efficacy Analysis

The AUC<sub>ANC</sub> and/or AUC<sub>ALC</sub> will be analyzed by week using descriptive statistics and presented by dose level. A patient listing of the AUC values will be provided.

The primary efficacy analysis will be performed with the missing data handling method described in Section 6.1.1 and without imputations.

#### 8.2. Exploratory Efficacy Analysis

The following exploratory analyses will be performed:

- Time above threshold values for ANC, AMC, and ALC, as applicable, will be calculated using the ANC, AMC, and ALC assessments collected during the 24-hour collection times and analyzed as percentage of time (from initial to final value obtained during each of these visits) above the clinically meaningful thresholds of 500/µL and 1000/µL (Time (hours) >ANC Threshold<sub>500</sub>, Time (hours) >ALC Threshold<sub>1000</sub>, and age and gender specific AMC thresholds), respectively. These parameters will be compared between dose levels to determine if there is a dose-dependent change in the respective Time (hours)>Thresholds.
- **Frequency and severity of infections** (severity assessed as Grade 1 to 5 using NCI CTCAE Version 4.03 or higher).

- Number of warts applicable only to patients with cutaneous warts at baseline and comparing number of warts to that at end of Treatment Period.
- **Severity of genital warts** applicable only to patients with genital warts, and comparing number of lesions, size of largest lesion, and patient-reported morbidity.
- Improvement in antibody levels following revaccination applicable only to patients who were (a) previously administered approved vaccines, (b) found at baseline to have predefined sub-protective levels of antibody, and (c) agree to repeat administration of the vaccine after 12 weeks of treatment.
- Frequency of events requiring rescue therapy (granulocyte-colony stimulating factor [G-CSF] and/or intravenous immunoglobulins [Ig]).
- Rate of hospitalization events for the X4P-001 treated patients will be evaluated based on the information collected in the 12 months prior to start of participation in Study X4P-001-MKKA through end of Phase 2 Treatment Period or data cutoff for the iCSR.
- Circulating white blood cells (WBCs) Absolute and fold change from baseline in total WBC counts, and in absolute numbers of lymphocytes, neutrophils, monocytes, and lymphocyte subpopulations cells. Correlation of ANC and ALC levels with plasma drug levels

# • Ig and specific antibodies

- Changes from baseline in levels of total IgG, IgG subclasses, IgA, IgD, IgE and IgM.
- **Bone marrow aspirates** (analyzed centrally by a blinded reviewer) Change from baseline in cellularity. Change from baseline in frequency of apoptotic cells.
- Quality of Life as assessed by SF-36, LQI and HIP.

The Safety population will be used to perform all the exploratory analyses.

# 8.3. Subgroup Analysis

There are no planned subgroup analyses for the Phase 2 study.

#### 9. Safety and Tolerability Analysis

Safety variables will include TEAEs, SAEs, deaths, discontinuations due to AEs, vital signs, physical examinations, ophthalmology, laboratory tests, 12-Lead electrocardiograms (ECG), , concomitant medications and study drug exposure. The safety population will be used to perform these analyses.

### 9.1. Adverse Events

Adverse events will be coded using MedDRA Version 19.0 or higher. The severity of an AE will be graded according to the NCI CTCAE, Version 4.03 or higher.

The causal relationship of an AE to the study drug is determined by the investigator as Unrelated, Unlikely Related, Possibly Related, Probably Related, and Definitely Related. These will be mapped to Unrelated (Unrelated and Unlikely Related) and Related (Possibly Related, Probably Related, and Definitely Related). A summary table will be presented for the following:

- All TEAEs
- TEAEs all grades and grade 3 or higher
- TEAEs by relationship to study drug all grades and grade 3 or higher
- TEAEs leading to discontinuation of study drug
- SAEs regardless of causality and treatment related
- AEs leading to death
- AEs of special interest
- TLTs

TEAEs are defined as any AEs that begin or worsen on or after the start of study drug through 10 days after the last dose of study drug.

The incidence of TEAEs will be summarized by SOC and PT. TEAEs will also be summarized using Investigator assessment of the relationship to study drug (related or not related) and by maximum severity. TEAEs leading to study drug discontinuation and those resulting in premature withdrawal from study will be tabulated and listed.

If a patient experiences multiple AEs under the same PT within a SOC, then the patient will be counted only once for that PT within that SOC. If a patient experiences the same AE more than once with different intensity or grade, then the event with the highest grade will be tabulated in "by grade" tables.

# 9.1.1. Adverse Events Leading to Withdrawal

Summary tables of TEAEs leading to the discontinuation of the study drug and AEs leading to premature withdrawal from the study will be provided. Data listings will be provided as well.

#### 9.1.2. Deaths and Serious Adverse Events

A summary of serious adverse events will be provided by SOC and PT and presented by dose level. The SAEs will also be listed. In addition, any deaths that occur during the study will be listed.

#### 9.1.3. Treatment Limiting Toxicities

A TLT event for X4P-001 is defined as an AE that meets *both* of the following criteria:

- 1. Is assessed by the Investigator as possibly or probably related, or related to X4P-001 (see Section 8.2.3 of the study Protocol).
- 2. Represents one of the following events (grading as defined by the NCI CTCAE, v4.03 or higher) (see Section 8.2.1 of the study Protocol):
  - Is a Grade 3 or Grade 4 clinical event, except grade 3 nausea, vomiting, or diarrhea lasting <48 hrs in patients who have received suboptimal medical management.
  - Is a confirmed Grade 3 or Grade 4 laboratory event with the following exceptions:
    - Grade 3 electrolyte abnormalities that persist <72 hrs and do not require hospitalization.

- o Grade 3 AST/ALT increases that persist <5 days and with total bilirubin ≤1.5x ULN.
- Is one of the following, which are designated as critical TLT events:
  - o AST/ALT increased >3x ULN (Grade 2) with total bilirubin increased >2x ULN in the absence of cholestasis.
  - o Retinopathy confirmed treatment-emergent retinopathy.
  - o Platelets <50,000/mm<sup>3</sup> (Grade 3) with bleeding or <25,000/mm<sup>3</sup> (Grade 4).

A summary of TLTs will be provided by SOC and PT and presented by dose level.

# 9.2. Clinical Laboratory Evaluations

Laboratory safety tests will be performed by central (CRL and Cerba Research) and local lab facilities. Descriptive summaries of actual (absolute) values and changes from baseline values will be provided for hematology and chemistry by dose level and visit.

For tests with categorical results, the number and percentage of patients in each category will be provided by dose level. In the event of repeat test results, the last non-missing value per study day/time will be used.

A shift table presenting the number and percentage of patients with clinical laboratory values classified as below, within, or above the normal range at post baseline visit and in relation to baseline will be provided for each clinical laboratory analyte (i.e., hematology and chemistry).

A listing for the laboratory test results will be provided and all values that are outside the normal range will be flagged.

As central labs changed from CRL to Cerba Research during the study a correction factor needs to be applied to the test results from Cerba Research as specified in the table below to standardise the results and align them with the original central lab data. The correction will not need to be applied to the normal ranges.

For the local lab values, no conversion will be performed.

**Table 3: Overview of Conversion Factors** 

| | USA patients | | | AUS patients | | |
|---|---|---|---|---|---|---|
| Test | Testing lab<br>at CRL | Testing lab at<br>Cerba Research | Correction factor | Testing lab<br>at CRL | Testing lab at Cerba<br>Research | Correction factor |
| Rubella<br>IgG | LabCorp | Cerba (France) Paris | N A | Sydpath | Cerba (France) Paris | N A |
| Rubeola<br>IgG | CRL USA | Cerba (France) Paris | N A | Sydpath | Cerba (France) Paris | N A |
| IgG1 | LabCorp | Cerba (France) Paris | LabCorp (g/L) = 1.310804<br>+ 0.791798 * CerbaCR FRA<br>(g/L) | Sydpath | Cerba (France) Paris | Sydpath (g/L) = 1.411672+<br>1.037855 * CerbaCR FRA<br>(g/L) |
| IgG2 | LabCorp | Cerba (France) Paris | LabCorp (g/L) = 0.746442<br>+ 0.817308 * CerbaCR FRA<br>(g/L) | Sydpath | Cerba (France) Paris | N A |
| IgG3 | LabCorp | Cerba (France) Paris | LabCorp $(g/L) = 0.08375 + 0.875 * CerbaCR FRA (g/L)$ | Sydpath | Cerba (France) Paris | Sydpath (g/L) = 0.0304221 -<br>0.466234 * CerbaCR FRA<br>(g/L) |
| IgG4 | LabCorp | Cerba (France) Paris | LabCorp (g/L) = 0.0590315 + 0.788288 * CR FRA (g/L) | Sydpath | Cerba (France) Paris | Sydpath (g/L) = 0.0226538 - 1.230769 * CR FRA (g/L) |
| IgG | LabCorp | NWHL | LabCorp (mg/dL) = 17.410089<br>+ 1.074362 * CR USA (mg/dL) | Sydpath | SDS<br>Laverty | N A |
| IgA | LabCorp | NWHL | LabCorp (mg/dL) = -8.2 +<br>1.085714 * CR USA (mg/dL) | Sydpath | SDS<br>Laverty | N A |
| IgE | CRL USA | NWHL | CRL USA (IU/mL) =-0.858757<br>+ 0.817047 * CR USA (IU/mL) | Sydpath | SDS<br>Laverty | Sydpath (IU/mL) =<br>11.903864 + 1.005829 * CF<br>AUS (IU/mL) |
| IgM | CRL USA | NWHL | N A | Sydpath | SDS<br>Laverty | N A |

# 9.3. Vital Signs

Descriptive summaries of actual (absolute) values and changes from baseline values will be provided for vital signs including weight (kg), heart rate (bpm), systolic blood pressure (mmHg), diastolic blood pressure (mmHg), and temperature (°C) by dose level.

A listing of the vital sign measurements will also be provided. Results outside the normal range will be flagged.

#### 9.4. Electrocardiograms

The following ECG parameters will be recorded: HR, RR, PR interval, QRS, QT, QTc interval (the correction method QTcF will be calculated).

Descriptive summaries of actual values and changes from baseline to each visit will be presented for ECG measures of HR (bpm), RR interval (ms), PR interval (ms), QRS (ms), QT (ms), and QTc interval (ms). These summaries will be presented by treatment group as appropriate.

Shift tables comparing baseline ECG investigator interpretation (normal, abnormal, not clinically significant or abnormal, clinically significant) to each study visit will be summarized by dose level.

#### 9.5. Concomitant Medication

Prior medications as well as prior WHIM treatment, and concomitant medications will be summarized descriptively using counts and percentages of patients taking each medication, classified using World Health Organization Drug Dictionary (WHO-DD) Anatomical Therapeutic Chemical (ATC) classes and PT. Prior WHIM medications, prior medications and concomitant medications will be presented separately. The use of antibiotics, G-CSF, Immunoglobulins, and imiquamod will be tabulated separately.

- A prior medication is any medication that is started or ended prior to the first dose of the study medication.
- A concomitant medication is any medication taken or ongoing on or after the first dose of the study medication.
- A medication is both prior and concomitant if it started prior to and is ongoing on or after the first dose of the study medication.

# 9.6. Exposure and Compliance

The study drug will be dispensed in bottles and using a web-based treatment diary, each patient will record the number of capsules taken. The bottles will be examined visually at each clinic visit for the purpose of assessing study drug compliance. Percent compliance will be calculated as follows:  $[1 - (\text{Total number of capsules returned/Total number of capsules dispensed})] \times 100$ . Patient compliance with study drug will be summarized by patient, treatment duration overall, dose, treatment duration by dose and capsule strength. All study drug administration data will be displayed in a listing.

# 10. Changes from Planned Analysis

The following analyses were not described in the protocol but will be presented in the TLFs:

- A separate table for AUC for ANC by dose level will be presented where the threshold of  $AUC_{ANC} \ge 500/\mu L$ .
- As a sensitivity analysis, separate summary tables of TAT will be presented including the dense sample data for ...

# 11. Other Planned Analysis

#### 11.1. Pharmacokinetic and Pharmacodynamic (PK/PD) Analysis

# Pharmacokinetic Analysis

The PK parameters (AUC,  $T_{max}$  and  $C_{max}$ ), will be determined for each patient following each specified visit, using a non-compartmental analysis based on the plasma concentration versus time dataset. Additional parameters may be estimated if warranted and if data permit.

Plasma X4P-001 concentration and PK parameters (AUC, C<sub>max</sub>, T<sub>max</sub>) will be summarized at each timepoint using descriptive statistics, including number of patients, arithmetic mean, geometric mean, SD, median, maximum, minimum, and coefficient of variation (%CV). These summaries will be presented by dose level. All figures will be presented using both linear and semi-logarithmic scales. All plasma concentration data and PK parameters will be displayed in data listings.

Plasma concentration of X4P-001 below the limit of quantification (BLQ) occurring before  $T_{max}$  will be set to 0. BLQ plasma concentrations occurring after  $T_{max}$  will be set to missing. If sufficient data are missing for a given patient, that patient may be considered non-evaluable for PK analysis. All plasma concentration data and PK parameters will be displayed in data listings. The above descriptive summary will be performed using the PK population.

#### Pharmacodynamic Analysis

AUC of ANC and ALC will be determined for each patient and each dose level. Individual ANC/ALC values vs time will be plotted. Mean ANC/ALC values vs time will be plotted by dose level. X4P-001 concentration vs ANC/ALC by timepoint will be presented in scatter plots by dose.

The PK and PD data collected in this study may be combined with data from other studies in a population pharmacokinetic (pop PK) analysis to assess covariate effects on the PK of X4P-001 and the PKPD correlation between exposure and ANC/ALC to support dose selection. A separate PK analysis plan will be developed.

#### 11.2. Biomarker Analysis

Biomarker data will be summarized descriptively, including actual value and change from baseline. Summaries will be presented overall. All biomarker data will be displayed in data listings with the cell subset name such as naïve T cells, memory T cells, B cells, transitional B cells, NK cells, and monocytes mentioned in the protocol. The above descriptive summary will be performed using the safety population

#### 12. References

- 1. Study protocol X4P-001-MKKA version 5.0 dated 21 December 2020
- 2. Study eCRF version 12.0 dated 17 February 2021
- 3. ASA. (1999) Ethical Guidelines for Statistical Practice. Prepared by the Committee on Professional Ethics, August 7, 1999. http://www.amstat.org/about/ethicalguidelines.cfm
- 4. US Federal Register. (1998) International Conference on Harmonization; Guidance on Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration [Docket No. 97D-0174]. Federal Register Volume 63, Number 179, pages 49583-49598. September 16, 1998.
- 5. McDermott DH, Liu Q, Velez D, et al. A phase 1 clinical trial of long-term, low-dose treatment of WHIM syndrome with the CXCR4 antagonist plerixafor. Blood. 2014;123 (15):2308-16.
## 13. Tables, Listings, and Figures

## 13.1. Planned Table Descriptions

The following are planned summary tables for protocol X4P-001-MKKA. Tables will be numbered according to the nomenclature used to support the CSR when the Premier Research CSR template is used. However, the table numbering structure can be modified per the sponsor's request to meet compatibility with the sponsor's CSR template.

### 13.2. Demographic Data

**Table 1: Demographic Data Summary Tables** 

| Table 1. Demographic Data Summary Tables | | |
|---|---|---|
| Table<br>Number | Population | Table Title/Summary |
| 14.1 Display | s of Demographics an | d Disposition Data |
| 14.1.1 | Informed Consent<br>Signed | Subject Disposition |
| 14.1.2 | Safety Population | Summary of Protocol Deviations |
| 14.1.3 | Safety Population | Demographics and Baseline Characteristics |
| 14.1.4 | Safety Population | Summary of Study Drug Exposure |
| 14.1.5 | Safety Population | Summary of Medical History |

## 13.3. Efficacy Data

**Table 2: Efficacy Data Summary Tables** 

| Table<br>Number | Population | Table Title/Summary |
|---|---|---|
| 14.2 Display | s of Exploratory Sum | maries |
| 14.2.1.1 | Safety Population | Summary of AUCs and Mean of AUCs for ANC by Dose Level - $AUC_{ANC} \ge 600/\mu L$ Threshold |
| 14.2.1.1.1 | Safety Population | Summary of AUCs and Mean of AUCs for ANC by Dose Level - $AUC_{ANC} \ge 500/\mu L$ Threshold |
| 14.2.1.2 | Safety Population | Summary of AUCs and Mean of AUCs for ALC by Dose Level |
| 14.2.2.1 | Safety Population | Summary of Infection Rates |
| 14.2.2.2 | Safety Population | Summary of Infections by Severity |
| 14.2.2.3 | Safety Population | Summary of Highest Grade Infections |
| 14.2.2.4 | Safety Population | Summary of Infection Scores |
| 14.2.3.1 | Safety Population | Summary of Non-Genital Warts |
| 14.2.3.2 | Safety Population | |
| 14.2.4.1 | Safety Population | Summary of Genital Warts |
| 14.2.5 | Safety Population | Summary of Antibody levels Following Revaccination |
| 14.2.6 | Safety Population | Summary of Rescue Medications |
| 14.2.7 | Safety Population | Summary of Hospitalizations |
| 14.2.8 | Safety Population | Summary of Ig and Specified Antibodies |
| 14.2.9 | Safety Population | Time above Threshold for ANC by Dose Level |
| 14.2.9.1 | Safety Population | Time above Threshold for ANC by Dose Level Sensitivity |
| 14.2.10 | Safety Population | Time above Threshold for ALC by Dose Level |
| 14.2.10.1 | Safety Population | Time above Threshold for ALC by Dose Level – Sensitivity<br>Analysis |
| 14.2.11 | Safety Population | Time above Threshold for Monocytes by Dose Level |

| 142111 | G C . B 1 .: | Time above Threshold for Monocytes by Dose Level – Sensitivity |
|---|---|---|
| 14.2.11.1 | Safety Population | Time above Threshold for Monocytes by Dose Level – Sensitivity Analysis |

## 13.4. Safety Data

| Table 3: Safety Data Summary Tables | | |
|---|---|---|
| Table<br>Number | Population | Table Title/Summary |
| | | ergent Adverse Events |
| 14.3.1.1 | Safety Population | Overall Summary of Treatment-Emergent Adverse Events |
| 14.3.1.2 | Safety Population | Summary of Treatment-Emergent Adverse Events by System<br>Organ Class and Preferred Term |
| 14.3.1.3 | Safety Population | Summary of Treatment-Emergent Adverse Events Related to<br>Study Treatment by System Organ Class and Preferred Term |
| 14.3.2 Sumn | nary of Deaths, Other | Serious and Significant Adverse Events |
| 14.3.2.1 | Safety Population | Summary of Serious Adverse Events by System Organ Class and Preferred Term |
| 14.3.2.2 | Safety Population | Summary of Serious Adverse Events Related to Study Treatment<br>by System Organ Class and Preferred Term |
| 14.3.2.3 | Safety Population | Summary of treatment-limiting toxicities by System Organ Class and Preferred Term |
| 14.3.2.4 | Safety Population | Summary of Grade 3 or Higher Treatment-Emergent Adverse<br>Events by System Organ Class and Preferred Term |
| 14.3.2.5 | Safety Population | Rate of Treatment Emergent Adverse Events by System Organ<br>Class and Preferred Term |
| 14.3.2.6.1 | Safety Population | Summary of Yearly Infection Rate for Subjects on 300mg and 400mg Dose Levels by 6 Month Intervals |
| 14.3.2.6.2 | Safety Population | Summary of Yearly Infection Score for Subjects on 300mg and 400mg Dose Levels by 6 Month Intervals |
| 14.3.2.7.1 | Safety Population | Summary of Yearly Infection Rate by Dose Level - Method 1 |
| 14.3.2.7.2 | Safety Population | Summary of Yearly Infection Rate by Dose Level – Method 2 |
| 14.3.3 Narra | tives of Deaths, Other | Serious and Certain Other Significant Adverse Events |
| 14.3.3.1 | Safety Population | Listing of Serious Adverse Events |
| 14.3.3.2 | Safety Population | Listing of Treatment Emergent Adverse Events Leading to Discontinuation |
| 14.3.4 Abno | rmal Laboratory Valu | ie |
| 14.3.4.1 | Safety Population | Listing of Out of Reference Range Laboratory Values |
| 14.3.5 Labor | ratory Data Summary | Tables |
| 14.3.5.1.1 | Safety Population | Summary of actual and Change from Baseline in Hematology<br>Results |
| 14.3.5.1.2 | Safety Population | Shift from Baseline in Hematology Results |
| 14.3.5.2.1 | Safety Population | Summary of actual and Change from Baseline in Serum<br>Chemistry Results |
| 14.3.5.2.2 | Safety Population | Shift from Baseline in Serum Chemistry Results |
| 14.3.5.3.1 | Safety Population | Summary of actual and Change from Baseline in Coagulation Results |
| 14.3.5.3.2 | Safety Population | Shift from Baseline in Coagulation Results |
| 14.3.5.4.1 | Safety Population | Summary of actual and Change from Baseline in Cytometry Results |
| 14.3.6 Other | Safety Data Summar | y Tables |
| 14.3.6.1.1 | Safety Population | Summary of actual and Change from Baseline in Vital Signs |
| 14.3.6.2.1 | Safety Population | Summary of actual and Change from Baseline of 12-Lead<br>Electrocardiogram (ECG) Parameters |

| 14.3.6.3.1 | Safety Population | Summary of Ophthalmologic Examination Results (Local Reader) |
|---|---|---|
| 14.3.6.3.2 | Safety Population | Summary of Ophthalmologic Examination Results (Central |
| | | Retinal Findings) |
| 14.3.6.4 | Safety Population | Summary of Concomitant Medications |
| 14.3.6.5.1 | Safety Population | Summary of Use of Antibiotics, G-CSF, Immunoglobulins, and |
| | | imiquamod - Concomitant Medications |
| 14.3.6.5.2 | Safety Population | Summary of Use of Antibiotics, G-CSF, Immunoglobulins, and |
| | | imiquamod – Prior Medications |
| 14.3.6.6 | Safety Population | Summary of SF-36 QOL |
| 14.3.6.7 | Safety Population | Summary of HPV Impact Profile (HIP) Questionnaire |

### 13.5. Pharmacokinetic Data

**Table 4: Pharmacokinetic Data Summary Tables** 

| <b>Table Number</b> | Population | Table Title/Summary |
|---|---|---|
| 14.4 Pharmacok | inetic Data Summary Ta | ables |
| 14.4.1 | Safety Population | Summary of Plasma X4P-001 Concentrations by Dose Level |
| 14.4.2 | Safety Population | Summary of Plasma X4P-001 Pharmacokinetic Parameters by Dose Level |

### 13.6. Planned Listing Descriptions

The following are planned patient data listings for protocol X4P-001-MKKA. Data listings will be numbered according to the nomenclature used to support the CSR when the Premier Research CSR template is used. However, the listing numbering structure can be modified per the sponsor's request to meet compatibility with the sponsor's CSR template.

**Table 5: Planned Listings** 

| Data Listing<br>Number | Population | Data Listing Title / Summary |
|---|---|---|
| 16.2.1 Patient D | iscontinuations/Completi | ons |
| 16.2.1 | All Enrolled Patients | Subject Disposition |
| 16.2.2 Protocol | Deviations | |
| 16.2.2.1 | All Enrolled Patients | Eligibility Criteria Not Met |
| 16.2.2.2 | Safety Population | Protocol Deviations |
| 16.2.3 Analyses | Populations | |
| 16.2.3 | All Enrolled Patients | Analysis Populations |
| 16.2.4 Demogra | phic Data and Other Bas | eline Characteristics |
| 16.2.4.1 | Safety Population | Demographics and Baseline Characteristics |
| 16.2.4.2 | Safety Population | Medical History |
| 16.2.4.3.1 | Safety Population | History of WHIM Syndrome - Hospitalizations |
| 16.2.4.3.2 | Safety Population | History of WHIM Syndrome - Infections Managed as Out-<br>Patient |
| 16.2.4.3.3 | Safety Population | History of WHIM Syndrome - Prior Treatments of WHIM Syndrome |
| 16.2.4.3.4 | Safety Population | WHIM Syndrome Genotyping |
| 16.2.4.4.1 | Safety Population | Study Drug Administration |
| 16.2.4.4.2 | Safety Population | Study Drug Exposure |
| 16.2.4.5 | Safety Population | Assessment of Warts |
| 16.2.4.6 | Safety Population | Revaccination |
| 16.2.4.7 | Safety Population | Bone Marrow Aspirate |

| 16.2.5 Drug Concentration Data | | |
|---|---|---|
| 16.2.5.1 | Safety Population | Pharmacokinetic Blood Collection and Concentrations |
| 16.2.5.2 | Safety Population | Calculated Pharmacokinetic Parameters |
| 16.2.5.3 | Safety Population | PK Sample Collection |
| | al Efficacy Response Dat | |
| 16.2.6.1 | Safety Population | ANC/ALC Sample Collection |
| 16.2.6.2.1 | Safety Population | Threshold Adjusted AUC values for ANC |
| 16.2.6.2.2 | Safety Population | Threshold Adjusted AUC values for ALC |
| 16.2.6.2.3 | Safety Population | Time Above Threshold by Dose Level - Assessment of |
| 160604 | | ANC/ALC/AMC |
| 16.2.6.2.4 | Safety Population | Time Above Threshold - Pharmacodynamic Assessment of ANC/ALC/AMC with Time Crossed |
| <b>16.2.7</b> Adverse | <b>Event Listings (by Patier</b> | nt) |
| 16.2.7.1 | Safety Population | Treatment Emergent Adverse Events |
| 16.2.7.2 | Safety Population | Adverse Events that occur during Screening and ended before Exposure to study Drug |
| 16.2.7.3 | Safety Population | Infections Reported as Adverse Events |
| 16.2.7.4 | Safety Population | Deaths |
| 16.2.7.5 | Safety Population | Treatment Limiting Toxicities |
| 16.2.7.6 | Safety Population | Infections in Subjects Treated on 300mg or 400mg Dose by Time Period |
| 16.2.7.7 | Safety Population | Infections by Dose Level |
| 16.2.7.8 | Safety Population | Infections by Subject |
| | ory Values by Patient | |
| 16.2.8.1 | Safety Population | Clinical Laboratory Data: Serum Chemistry |
| 16.2.8.2 | Safety Population | Clinical Laboratory Data: Hematology |
| 16.2.8.3 | Safety Population | Serology and Other Laboratory Test Results |
| 16.2.8.4 | Safety Population | Serum Ig and Specific Antibody Laboratory Test Results |
| 16.2.8.5 | Safety Population | Pregnancy Test Results |
| 16.2.8.6 | Safety Population | Coagulation Laboratory Test Results |
| 16.2.8.7 | Safety Population | Urinalysis Laboratory Test Results |
| 16.2.8.8 | Safety Population | Cytometry Test Results |
| | | Measurements (by Patient) |
| 16.2.9.1 | Safety Population | Prior or Concomitant Medications |
| 16.2.9.2 | Safety Population | Vital Signs Measurements |
| 16.2.9.3 | Safety Population | 12-Lead Electrocardiograms |
| 16.2.9.4 | Safety Population | Physical Examinations |
| 16.2.9.5 | Safety Population | Ophthalmologic Examination (Site Assessment) |
| 16.2.9.6 | Safety Population | Ophthalmologic Examination (Central Readings) |
| 16.2.9.7 | Safety Population | Rescue Medications |
| 16.2.9.8 | Safety Population | SF-36 QOL |
| 16.2.9.9.1 | Safety Population | HPV Impact Profile (HIP) Questionnaire |
| 16.2.9.9.1 | Safety Population | HPV Impact Profile (HIP) Questionnaire - Domain Scores |

## 13.7. Planned Figure Descriptions

The following are planned summary figures for protocol X4P-001-MKKA. They will be numbered according to the nomenclature used to support the CSR when the Premier Research CSR template is used. However, the figure numbering structure can be modified per the sponsor's request to meet compatibility with the sponsor's CSR template.

**Table 6: Planned Figures** 

| Figure Number | Population | Figure Title/Summary |
|---|---|---|
| Figure 14.4.1.1 | Safety Population | WBC Over Time by Patient |
| Figure 14.4.1.2a | Safety Population | ANC Over Time by Patient |
| Figure 14.4.1.2b | Safety Population | ANC Over Time by Dose Level |
| Figure 14.4.1.3a | Safety Population | ALC Over Time by Patient |
| Figure 14.4.1.3b | Safety Population | ALC Over Time by Dose Level |
| Figure 14.4.1.4a | Safety Population | Monocytes Over Time by Patient |
| Figure 14.4.1.4b | Safety Population | Monocytes Over Time by Dose Level |
| Figure 14.4.1.5 | Safety Population | Mean (+/- SE) Plasma Concentration - Time Profile of X4P-001 by Dose Level |
| Figure 14.4.1.6 | Safety Population | Mean Dose Response of ANC-Time Profile |
| Figure 14.4.1.7 | Safety Population | Mean Dose Response of ALC-Time Profile |
| Figure 14.4.1.8 | Safety Population | Mean Dose Response of Monocytes-Time Profile |
| Figure 14.4.1.9 | Safety Population | Box plots of WBC change from baseline ratio at 300mg |
| riguic 14.4.1.) | Safety Topulation | and 400mg by Dose Level |
| Figure 14.4.1.10 | Safety Population | Box plots of AUC for ANC by Dose Level |
| Figure 14.4.1.11 | Safety Population | Scatter Plot of Time above Threshold values for ANC |
| | | versus AUC for ANC |
| Figure 14.4.1.12 | Safety Population | Scatter Plot of Time above Threshold values for ALC |
| | | versus AUC for ALC |
| Figure 14.4.1.13.1 | Safety Population | Plot of Yearly Infection Rate by Dose Level |
| Figure 14.4.1.13.2 | Safety Population | Plot of Yearly Infection Score by Dose Level |
| Figure 14.4.1.14.1 | Safety Population | Plot of Yearly Infection Rate for Subjects on 300mg and 400mg Dose Levels by 6 Month Intervals |
| Figure 14.4.1.14.2 | Safety Population | Plot of Yearly Infection Score for Subjects on 300mg |
| rigure 14.4.1.14.2 | Safety Population | and 400mg Dose Levels by 6 Month Intervals |
| Figure 14.4.2.1 | Safety Population | Scatter Plot of Plasma Drug Level and ANC |
| Figure 14.4.2.2 | Safety Population | Scatter Plot of Plasma Drug Level and ALC |
| Figure 14.4.3.1 | Safety Population | Mean Plasma Concentrations of X4P-001 vs Nominal |
| 11guic 14.4.5.1 | Surety Topulation | Time (Dense Sampling Visits) by Dose Level - Linear |
| | | Scale |
| Figure 14.4.3.2 | Safety Population | Mean Plasma Concentrations of X4P-001 vs Nominal |
| | J 1 | Time (Dense Sampling Visits) by Dose Level - |
| | | Semi-logarithmic Scale |
| Figure 14.4.4.1 | Safety Population | Subject Plasma Concentrations of X4P-001 vs Nominal |
| _ | | Time (Dense Sampling Visits) by Dose Level - Linear |
| | | Scale |
| Figure 14.4.4.2 | Safety Population | Subject Plasma Concentrations of X4P-001 vs Nominal |
| | | Time (Dense Sampling Visits) by Dose Level - |
| | | Semi-logarithmic Scale |

## 14. Tables, Listings, and Figure Shells

## 14.1. Standard Layout for all Tables, Listings, and Figures

The following standard layout will be applied to all Tables, Listings, and Figures in support of this study. Note that programming notes may be added if appropriate after each TLF shell.

## 14.2. Planned Table Shells

## Table 14.1.1 Subject Disposition Informed Consent Signed

| Disposition | Overall<br>(N=XX) |
|-------------------------------------------------|-------------------|
| Study Populations [1] | |
| All Enrolled Patients | X (XX.X%) |
| ITT Population | X (XX.X%) |
| Safety Population | X (XX.X%) |
| Per Protocol Population | X (XX.X%) |
| Completion Status [2] | |
| Completed Initial Treatment Period | X (XX.X%) |
| Prematurely Discontinued from Study | X (XX.X%) |
| < <ongoing>&gt;</ongoing> | X (XX.X%) |
| In the Extension Phase | X (XX.X%) |
| Reasons for discontinuation | |
| Lost to Follow-up | X (XX.X%) |
| Protocol Violation | X (XX.X%) |
| Adverse Event | X (XX.X%) |
| Death | X (XX.X%) |
| Patient Withdrew Consent | X (XX.X%) |
| Principal Investigator Decision | X (XX.X%) |
| Study Terminated by Sponsor | X (XX.X%) |
| Treatment Limiting Toxicity (TLT) Event | X (XX.X%) |
| Pregnancy | X (XX.X%) |
| Other | X (XX.X%) |
| Reason for discontinuation from Extension Phase | |
| Reason1 | X (XX.X%) |
| Reason2 | X (XX.X%) |

<sup>[1]</sup> Percentages are based on the number of all patients who signed the Informed Consent form. [2] Percentages are based on the number of patients in the Safety Population. SOURCE: Listing 16.2.1

Programming note: only present 'Ongoing' in Completion Status section if patient is still in active treatment phase.

### Table 14.1.2 Summary of Protocol Deviations Safety Population

| Violation Level COVID-19 Relatedness Deviation Category | Overall<br>(N=X) [1] | Number of Protocol Deviations n (%) |
|---|---|---|
| Total number of protocol deviations reported | < <leave blank="">&gt;</leave> | XXX (100.0%) |
| Important [2] | XXX | XX (XX.X%) |
| Non COVID-19 Deviations | XX | XX (XX.X%) |
| Study Drug Compliance | X | XX (XX.X%) |
| < <list all="" categories="" major="" relevant="">&gt;</list> | X | XX (XX.X%) |
| Important (CS) | XXX | XX (XX.X%) |
| Non COVID-19 Deviations | XX | XX (XX.X%) |
| Study Drug Compliance | X | XX (XX.X%) |
| Procedure/Assessment Not Done/Done Incorrectly | X | XX (XX.X%) |
| < <list all="" categories="" cs="" major="" relevant="">&gt;</list> | x | XX (XX.X%) |
| COVID-19 Deviations | xx | XX (XX.X%) |
| Study Drug Compliance | X | XX (XX.X%) |
| Visit Window | X | XX (XX.X%)<br>XX (XX.X%) |
| Procedure/Assessment Not Done/Done Incorrectly | X | XX (XX.X%) |
| < <list all="" categories="" cs="" major="" relevant="">&gt;</list> | X | XX (XX.X%)<br>XX (XX.X%) |
| NEIST All Televant Major 63 Categories | ^ | XX (XX.X 76) |
| Important (NCS) | XXX | XX (XX.X%) |
| Non COVID-19 Deviations | XX | XX (XX.X%) |
| Informed consent | X | XX (XX.X%) |
| Procedure/Assessment Not Done/Done Incorrectly | X | XX (XX.X%) |
| < <list all="" categories="" major="" ncs="" relevant="">&gt;</list> | X | XX (XX.X%) |
| COVID-19 Deviation | XX | XX (XX.X%) |
| Study Drug Compliance | Χ | XX (XX.X%) |
| Visit Window | X | XX (XX.X%) |
| Procedure/Assessment Not Done/Done Incorrectly | X | XX (XX.X%) |
| < <list all="" categories="" major="" ncs="" relevant="">&gt;</list> | X | xx (xx.x%) |
| Non-Important | XXX | XX (XX.X%) |
| Non COVID-19 Deviations | XX | XX (XX.X%)<br>XX (XX.X%) |
| Informed consent | X | XX (XX.X%) |
| Procedure/Assessment Not Done/Done Incorrectly | X | XX (XX.X%) |
| < <list all="" categories="" minor="" relevant="">&gt;</list> | X | XX (XX.X%) |
| Est an folovant minor odtogorios | ^ | 70(70(.7070) |
| COVID-19 Deviations | XX | XX (XX.X%) |
| Study Drug Compliance | X | XX (XX.X%) |
| Visit Window | X | XX (XX.X%) |
| < <list all="" categories="" minor="" relevant="">&gt;</list> | Χ | XX (XX.X%) |

Abbreviations: CS = Clinically significant, NCS = Not clinically significant.

Note: Percentage are based on the total number of protocol deviations (n) reported in the Safety Population.

Note: N is the number of patient in the Safety Population.

[1] Each patient is counted once per Violation Level and once per COVID-19 Relatedness, with patient being counted once within the Deviation Category, e.g., if patient had a procedure done incorrectly due to COVID-19 and also had a compliance issue due to COVID-19 both of which were classed as Important (CS) events, then the patient would have the following records: 1=Important (CS); 1=COVID-19 Deviations; 1=Study Drug Compliance and 1=Procedure... as patient's entries.

[2] Protocol deviation was not classified as CS or NCS at the time of the datacut.

SOURCE: Listing 16.2.2.2

Programming note: <<Leave blank>> cell in the shells should not be populated. Total number of 'Deviation Categories' present for one subject will not add up to the 'COVID-19 Relatedness', it should be higher as accounts for each individual PD category while relatedness counts the patient once irrespective of now many individual PDs have occurred.

If category is not present in the data, skip outputting to the table (mostly will refer to Important [2] once data is corrected).

Identify COVID deviations using COVID19 variable.

Present in descending count order of PDs, if ties present, sort alphabetically.

## Table 14.1.3 Demographics and Baseline Characteristics Safety Population

| Variable<br>Statistic or Category | Overall<br>(N=XX) |
|---|---|
| Age (years) n Mean (SD) Median Min, Max | XX<br>XX.X (XX.XX)<br>XX.X<br>XX, XX |
| Gender<br>Male<br>Female | X (XX.X%)<br>X (XX.X%) |
| Ethnicity Hispanic or Latino Not Hispanic or Latino | X (XX.X%)<br>X (XX.X%) |
| Race American-Indian or Alaska Native Asian Black or African-American Native Hawaiian or Other Pacific Islander White Other | X (XX.X%) X (XX.X%) X (XX.X%) X (XX.X%) X (XX.X%) X (XX.X%) |
| Height (cm) n Mean (SD) Median Min, Max | XX<br>XX.X (XX.XX)<br>XX.X<br>XX, XX |
| Weight (kg) n Mean (SD) Median Min, Max | XX<br>XX.X(XX.XX)<br>XX.X<br>XX, XX |

Abbreviations: BMI = Body mass index; SD= Standard deviation.

Note: Percentage are based on the number of patients in the Safety Population SOURCE: Listing 16.2.4.1

## Table 14.1.3 Demographics and Baseline Characteristics Safety Population

| Variable<br>Statistic or Category | Overall<br>(N=XX) |
|-----------------------------------|-------------------|
| BMI (kg/m2) | |
| n | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Min, Max | XX, XX |
| Capsule Strength Received | |
| 25 mg | X (XX.X%) |
| 100 mg | X (XX.X%) |

Abbreviations: BMI = Body mass index; SD= Standard deviation.

Note: Percentage are based on the number of patients in the Safety Population.

### Table 14.1.4 Summary of Study Drug Exposure Safety Population

| | Overall |
|-----------------------------------|--------------|
| Drug Exposure | (N=XX) |
| Number of Doses Taken | |
| n | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Min, Max | XX, XX |
| Treatment Duration (Days) [1] | |
| n | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Min, Max | XX, XX |
| Total Study Drug Administerd (mg) | |
| n | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Min, Max | XX, XX |
| Intra Dose Escalation | |
| 50 mg to 100 mg | X (XX.X%) |
| 100 mg to 150 mg | X (XX.X%) |
| 150 mg to 200 mg | X (XX.X%) |
| 200 mg to 300 mg | X (XX.X%) |
| 300 mg to 400 mg | X (XX.X%) |

Note: The data cut off date is used if study medication is ongoing (i.e., missing study medication end date in CRFs). A cut off date of XXMMMYYYY is used to calculate dose duration.
[1] Duration = Date of last dose administered – Date of first dose administered + 1.
SOURCE: Listing 16.2.4.4.1

## Table 14.1.5 Summary of Medical History Safety Population

| System Organ Class<br>Preferred Term | Overall<br>(N=XX) |
|--------------------------------------------|-------------------|
| Patients with at least one Medical History | X (XX.X%) |
| System Organ Class 1 | |
| Preferred Term 1 | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) |
| | X (XX.X%) |
| System Organ Class 2 | , |
| Preferred Term 1 | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) |

Note: Percentages are based on the number of patients in the Safety Population.

Medications coded using WHO-DD B2E version March 2017.

Medications are displayed by descending frequency of System Organ Class (SOC), by Preferred Term (PT) within SOC and then alphabetically. Patients were counted only once for each SOC and PT. SOURCE: Listing 16.2.4.2

Table 14.2.1.1 Summary of AUCs and Mean of AUCs for ANC by Dose Level -  $AUC_{ANC} \ge 600/\mu L$  Threshold Safety Population

| | | | | Dose Levels | | | |
|---|---|---|---|---|---|---|---|
| Visit/<br>Statistics | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) | 300/400 mg<br>(N=XX) |
| Week 5 | , , , | | , | , , | | | |
| Mean (SD)<br>Median<br>Min, Max<br>P-value<br>95% CI | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X<br>X.XXX<br>[XX.X; XX.X] |
| Week 13<br>n<br>Mean (SD)<br>Median<br>Min, Max<br>P-value<br>95% CI | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X<br>X.XXX<br>[XX.X; XX.X] |
| Week 21<br>n<br>Mean (SD)<br>Median<br>Min, Max<br>P-value<br>95% CI | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X<br>X.XXX<br>[XX.X; XX.X] |

Abbreviations: AUC = Area under the plasma concentration; CI = Confidence interval; NE = Not estimable; SD = Standard deviation.

Note: AUC is calculated using the trapezoidal rule with area above the threshold being positive and the area below the threshold being negative. The threshold is defined as 600 /ul for ANC. P-value is obtained from two-sided one sample t-test.

[\*] The summary is based on the mean of AUCs that is, the per-patient average of the AUC<sub>ANC</sub> where patient was treated with at least 300/400mg dose. Missing AUCs are not imputed. For a given patient, if all 3 AUCs are missing then per-patient average is missing.

[#] Extension Visits occur every 6 months from the EOS until the drug becomes commercially available.

SOURCE: Listing 16.2.6.1

Programming Note: P-value and 95% CI are computed only for 300/400mg dose, NOT for each dose level.

For dose 300/400mg: "Mean AUC (cell.hr/uL) for ALC (cell/uL) - Weeks 5, 13, 21 - Dose 300 or 400" and "Mean AUC (cell.hr/uL) for ALC (cell/uL) - Extension Visits - Dose 300 or 400". The first parameter will then be used for "All Visits" section and the 2nd parameter will be used for "Extension Visits" section.

### Table 14.2.1.1 Summary of AUCs and Mean of AUCs for ANC by Dose Level Safety Population

| | | | | Dose Levels | | | |
|---|---|---|---|---|---|---|---|
| Visit/<br>Statistics | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) | 300/400 mg<br>(N=XX) |
| All Visits[*] n Mean (SD) Median Min, Max P-value 95% CI Extension Visits | | | | | | | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X<br>X.XXX<br>[XX.X; XX.X] |
| [#] n Mean (SD) Median Min, Max P-value 95% CI | | | | | | | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X<br>X.XXX<br>[XX.X; XX.X] |

Abbreviations: AUC = Area under the plasma concentration; CI = Confidence interval; NE = Not estimable; SD = Standard deviation.

Note: AUC is calculated using the trapezoidal rule with area above the threshold being positive and the area below the threshold being negative. The threshold is defined as 500 /ul for ANC. P-value is obtained from two-sided one sample t-test.

[\*] The summary is based on the mean of AUCs that is, the per-patient average of the AUC<sub>ANC</sub> where patient was treated with at least 300/400mg dose. Missing AUCs are not imputed. For a given patient, if all 3 AUCs are missing then per-patient average is missing.

[#] Extension Visits occur every 6 months from the EOS until the drug becomes commercially available.

Patient , Extension Phase - Residence Visit 1 Post EOS and Extension Phase - Residence Visit 3 occurred during episodes of infection. These values were excluded from the analysis.

Patient Week 21 occurred during an episode of infection. These values were excluded from the analysis.

SOURCE: Listing 16.2.6.1

Programming Note: P-value and 95% CI are computed only for 300/400mg dose, NOT for each dose level.

# Table 14.2.1.1.1 Summary of AUCs and Mean of AUCs for ANC by Dose Level - AUC $_{ANC} \ge 500/\mu L$ Threshold Safety Population

(Same shell as Table 14.2.1.1. Update footnote to: The threshold is defined as 600 /ul for ANC.)

Table 14.2.1.2

Summary of AUCs and Mean of AUCs for ALC by Dose Level
Safety Population

| | Dose Levels | | | | | | |
|---|---|---|---|---|---|---|---|
| Visit/<br>Statistics | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) | 300/400 mg<br>(N=XX) |
| Week 5 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| P-value | , | , | , | • | , | , | X.XXX |
| 95% CI | | | | | | | [XX.X; XX.X] |
| Week 13 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X(XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | xx.x | xx.x | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| P-value | | | | | | | X.XXX |
| 95% CI | | | | | | | [XX.X; XX.X] |
| Week 21 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | xx.x | xx.x | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| P-value | , | • | • | • | • | , | X.XXX |
| 95% CI | | | | | | | [XX.X; XX.X] |

Abbreviations: AUC = Area under the plasma concentration; CI = Confidence interval; NE = Not estimable; SD = Standard deviation.

Note: AUC is calculated using the trapezoidal rule with area above the threshold being positive and the area below the threshold being negative. The threshold is defined as 1000 /ul for ALC. P-value is obtained from two-sided one sample t-test.

[\*] The summary is based on the mean of AUCs that is, the per-patient average of the AUC<sub>ALC</sub> where patient was treated with at least 300/400mg dose. Missing AUCs are not imputed. For a given patient, if all 3 AUCs are missing then per-patient average is missing.

[#] Extension Visits occur every 6 months from the EOS until the drug becomes commercially available.

Patient , Extension Phase - Residence Visit 1 Post EOS and Extension Phase - Residence Visit 3 occurred during episodes of infection. These values were excluded from the analysis.

Patient Week 21 occurred during an episode of infection. These values were excluded from the analysis.

SOURCE: Listing 16.2.6.1

Programming Note: P-value and 95% CI are computed only for 300/400mg dose, NOT for each dose level.

## Table 14.2.1.2 Summary of AUCs and Mean of AUCs for ALC by Dose Level Safety Population

| | | | | Dose Levels | | | |
|---|---|---|---|---|---|---|---|
| Visit/<br>Statistics | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) | 300/400 mg<br>(N=XX) |
| All Visits[*] n Mean (SD) Median Min, Max P-value 95% CI Extension Visits | | | | | | | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X<br>X.XXX<br>[XX.X; XX.X] |
| [#] n Mean (SD) Median Min, Max P-value 95% CI | | | | | | | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X<br>X.XXX<br>[XX.X; XX.X] |

Abbreviations: AUC = Area under the plasma concentration; CI = Confidence interval; SD = Standard deviation.

Note: AUC is calculated using the trapezoidal rule with area above the threshold being positive and the area below the threshold being negative. The threshold is defined as 1000 /ul for ALC. P-value is obtained from two-sided one sample t-test.

[\*] The summary is based on the mean of AUCs that is, the per-patient average of the AUC<sub>ALC</sub> where patient was treated with at least 300/400mg dose. Missing AUCs are not imputed. For a given patient, if all 3 AUCs are missing then per-patient average is missing.

[#] Extension Visits occur every 6 months from the EOS until the drug becomes commercially available.

Patient , Extension Phase - Residence Visit 1 Post EOS and Extension Phase - Residence Visit 3 occurred during episodes of infection. These values were excluded from the analysis.

Patient Week 21 occurred during an episode of infection. These values were excluded from the analysis.

SOURCE: Listing 16.2.6.1

Programming Note: P-value and 95% CI are computed only for 300/400mg dose, NOT for each dose level.

Table 14.2.2.1 Summary of Infection Rates Safety Population

| | | | Dose | Levels | | | |
|---|---|---|---|---|---|---|---|
| | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) | Overall<br>(N=XX) |
| Rate of Infection by type [1] | | | | | | | |
| Number of events (Rate of | XX (X.XX) | XX (X.XX) | XX (X.XX) | XX (X.XX) | XX (X.XX) | XX (X.XX) | XX (X.XX) |
| Infection) by type 1 / [95% CI] | [X.XX; X.XX] | [X.XX; X.XX] | [X.XX; X.XX] | [X.XX; X.XX] | [X.XX; X.XX] | [X.XX; X.XX] | [X.XX; X.XX] |
| Number of events (Rate of Infection) | XX (X.XX) | XX (X.XX) | XX (X.XX) | XX (X.XX) | XX (X.XX) | XX (X.XX) | XX (X.XX) |
| type 2 / [95% CI] | [X.XX; X.XX] | [X.XX; X.XX] | [X.XX; X.XX] | [X.XX; X.XX] | [X.XX; X.XX] | [X.XX; X.XX] | [X.XX; X.XX] |
| Number of events (Rate of Infection) | XX (X.XX) | XX (X.XX) | XX (X.XX) | XX (X.XX) | XX (X.XX) | XX (X.XX) | XX (X.XX) |
| by type k / [95% CI] | [X.XX; X.XX] | [X.XX; X.XX] | [X.XX; X.XX] | [X.XX; X.XX] | [X.XX; X.XX] | [X.XX; X.XX] | [X.XX; X.XX] |
| Number of events (Rate of All types of | XX (X.XX) | XX (X.XX) | XX (X.XX) | XX (X.XX) | XX (X.XX) | XX (X.XX) | XX (X.XX) |
| Infections) / [95% CI] | [X.XX; X.XX] | [X.XX; X.XX] | [X.XX; X.XX] | [X.XX; X.XX] | [X.XX; X.XX] | [X.XX; X.XX] | [X.XX; X.XX] |

Note: XX (X.XX) [X.XX; X.XX] syntax refers to the number of infections – XX, followed by the infection rate (X.XX) and 95% CI [X.XX; X.XX].

Note: Percentages are based on number of patients in the Safety Population. Two-sided 95% CI is computed using the Normal approximation of the Negative Binomial Distribution. [1] Rate of infection, per year, is defined as the total number of infections divided by the total number of person-years.

Table 14.2.2.2 Summary of Infections by Severity Safety Population

| | | | Dose | Levels | | | _ |
|---|---|---|---|---|---|---|---|
| Infections/<br>Grade [1] | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) | Overall (N=XX) |
| Patients with at least one Infection | , , , | | | | | , , , | |
| Grade 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | V (VV V0/.) |
| | ` , | ` , | , | ` , | ` , | ` , | X (XX.X%) |
| Grade 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Grade 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Grade 4 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Grade 5 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Infection 1 | | | | | | | |
| Grade 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Grade 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Grade 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Grade 4 | X (XX.X%) | X (XX.X%) | X (XX.X%) | x (xx.x%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Grade 5 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Infection 2 | | | | | | | |
| Grade 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Grade 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Grade 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Grade 4 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Grade 5 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Grade 5 | A (AA.A /0) | A (AA.A 70) | A (AA.A 70) | Λ (ΛΛ.Λ /0) | A (AA.A /0) | A (AA.A 70) | A (AA.A 70) |

Note: XX (X.XX) syntax refers to the number of infections – XX, followed by the infection rate (X.XX).

Note: Percentages are based on number of patients in the Safety Population. Two-sided 95% CI is computed using the Normal approximation of the Negative Binomial Distribution.

[1] The severity is assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (v4.03).

### Table 14.2.2.3 Summary of Highest Grade Infections Safety Population

| Infections/<br>Grade [1] | Dose Levels | | | | | |
|---|---|---|---|---|---|---|
| | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) |
| Patients with at least one Infection | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| nfection 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| nfection 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Note: Percentages are based on number of patients in the Safety Population.

Note: This table summarizes only infections which meet the highest severity grade criteria at the given dose level for each patient. An infection is considered to have met the criteria if the severity of infection is same as the maximum severity grade experienced by the patient at the given dose level. [1] The severity is assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (v4.03).

### Table 14.2.2.4 Summary of Infection Scores Safety Population

| | X4P-001 | X4P-001 | X4P-001 | X4P-001 | X4P-001 |
|---|---|---|---|---|---|
| | 50/100/150 mg | 200 mg | 300 mg | 400 mg | 300/400 mg |
| Statistics | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Overall Infection Score [1] | | | | | |
| Number of Infection Events | XX | XX | XX | XX | XX |
| Mean (SD) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) |
| Standard Error | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min, Max | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| 95% CI | (XX.XX,XX.XX) | (XX.XX,XX.XX) | (XX.XX,XX.XX) | (XX.XX,XX.XX) | (XX.XX,XX.XX) |

Note: Percentages are based on number of patients in the Safety Population. Two-sided 95% CI is computed using the Normal Distribution.

Note: n is the number of patients who had an infection whilst on the reported dose of the study drug.

[1] Infection Score = (# of infection events × severity) / duration of exposure in years. SOURCE: Listings 16.2.7.1 and 16.2.7.3

Programming note: use OINFSC from ADIR dataset. n is the number of patients who had an event while on IMP dose at the time.

Table 14.2.3.1 Summary of Non-Genital Warts Safety Population

| | Dose Levels | | | | | | |
|---|---|---|---|---|---|---|---|
| Study Week/<br>Statistic | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) | Overall<br>(N=XX) |
| Baseline [1] | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Week 5 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| CFB to Week 5 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Week 13 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median <sup>′</sup> | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| CFB to Week 13 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median <sup>′</sup> | xx.x | XX.X | xx.x | XX.X | XX.X | XX.X | xx.x |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |

Note: An out of schedule assessment of warts was done at end of study visit for subject SOURCE: Listing 16.2.4.5.

> Confidential Page 59 of 172

Abbreviations: CFB = Change from Baseline; NE = Not estimable; SD = Standard deviation.
[1] Baseline is the last non-missing observation recorded before the first dose on Day 1. Baseline visit is displayed for all dose levels irrespective of whether they were receiving that dose level at baseline.

### Table 14.2.3.1 Summary of Non-Genital Warts Safety Population

| Dose Levels | | | | | | |
|---|---|---|---|---|---|---|
| 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) | Overall (N=XX) |
| XX | XX | XX | XX | XX | XX | XX |
| XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| XX | XX | XX | XX | XX | XX | XX |
| XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| xx.x | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | | | | | | XX |
| | | | | | | XX.X (XX.XX) |
| | | | | | | XX.X |
| | | | | | | XX.X, XX.X |
| | | | | | | XX |
| | | | | | | XX.X (XX.XX) |
| | | | | | | XX.X |
| | | | | | | XX.X, XX.X |
| | (N=XX) XX XX.X (XX.XX) XX.X XX.X, XX.X XX XX.X (XX.XX) XX.X (XX.XX) | (N=XX) | 50 mg (N=XX) 100 mg (N=XX) 150 mg (N=XX) XX XX XX XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X XX.X XX.X XX.X XX.X XX.X XX XX XX XX XX XX XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) | 50 mg (N=XX) 100 mg (N=XX) 150 mg (N=XX) 200 mg (N=XX) XX XX XX XX XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX XX XX XX XX XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) | 50 mg (N=XX) 100 mg (N=XX) 150 mg (N=XX) 200 mg (N=XX) 300 mg (N=XX) XX XX XX XX XX XX XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX XX XX XX.X (XX.XX) XX.X (XX.XX) | 50 mg (N=XX) 100 mg (N=XX) 150 mg (N=XX) 200 mg (N=XX) 300 mg (N=XX) 400 mg (N=XX) XX XX XX XX XX XX XX XX.X (XX.XX) XX.X (XX.X |

Note: An out of schedule assessment of warts was done at end of study visit for subject SOURCE: Listing 16.2.4.5



Abbreviations: CFB = Change from Baseline; NE = Not estimable; SD = Standard deviation.
[1] Baseline is the last non-missing observation recorded before the first dose on Day 1. Baseline visit is displayed for all dose levels irrespective of whether they were receiving that dose level at baseline.

### Table 14.2.3.2 Summary of Non-Genital Warts by location Safety Population

Location: XXXXXX

| | | | Dose | Levels | | | |
|---|---|---|---|---|---|---|---|
| Study Week/<br>Statistic | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) | Overall<br>(N=XX) |
| Baseline [1] | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median ´ | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Week 5 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| CFB to Week 5 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Week 13 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| CFB to Week 13 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |

Abbreviations: CFB = Change from Baseline; NE = Not estimable; SD = Standard deviation.

Note: An out of schedule assessment of warts was done at end of study visit for subject SOURCE: Listing 16.2.4.5.

<sup>[1]</sup> Baseline is the last non-missing observation recorded before the first dose on Day 1. Baseline visit is displayed for all dose levels irrespective of whether they were receiving that dose level at baseline.

## Table 14.2.3.2 Summary of Non-Genital Warts by location Safety Population

Location: XXXXXX

| | | | Dose L | evels | | | |
|---|---|---|---|---|---|---|---|
| Study Week/<br>Statistic | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) | Overall (N=XX) |
| Week 21 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| CFB to Week 21 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median ´ | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Extension Visits | | | | | | | |
| n | | | | | | | XX |
| Mean (SD) | | | | | | | XX.X (XX.XX) |
| Median ´ | | | | | | | XX.X |
| Min, Max | | | | | | | XX.X, XX.X |
| CFB to Extension visits | | | | | | | |
| n | | | | | | | XX |
| Mean (SD) | | | | | | | XX.X (XX.XX) |
| Median | | | | | | | XX.X |
| Min, Max | | | | | | | XX.X, XX.X |
| , | | | | | | | , / 0 11/1 |

Abbreviations: CFB = Change from Baseline; NE = Not estimable; SD = Standard deviation.
[1] Baseline is the last non-missing observation recorded before the first dose on Day 1. Baseline visit is displayed for all dose levels irrespective of whether they were receiving that dose level at baseline.

Note: An out of schedule assessment of warts was done at end of study visit for subject

### Table 14.2.4.1 Summary of Genital Warts Safety Population

(Same shell as Table 14.2.3: SOURCE: Listing 16.2.4.5)

### Table 14.2.5 Summary of Antibody Levels following Revaccination Safety Population

Antibodies: Haemophilus Influenzae B Polysaccharide (mg/L)

| | | | Dose L | evels | | | |
|---|---|---|---|---|---|---|---|
| Study Week /<br>Statistics | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) | Overall<br>(N=XX) |
| Baseline [1] | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX |
| Median | xx.x | xx.x | xx.x | xx.x | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Week 9 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | xx.x | xx.x | xx.x | xx.x | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| CFB to Week 9 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX |
| Median | xx.x | xx.x | xx.x | xx.x | XX.X | XX.X | xx.x |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Week 17 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| CFB to Week 17 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX |
| Median | xx.x | xx.x | xx.x | xx.x | XX.X | XX.X | xxx.x |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Week 25 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |

Abbreviations: CFB = Change from Baseline; NE = Not estimable; SD = Standard deviation.

<sup>[1]</sup> Baseline is the last non-missing observation recorded on or before treatment start date. Baseline visit is displayed for all dose levels irrespective of whether they were receiving that dose level at baseline.

## Table 14.2.5 Summary of Antibody Levels following Revaccination Safety Population

Antibodies: <<pre><<pre><<pre>

| | | | Dose L | evels | | | |
|---|---|---|---|---|---|---|---|
| Study Week /<br>Statistics | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) | Overall<br>(N=XX) |
| CFB to Week 25 | | | | | | | |
| n<br>Mean (SD)<br>Median<br>Min, Max | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, XX.X |
| Extension Visits | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD)<br>Median | XX.X (XX.XX)<br>XX.X | XX.X (XX.XX)<br>XX.X | XX.X (XX.XX)<br>XX.X | XX.X (XX.XX)<br>XX.X | XX.X (XX.XX)<br>XX.X | XX.X (XX.XX)<br>XX.X | XX.X (XX.XX)<br>XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| CFB to Extension Visits | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median <sup>′</sup> | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |

Abbreviations: CFB = Change from Baseline; NE = Not estimable; SD = Standard deviation.

<sup>[1]</sup> Baseline is the last non-missing observation recorded on or before treatment start date. Baseline visit is displayed for all dose levels irrespective of whether they were receiving that dose level at baseline. SOURCE: Listing 16.2.4.6

Table 14.2.6 Summary of Rescue Medications Safety Population

| | Dose Levels | | | | | | |
|---|---|---|---|---|---|---|---|
| ATC Class Level 4 Preferred Term (ATC Class Level 5) | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) | Overall (N=XX) |
| · | | | | | | | • |
| Patients with at least one Rescue Medication | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| ATC Class 1 | | | | | | | |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| ATC Class 2 | , | , | , , | , | , | , , | , |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | x (xx.x%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | x (xx.x%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | X (XX.X%) |

Note: Percentages are based on the number of patients in the Safety Population.

Medications coded using WHO-DD B2E version March 2017.

Medications are displayed by descending frequency of Anatomic Therapeutic Chemical (ATC) Level 4 classification, by Preferred Term (PT) within ATC and then alphabetically. Patients were counted only once for each ATC and PT.

Table 14.2.7 Summary of Hospitalizations Safety Population

| | | | Dose | Levels | | | |
|---|---|---|---|---|---|---|---|
| Hospitalization | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) | Overall<br>(N=XX) |
| Hospitalized | | | | | | | |
| Yes | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| No | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Hospitalized WHIM Related | | | | | | | |
| Yes | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| No | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Hospitalized AE Related | | | | | | | |
| Yes | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| No | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Total Number of hospitalizations | | | | | | | |
| n · | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Duration of hospitalization (in Days) | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |

Abbreviations: AE = Adverse event; NE = Not estimable; SD = Standard deviation. Note: Percentages are based on the number of patients in the Safety Population. SOURCE: Listing 16.2.7.1, 16.2.7.3

Table 14.2.8 Summary of Ig and Specified Antibodies Safety Population

Antibody: XXXXXXX

| | | | | Levels | | | |
|---|---|---|---|---|---|---|---|
| Study Week/<br>Statistics | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) | Overall<br>(N=XX) |
| Baseline | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Veek 2 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| CFB to Week 2 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Veek 3 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| CFB to Week 3 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Veek 25 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XXX |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |

Abbreviations: CFB Change from Baseline; NE = Not estimable; SD = Standard deviation. Note: Change is calculated as post baseline - baseline.

<sup>[1]</sup> Baseline is the last non-missing observation recorded before the first dose on Day 1. Baseline visit is displayed for all dose levels irrespective of whether they were receiving that dose level at baseline.

### Table 14.2.8 Summary of Ig and Specified Antibodies Safety Population

Antibody: XXXXXXX

| | | | Dose | Levels | | | |
|---|---|---|---|---|---|---|---|
| Study Week/ | 50 mg | 100 mg | 150 mg | 200 mg | 300 mg | 400 mg | Overall |
| Statistics | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| CFB to Week 25 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Extension Visits | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median <sup>′</sup> | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| CFB to Extension Visits | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |

Abbreviations: CFB Change from Baseline; NE = Not estimable; SD = Standard deviation.

Note: Change is calculated as post baseline - baseline.

<sup>[1]</sup> Baseline is the last non-missing observation recorded before the first dose on Day 1. Baseline visit is displayed for all dose levels irrespective of whether they were receiving that dose level at baseline.

# Table 14.2.9 Time above Threshold (Hours) for ANC by Dose Level Safety Population

| | X4P-001 | X4P-001 | X4P-001 | X4P-001 | X4P-001 |
|---|---|---|---|---|---|
| | 50/100/150 mg | 200 mg | 300 mg | 400 mg | 300/400 mg |
| Statistics | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Number of Subjects | XX | XX | XX | XX | XX |
| Mean (SD) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX |
| Standard Error | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min, Max | XX.X.XX.X | XX.X,XX.X | XX.X.XX.X | XX.X,XX.X | XX.X,XX.X |

Abbreviation: SD = Standard deviation.

Note: Time above threshold is defined as total time a subjects ANC result was above 500/uL. If time above threshold was >24 hours, it was rounded off to 24. Baseline observation carried forward (BOCF) imputation was used if a subjects 24 hour assessment was missing. Imputation is not used for intermediate missing assessments.

Patient , Extension Phase - Residence Visit 1 Post EOS and Extension Phase - Residence Visit 3 occurred during episodes of infection. These values were excluded from the analysis.

Patient Week 21 occurred during an episode of infection. These values were excluded from the analysis.

Dense sample data for subject will be excluded from the TAT summary tables and figures since the WBC, ANC, ALC, and AMC levels were normal at screening.

SOURCE: Listing 16.2.6.2.3

Table 14.2.9.1
Time above Threshold (Hours) for ANC by Dose Level – Sensitivity Analysis
Safety Population

(Same shell as Table 14.2.9: SOURCE: Listing 16.2.6.2.3. Do not display the footnote 'Dense sample data for subject will be excluded from the TAT summary tables and figures since the WBC, ANC, ALC, and AMC levels were normal at screening.')

Table 14.2.10
Time above Threshold (Hours) for ALC by Dose Level
Safety Population

(Same shell as Table 14.2.9: SOURCE: Listing 16.2.6.2.3)

Programming Note: Use ALC instead of ANC in the footnote and use threshold as 1000/uL.

# Table 14.2.10.1 Time above Threshold (Hours) for ALC by Dose Level – Sensitivity Analysis Safety Population

(Same shell as Table 14.2.9: SOURCE: Listing 16.2.6.2.3 Do not display the footnote. 'Dense sample data for subject will be excluded from the TAT summary tables and figures since the WBC, ANC, ALC, and AMC levels were normal at screening.')

# Table 14.2.11 Time above Threshold (Hours) for AMC by Dose Level Safety Population

(Same shell as Table 14.2.9: SOURCE: Listing 16.2.6.2.3)

Programming Note: Use AMC instead of ANC in the footnote and use threshold and categorize by age ranges; 12-18yrs and >=18yrs, and gender; Male and Female as follows:

| Age (year) | Gender | Threshold (/uL) |
|------------|--------|-----------------|
| 12-18 | F | 190 |
| | М | 180 |
| >=18 | F | 250 |
| | М | 290 |

#### Add footnote:

Note: Time above threshold is defined as total time a subject's AMC result was above 190/uL for females aged 12 to 18, above 180/uL for males aged

12 to 18, above 250/uL for females aged>=18 and above 290/uL for males aged >=18. If time above threshold was >24 hours, it was rounded off to 24. Baseline observation carried fo rward (BOCF) imputation was used if a subject's 24 hour assessment was missing. Imputation is not used for intermediate missing assessments.

Patient , Extension Phase - Residence Visit 1 Post EOS and Extension Phase - Residence Visit 3 occurred during episodes of infection. These values were excluded from the analysis.

Patient , Week 21 occurred during an episode of infection. These values were excluded from the analysis.

Dense sample data for subject will be excluded from the TAT summary tables and figures since the WBC, ANC, ALC, and AMC levels were normal at screening.

SOURCE: Listing 16.2.6.2.3

# Table 14.2.11.1 Time above Threshold (Hours) for AMC by Dose Level – Sensitivity Analysis Safety Population

(Same shell as Table 14.2.11: SOURCE: Listing 16.2.6.2.3. Do not display the footnote 'Dense sample data for subject will be excluded from the TAT summary tables and figures since the WBC, ANC, ALC, and AMC levels were normal at screening.')

Table 14.3.1.1 Overall Summary of Treatment-Emergent Adverse Events Safety Population

| | | | | Dose Lev | /els | | | |
|---|---|---|---|---|---|---|---|---|
| Treatment-Emergent Adverse Events | 50 mg<br>(N=XX) | | 100 mg<br>(N=XX) | | 150 mg<br>(N=XX) | | 200 mg<br>(N=XX) | |
| | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] |
| Patients with at least one TEAE | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Total Number of Events | XX | XX | XX | XX | XX | XX | XX | XX |
| TEAE by Relationship [2]<br>Unrelated<br>Related | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) |
| AE leading to Discontinuation from study | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| SAE | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| AE leading to Death | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Abbreviations: AE = Adverse event; SAE = Serious AE; TEAE = Treatment emergent adverse event.

Note: Percentages are based on the number of patients in the Safety Population. TEAEs were coded using MedDRA version 23.1.

A TEAE is defined as any AE that begins or worsens in severity or frequency on or after the start of study drug through 10 days after the last dose of the study drug.

[1] The severity is assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCÁE) (v4.03). "All Grades" includes all TEAEs with CTCAE Grade 1 to 5, "≥ Grade 3" is a subset of "All Grades" reported.

[2] Unrelated TEAEs are those marked as not related on the case report form (CRF); Related TEAEs are those marked as possibly related or related on the CRF.
Table 14.3.1.1

Overall Summary of Treatment-Emergent Adverse Events
Safety Population

| | Dose Levels | | | | | |
|---|---|---|---|---|---|---|
| Treatment-Emergent Adverse Events | | 0 mg<br>=XX) | | ) mg<br>=XX) | Ove<br>(N= | |
| - | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] |
| Patients with at least one TEAE | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Total Number of Events | XX | XX | XX | XX | XX | XX |
| TEAE by Relationship [2] | | | | | | |
| Unrelated | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Related | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| AE leading to Discontinuation from study | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| SAE | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| AE leading to Death | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Abbreviations: AE = Adverse event; SAE = Serious AE; TEAE = Treatment emergent adverse event.

Note: Percentages are based on the number of patients in the Safety Population. TEAEs were coded using MedDRA version 23.1.

A TEAE is defined as any AE that begins or worsens in severity or frequency on or after the start of study drug through 10 days after the last dose of the study drug.

<sup>[1]</sup> The severity is assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (v4.03). "All Grades" includes all TEAEs with CTCAE Grade 1 to 5, "> Grade 3" is a subset of "All Grades" reported.

<sup>[2]</sup> Unrelated TEAEs are those marked as not related on the case report form (CRF); Related TEAEs are those marked as possibly related or related on the CRF. SOURCE: Listing 16.2.7.1

Table 14.3.1.2
Summary of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Safety Population

| | | | | Dose Lev | /els | | | |
|---|---|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | 50 mg<br>(N=XX) | | 100 mg<br>(N=XX) | | 150<br>(N= | 9 | 200 mg<br>(N=XX) | |
| | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] |
| Patients with at least One TEAE | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| System Organ Class 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | x (xx.x%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| System Organ Class 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Note: Percentages are based on the number of patients in the Safety Population. TEAEs were coded using MedDRA version 23.1.

A TEAE is defined as any AE that begins or worsens in severity or frequency on or after the start of study drug through 10 days after the last dose of the study drug.

[1] The severity is assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (v4.03).

Table 14.3.1.2
Summary of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Safety Population

| | Dose Levels | | | | | |
|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | 300 mg<br>(N=XX) | | | mg<br>XX) | Overall<br>(N=XX) | |
| | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] |
| Patients with at least One TEAE | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| System Organ Class 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| System Organ Class 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Note: Percentages are based on the number of patients in the Safety Population. TEAEs were coded using MedDRA version 23.1.

A TEAE is defined as any AE that begins or worsens in severity or frequency on or after the start of study drug though 10 days after the last dose of the study drug.

[1] The severity is assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (v4.03).

Table 14.3.1.3 Summary of Treatment-Emergent Adverse Events Related to Study Treatment by System Organ Class and Preferred Term Safety Population

| TEAEs Related to Study Drug** | | Dose Levels | | | | | | |
|---|---|---|---|---|---|---|---|---|
| System Organ Class | 50 mg | | 100 mg | | 150 mg | | 200 mg | |
| Preferred Term | (N= | XX) | (N= | :XX) | (N= | XX) | (N= | XX) |
| | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] |
| Patients with at least One TEAE | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| System Organ Class 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | x (xx.x%) | X (XX.X%) | X (XX.X%) |
| System Organ Class 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Note: Percentages are based on the number of patients in the Safety Population. TEAEs were coded using MedDRA version 23.1.

A TEAE is defined as any AE that begins or worsens in severity or frequency on or after the start of study drug through 10 days after the last dose of the study drug. [1] The severity is assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (v4.03).

<sup>\*\*</sup>A related TEAE is one that is marked as possibly related, probably related, or definitely related as assessed by the Investigator.

Table 14.3.1.3

Summary of Treatment-Emergent Adverse Events Related to Study Treatment by System Organ Class and Preferred Term Safety Population

| TEAEs Related to Study Drug** | | | Dose L | evels | | |
|---|---|---|---|---|---|---|
| System Organ Class | 300 | ) mg | 400 | mg | Overall | |
| Preferred Term | (N= | =XX) | (N= | XX) | (N=) | XX) |
| | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] |
| Patients with at least One TEAE Related to | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Study Drug | , , | , , | , , | , | , , | , , |
| System Organ Class 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| System Organ Class 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Note: Percentages are based on the number of patients in the Safety Population. TEAEs were coded using MedDRA version 23.1.

A TEAE is defined as any AE that begins or worsens in severity or frequency on or after the start of study drug though 10 days after the last dose of the study drug.

<sup>[1]</sup> The severity is assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (v4.03).

<sup>\*\*</sup> A related TEAE is one that is marked as possibly related, probably related, or definitely related as assessed by the Investigator.

Table 14.3.2.1 Summary of Serious Adverse Events by System Organ Class and Preferred Term Safety Population

| | Dose Levels | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | 50 mg<br>(N=XX) | | 100 mg<br>(N=XX) | | 150<br>(N= | 3 | 200 mg<br>(N=XX) | |
| | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] |
| Patients with at least One SAE | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| System Organ Class 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| System Organ Class 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Abbreviations: SAE = Serious adverse event.

Note: Percentages are based on the number of patients in the Safety Population. SAEs were coded using MedDRA version 23.1.
[1] The severity is assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (v4.03).

Table 14.3.2.1 Summary of Serious Adverse Events by System Organ Class and Preferred Term Safety Population

| | | | Dose L | evels | | |
|---|---|---|---|---|---|---|
| System Organ Class | 300 mg | | 400 | mg | Ove | rall |
| Preferred Term | (N= | =XX) | (N= | XX) | (N=) | XX) |
| | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] |
| Patients with at least One SAE | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| System Organ Class 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| System Organ Class 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | x (xx.x%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Abbreviations: SAE = Serious adverse event.

Note: Percentages are based on the number of patients in the Safety Population. SAEs were coded using MedDRA version 23.1.
[1] The severity is assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (v4.03). SOURCE: Listing 16.2.7.1

Table 14.3.2.2 Summary of Serious Adverse Events Related to Study Treatment by System Organ Class and Preferred Term Safety Population

| SAEs Related to Study Drug** | | | | Dose Lev | /els | | | |
|---|---|---|---|---|---|---|---|---|
| System Organ Class Preferred Term | | mg<br>:XX) | | 100 mg<br>(N=XX) | | 150 mg<br>(N=XX) | | mg<br>XX) |
| Troiding Tollin | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] |
| Patients with at least One SAE | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| System Organ Class 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 1 Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| System Organ Class 2 Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Abbreviation: SAE = Serious adverse event.

Note: Percentages are based on the number of patients in the Safety Population. SAEs were coded using MedDRA version 23.1.

<sup>[1]</sup> The severity is assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (v4.03).

\*\* A related SAE is one that is possibly related, probably related, or definitely related as assessed by the Investigator.

# Table 14.3.2.2 Summary of Serious Adverse Events Related to Study Treatment by System Organ Class and Preferred Term Safety Population

| SAEs Related to Study Drug** | | | Dose L | Dose Levels | | |
|---|---|---|---|---|---|---|
| System Organ Class | 300 | ) mg | 400 | mg | Overall | |
| Preferred Term | (N= | =XX) | (N= | XX) | (N=) | XX) |
| | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] | All Grades[1] | ≥ Grade 3[1] |
| Patients with at least One SAE | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| System Organ Class 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| System Organ Class 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | x (xx.x%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | x (xx.x%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Abbreviation: SAE = Serious adverse event.

Note: Percentages are based on the number of patients in the Safety Population.

SAEs were coded using MedDRA version 23.1.

<sup>[1]</sup> The severity is assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (v4.03).

<sup>\*\*</sup> A related SAE is one that is possibly related, probably related, or definitely related as assessed by the Investigator.

Table 14.3.2.3 Summary of Treatment-Limiting Toxicities by System Organ Class and Preferred Term Safety Population

| | Dose Levels | | | | | | |
|---|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) | Overall<br>(N=XX) |
| Patients with at least One TLT TEAE | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| System Organ Class 1 | | | | | | | |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| System Organ Class 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Abbreviations: TLT = Treatment-limiting toxicity; TEAE = Treatment emergent adverse event.

Note: Percentages are based on the number of patients in the Safety Population.TEAEs were coded using MedDRA version 23.1.

A TEAE is defined as any AE that begins or worsens in severity or frequency on or after the start of study drug through 10 days after the last dose of the study drug.

Table 14.3.2.4
Summary of Grade 3 or Higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Safety Population

| | | | Dose | Levels | | | |
|---|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) | Overall<br>(N=XX) |
| Patients with at least One Grade 3 or Higher TEAE | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| System Organ Class 1 | | | | | | | |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| System Organ Class 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | x (xx.x%) | x (xx.x%) | X (XX.X%) | x (xx.x%) | x (xx.x%) | X (XX.X%) | X (XX.X%) |

Abbreviation: TEAE = Treatment emergent adverse event.

Note: Percentages are based on the number of patients in the Safety Population. N under each dose level represents patients who got drug at that dose level. TEAEs were coded using MedDRA version 23.1.

A TEAE is defined as any AE that begins or worsens in severity or frequency on or after the start of study drug through 10 days after the last dose of study drug.

Table 14.3.2.5
Rate of Treatment Emergent Adverse Events by System Organ Class and Preferred Term Safety Population

| | | | Dose | Levels | | | |
|---|---|---|---|---|---|---|---|
| System Organ Class | 50 mg | 100 mg | 150 mg | 200 mg | 300 mg | 400 mg | Overall |
| Preferred Term | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Patients with at least One TEAE | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| System Organ Class 1 | | | | | | | |
| Preferred Term 1 | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) |
| | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] |
| Preferred Term 2 | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) |
| | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] |
| Preferred Term 3 | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) |
| | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] |
| System Organ Class 2 | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) |
| | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] |
| Preferred Term 1 | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) |
| | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] |
| Preferred Term 2 | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) |
| | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] |
| Preferred Term 3 | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) |
| | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] | [X.XX, X.XX] |

Abbreviation: AE = Adverse event; CI = Confidence interval; TEAE = Treatment emergent adverse event.

Note: XX (X.XX) [X.XX; X.XX] syntax refers to the number of TEAEs – XX, followed by the TEAE rate (X.XX) and 95% CI [X.XX; X.XX].

Percentages are based on the number of patients in the Safety Population. TEAEs were coded using MedDRA version 23.1.

A TEAE is defined as any AE that begins or worsens in severity or frequency on or after the start of study drug through 10 days after the last dose of study drug.

TEAE rate is the total number of TEAEs at that dose, divided by the total time (in years) all patients were treated at that dose. Two-sided 95% CI is computed using the Negative Binomial Distribution.

### Table 14.3.2.6.1 Summary of Yearly Infection Rate for Subjects on 300mg and 400mg Dose Levels by 6 Month Intervals Safety Population

| | X4P-001 |
|-------------------------------------------|----------------|
| Period | 300/400 mg |
| Rate Statistics | (N=XX) |
| Pre-Study (12 months prior to first dose) | |
| Number of Infection Events | XX |
| Mean (SD) | XX.XX (XX.XXX) |
| Standard Error | XX.XX |
| | XX.XX |
| Median | |
| Min, Max | XX.X, XX.X |
| 95% CI | (XX.XX, XX.XX) |
| 0-6 Months | |
| Number of Infection Events | XX |
| Mean (SD) | XX.XX (XX.XXX) |
| Standard Error | XX.XX |
| Median | XX.XX |
| Min, Max | XX.X, XX.X |
| 95% CI | (XX.XX, XX.XX) |

Abbreviation: CI = Confidence interval; NE = Not estimable; SD = Standard deviation.

Notes: Infections are identified as follows: for Prior 12 months, events are identified from the Medical History CRF under History of WHIM infections. While on study, infections are identified as all events with a MedDRA System Organ Class of "Infections and infestations". The reporting period starts on the 300 mg dose date. Rate is defined as number of infection events in a given period/duration of period in years. 95% CI is based on normal approximation. Only events with start date occurring within start and end dates of 300/400 mg dose for each subject are included. Time period assignment is based on the start date of the event.

SOURCE: Listing 16.2.7.6

Programming Note: Complete table until maximum duration in 6 month intervals
For Pre-study infection rate use ADIR.PARAMCD=PINFRATE
For 0-6 months, ADIR.PARAMCD=OINFRTBP and DOSEA in (300,400) and ETINFG1=0 – 6 Months.
For 6-12 months, ADIR.PARAMCD=OINFRTBP and DOSEA in (300,400) and ETINFG1=6 – 12 Months
Continue for all available data....

For 0-6 months, for Number of infection events- ADIR.NOINFBP and DOSEA in (300,400) and ETINFG1=0 – 6 Months. For 6-12 months, for Number of infection events- ADIR.NOINFBP and DOSEA in (300,400) and ETINFG1=6 – 12 Months Continue for all available data ....

### Table 14.3.2.6.2 Summary of Yearly Infection Score for Subjects on 300mg and 400mg Dose Levels by 6 Month Intervals Safety Population

| Period | X4P-001 |
|--------------------------------|----------------|
| Infection Score Statistics [1] | 300/400 mg |
| | (N=XX) |
| 0-6 Months | |
| Number of Infection Events | XX |
| Mean (SD) | XX.XX (XX.XXX) |
| Standard Error | xx.xx ′ |
| Median | XX.XX |
| Min, Max | XX.X, XX.X |
| 95% CI | (XX.XX, XX.XX) |
| 6-12 Months | |
| Number of Infection Events | XX |
| Mean (SD) | XX.XX (XX.XXX) |
| Standard Error | XX.XX |
| Median | XX.XX |
| Min, Max | XX.X, XX.X |
| 95% CI | (XX.XX, XX.XX) |

Abbreviation: CI = Confidence interval; NE = Not estimable; SD = Standard deviation.

Notes: Infections are identified as follows: On study infections are identified as all events with a MedDRA System Organ Class of "Infections and infestations". The reporting period starts on the 300 mg dose date. Only events with start date occurring within start and end dates of 300/400 mg dose for each patient are included. Time period assignment is based on the start date of the event.

[1] Infection Score = (# of infection events × severity) / duration of period in years.

SOURCE: Listing 16.2.7.6

Programming Note: Exposure in years is constant in this table, at 6 month intervals, so exposure is always 0.5.

For number of infection events, use PARAMCD=NOINFBP

Complete table until maximum duration in 6 month intervals up to last available interval

For 0-6 months Infection Score, ADIR.PARAMCD=OINFSCBP and DOSEA in (300,400) and ETINFG1=0-6 Months.

For 6-12 months Infection Score, ADIR.PARAMCD= OINFSCBP and DOSEA in (300,400) and ETINFG1=6-12 Months

Continue for all available data ....

Table 14.3.2.7.1 Summary of Yearly Infection Rate by Dose Level – Method 1 Safety Population

| Rate<br>Statistics | 12 Months<br>Prior to<br>First Dose<br>(N=XX) | X4P-001<br>50 mg<br>(N=XX) | X4P-001<br>100 mg<br>(N=XX) | X4P-001<br>150 mg<br>(N=XX) | X4P-001<br>50/100/150 mg<br>(N=XX) | X4P-001<br>200 mg<br>(N=XX) | X4P-001<br>300 mg<br>(N=XX) | X4P-001<br>400 mg<br>(N=XX) | X4P-001<br>300/400 mg<br>(N=XX) |
|---|---|---|---|---|---|---|---|---|---|
| Number of<br>Infection | XX | xx | xx | XX | xx | XX | XX | XX | XX |
| Events | V0/ V0/ | V// V// | V0/ V0/ | VO/ VO/ | V0/ V0/ | V// V// | V0/ V0/ | \0/\0/ | V0/ V0/ |
| Mean (SD) | XX.XX<br>(XX.XXX) | XX.XX<br>(XX.XXX) | XX.XX<br>(XX.XXX) | XX.XX<br>(XX.XXX) | XX.XX<br>(XX.XXX) | XX.XX<br>(XX.XXX) | XX.XX<br>(XX.XXX) | XX.XX<br>(XX.XXX) | XX.XX<br>(XX.XXX) |
| Standard<br>Error | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median<br>Min, Max<br>95% CI | XX.XX<br>XX.X,XX.X<br>(XX.XX,XX.XX) | XX.XX<br>XX.X,XX.X<br>(XX.XX,XX.XX) | XX.XX<br>XX.X,XX.X<br>(XX.XX,XX.XX) | XX.XX<br>XX.X,XX.X<br>(XX.XX,XX.XX) | XX.XX<br>XX.X,XX.X<br>(XX.XX,XX.XX) | XX.XX<br>XX.X,XX.X<br>(XX.XX,XX.XX) | XX.XX<br>XX.X,XX.X<br>(XX.XX,XX.XX) | XX.XX<br>XX.X,XX.X<br>(XX.XX,XX.XX) | XX.XX<br>XX.X,XX.X<br>(XX.XX,XX.XX |

Abbreviations: CI = Confidence interval; NE = Not estimable; SD = Standard deviation.

Notes: On study infections are identified as all events with a MedDRA System Organ Class of "Infections and infestations". Infection rate is calculated as the total number of infection events for all patients within each dose level ÷ total duration of exposure (in years) for all patient within each dose level. 95% Cl and Standard Error are based on Poisson approximation for each dose level. Events at dose level are assigned based on the start date of the event occurring within start and end dates of that dose for each subject. SOURCE: Listing 16.2.7.7

Programming Note: For Rate use ADIR.PARAMCD=OINFRAT1.

Table 14.3.2.7.2 Summary of Yearly Infection Rate by Dose Level – Method 2 Safety Population

| Rate<br>Statistics | 12 Months<br>Prior to<br>First Dose<br>(N=XX) | X4P-001<br>50 mg<br>(N=XX) | X4P-001<br>100 mg<br>(N=XX) | X4P-001<br>150 mg<br>(N=XX) | X4P-001<br>50/100/150 mg<br>(N=XX) | X4P-001<br>200 mg<br>(N=XX) | X4P-001<br>300 mg<br>(N=XX) | X4P-001<br>400 mg<br>(N=XX) | X4P-001<br>300/400 mg<br>(N=XX) |
|---|---|---|---|---|---|---|---|---|---|
| Number of<br>Infection | XX | xx | xx | XX | xx | XX | XX | XX | XX |
| Events | V0/ V0/ | V// V// | V0/ V0/ | VO/ VO/ | V0/ V0/ | V// V// | V0/ V0/ | \0/\0/ | V0/ V0/ |
| Mean (SD) | XX.XX<br>(XX.XXX) | XX.XX<br>(XX.XXX) | XX.XX<br>(XX.XXX) | XX.XX<br>(XX.XXX) | XX.XX<br>(XX.XXX) | XX.XX<br>(XX.XXX) | XX.XX<br>(XX.XXX) | XX.XX<br>(XX.XXX) | XX.XX<br>(XX.XXX) |
| Standard<br>Error | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median<br>Min, Max<br>95% CI | XX.XX<br>XX.X,XX.X<br>(XX.XX,XX.XX) | XX.XX<br>XX.X,XX.X<br>(XX.XX,XX.XX) | XX.XX<br>XX.X,XX.X<br>(XX.XX,XX.XX) | XX.XX<br>XX.X,XX.X<br>(XX.XX,XX.XX) | XX.XX<br>XX.X,XX.X<br>(XX.XX,XX.XX) | XX.XX<br>XX.X,XX.X<br>(XX.XX,XX.XX) | XX.XX<br>XX.X,XX.X<br>(XX.XX,XX.XX) | XX.XX<br>XX.X,XX.X<br>(XX.XX,XX.XX) | XX.XX<br>XX.X,XX.X<br>(XX.XX,XX.XX |

Abbreviations: CI = Confidence interval; NE = Not estimable; SD = Standard deviation.

Notes: On study infections are identified as all events with a MedDRA System Organ Class of "Infections and infestations". Infection rate is calculated as: for each patient calculate the infection rate for each dose level, then calculate the average for all patients for each dose level. 95% CI is based on normal approximation. Events at dose level are assigned based on the start date of the event occurring within start and end dates of that dose for each subject.

SOURCE: Listing 16.2.7.7

Programming Note: For Rate use ADIR.PARAMCD=OINFRAT2.

#### Table 14.3.3.1 Listing of Serious Adverse Events Safety Population

| Subject<br>Number | Dose<br>Level<br>(mg) | Gender | Age | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date/Time (Day)/<br>End Date/Time (Day)[1] | Severity/<br>Causality [2] | Outcome/<br>Action Taken |
|---|---|---|---|---|---|---|---|
| | 200 | Male | XX | xxxx/ xxxx/ xxxx | DDMMMYYYY/HH:MM (XX)/<br>DDMMMYYYY/HH:MM (XX) | Grade 4/<br>Related | XXX/<br>XXX |
| | 400 | Female | xx | xxxx/ xxxx/ xxxx | DDMMMYYYY/HH:MM (XX)/<br>DDMMMYYYY/HH:MM (XX) | Grade 3/<br>Related | XXX/<br>XXX |
| | 200 | Female | xx | xxxx/ xxxx/ xxxx | DDMMMYYYY/HH:MM (XX)/<br>DDMMMYYYY/HH:MM (XX) | Grade 2/<br>Not Related | XXX/<br>XXX |

Note: Adverse events were coded using MedDRA version 23.1.

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

<sup>[2]</sup> The severity is assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (v4.03).

Table 14.3.3.2
Listing of Treatment Emergent Adverse Events Leading to Discontinuation
Safety Population

| Subject | Dose | | | System Organ Class/<br>Preferred Term/ | Start Date/Time (Day)/ | Severity/ | Outcome/ |
|---|---|---|---|---|---|---|---|
| Number_ | Level (mg) | Gender | Age | Verbatim Term | End Date/Time (Day) | Causality [2] | Action Taken |
| | 200 | Male | XX | xxxx/ xxxx/ xxxx | DDMMMYYYY/HH:MM (XX)/ | Grade 4/ | XXX/ |
| | | | | | DDMMMYYYY/HH:MM (XX) | Related | XXX |
| | 400 | Female | XX | xxxx/ xxxx/ xxxx | DDMMMYYYY/HH:MM (XX)/ | Grade 3/ | XXX/ |
| | | | | | DDMMMYYYY/HH:MM (XX) | Related | XXX |
| | 200 | Female | XX | xxxx/ xxxx/ xxxx | DDMMMYYYY/HH:MM (XX)/ | Grade 2/ | XXX/ |
| | | | | | DDMMMYYYY/HH:MM`(XX) | Not Related | XXX |

Note: Adverse events were coded using MedDRA version 23.1.

SOURCE: 16.2.7.1

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

<sup>[2]</sup> The severity is assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (v4.03).

Table 14.3.4.1 Listing of Out of Reference Range Laboratory Values Safety Population

| Subject | | | | Reference | Dose Level | | Date/Time of Collection | Parameter | Test Result |
|---|---|---|---|---|---|---|---|---|---|
| Number | Age | Gender | Lab Parameter | Range | (mg) | Visit | (Day) [1] | Value | Assessment |
| | | Male | Hemoglobin | XX-XX | 200 | XXXX | DDMMMYYYY:HH:MM (XX) | XX | LOW |
| | | Female | Hemoglobin | XX-XX | 400 | xxxx | DDMMMYYYY:HH:MM (XX) | XX | HIGH |
| | | Female | Haematocrit | XX-XX | 200 | xxxx | DDMMMYYYY:HH:MM (XX) | XX | |

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

SOURCE: Listings 16.2.8.1, 16.2.8.2, 16.2.8.3, 16.2.8.6, 16.2.8.7

Table 14.3.5.1.1
Summary of Actual and Change from Baseline in Hematology Results
Safety Population

Parameter: XXXXXXX

| | | | Dose | Levels | | | _ |
|---|---|---|---|---|---|---|---|
| Study Week/<br>Statistics | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) | Overall<br>(N=XX) |
| Baseline [1] | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Week 2 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| CFB to Week 2 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Neek 3 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| CFB to Week 3 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Week 25 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |

Abbreviation: CFB = Change from Baseline; NE = Not estimable; SD = Standard deviation.

<sup>[1]</sup> Baseline is the last non-missing observation recorded before the first dose on Day 1. Baseline visit is displayed for all dose levels irrespective of whether they were receiving that dose level at baseline.

Table 14.3.5.1.1
Summary of Actual and Change from Baseline in Hematology Results
Safety Population

Parameter: XXXXXXX

| | | | Dose | Levels | | | |
|---|---|---|---|---|---|---|---|
| Study Week/ | 50 mg | 100 mg | 150 mg | 200 mg | 300 mg | 400 mg | Overall |
| Statistics | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| CFB to Week 25 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Extension Visits | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| CFB to Extension Visits | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median <sup>′</sup> | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |

Abbreviation: CFB = Change from Baseline; NE = Not estimable; SD = Standard deviation.

SOURCE: Listing 16.2.8.2

Programming Note: Repeat for ALL hematology parameters

<sup>[1]</sup> Baseline is the last non-missing observation recorded before the first dose on Day 1. Baseline visit is displayed for all dose levels irrespective of whether they were receiving that dose level at baseline.

### Table 14.3.5.1.2 Shift from Baseline in Hematology Results Safety Population

Parameter: XXXXXX; Dose level: XXX mg

| Study Week/ | | Bas | eline | | |
|------------------|-----------|-----------|-----------|-----------|-----------|
| Categories | Low | Normal | High | Missing | Total |
| Week 2 | | | | | |
| Low | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Normal | x (xx.x%) | X (XX.X%) | x (xx.x%) | x (xx.x%) | X (XX.X%) |
| High | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Total | x (xx.x%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | x (xx.x%) |
| Week 3 | | | | | |
| Low | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Normal | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | X (XX.X%) |
| High | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Total | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Week 25 | | | | | |
| Low | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Normal | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| High | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Total | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Extension Visits | | | | | |
| Low | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Normal | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| High | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Total | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Note: Data are presented by parameter and dose. SOURCE: Listing 16.2.8.2

**Programming Note:** Repeat table for **ALL** hematology parameters. Repeat table for 100 mg, 150 mg, 200 mg, 300 mg, 400 mg and Overall.

#### Table 14.3.5.2.1 Summary of Actual and Change from Baseline in Serum Chemistry Results Safety Population

(Same shell as Table 14.3.5.1.1: SOURCE: Listing 16.2.8.1)

Table 14.3.5.2.2 Shift from Baseline in Serum Chemistry Results Safety Population

(Same shell as Table 14.3.5.1.2: SOURCE: Listing 16.2.8.1)

Table 14.3.5.3.1
Summary of Actual and Change from Baseline in Coagulation Results
Safety Population

(Same shell as Table 14.3.5.1.1: SOURCE: Listing 16.2.8.6)

Table 14.3.5.3.2 Shift from Baseline in Coagulation Results Safety Population

(Same shell as Table 14.3.5.1.2: SOURCE: Listing 16.2.8.6)

Table 14.3.5.4.1
Summary of Actual and Change from Baseline in Cytometry Results
Safety Population

(Same shell as Table 14.3.5.1.1: SOURCE: Listing 16.2.8.8, add footnote: Note: Each sample was run 3 times producing triplicate results A, B, C for each laboratory test.

Table 14.3.6.1.1
Summary of Actual and Change from Baseline in Vital Signs
Safety Population

(Same shell as Table 14.3.5.1.1: SOURCE: Listing 16.2.9.2)

Table 14.3.6.2.1
Summary of Actual and Change from Baseline of 12-Lead Electrocardiogram (ECG) Parameters
Safety Population

ECG Parameter: XXXXX

| | | | Dose | Levels | | | _ |
|---|---|---|---|---|---|---|---|
| Study Week /<br>Statistics | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) | Overall<br>(N=XX) |
| Baseline [1] | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Week 5 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| CFB to Week 5 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Week 13 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| CFB to Week 13 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Week 21 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |

Abbreviations: CFB = Change from Baseline; NE = Not estimable; SD = Standard deviation.

<sup>[1]</sup> Baseline is the last non-missing observation recorded before the first dose on Day 1. Baseline visit is displayed for all dose levels irrespective of whether they were receiving that dose level at baseline.

SOURCE: Listing 16.2.9.3.

## Table 14.3.6.2.1 Summary of actual and Change from Baseline of 12-Lead Electrocardiogram (ECG) Parameters Safety Population

ECG Parameter: XXXXX

| | | | Dose Levels | | | | |
|---|---|---|---|---|---|---|---|
| Study Week / | 50 mg | 100 mg | 150 mg | 200 mg | 300 mg | 400 mg | Overall |
| Statistics | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| CFB to Week 21 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | xx.x | xx.x | xx.x | XX.X | XX.X | xx.x | xx.x |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Extension Visits | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | xx.x | XX.X | XX.X | xx.x | xx.x | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| CFB to Extension Visits | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |

Abbreviations: CFB = Change from Baseline; NE = Not estimable, SD = Standard deviation.

<sup>[1]</sup> Baseline is the last non-missing observation recorded before the first dose on Day 1. Baseline visit is displayed for all dose levels irrespective of whether they were receiving that dose level at baseline.

Table 14.3.6.3.1 Summary of Ophthalmologic Examination Results (Local Reader) Safety Populaion

| | Dose Levels | | | | | | |
|---|---|---|---|---|---|---|---|
| Study Week<br>Category | 50 mg<br>(N=X) | 100 mg<br>(N=X) | 150 mg<br>(N=X) | 200 mg<br>(N=X) | 300 mg<br>(N=X) | 400 mg<br>(N=X) | Overall<br>(N=X) |
| Baseline [1]<br>Normal<br>Abnormal - CS | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Abnormal - NCS | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Week 13 | | | | | | | |
| Normal | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Abnormal - CS | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Abnormal - NCS | X (XX.X%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | X (XX.X%) | X (XX.X%) |
| Week 25 EOT | | | | | | | |
| Normal | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Abnormal - CS | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | X (XX.X%) |
| Abnormal - NCS | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | , | , , | , | , | , , | , , | , |

Abbreviations: CS = Clinically significant; NCS = Not clinically significant.
[1] Baseline is the last non-missing observation recorded before the first dose on Day 1. Baseline visit is displayed for all dose levels irrespective of whether they were receiving that dose level at baseline.

Table 14.3.6.3.2 Summary of Ophthalmologic Examination Results (Central Retinal Findings)
Safety Populaion

| | | | Dose | Levels | | | |
|---|---|---|---|---|---|---|---|
| Study Week/ | 50 mg | 100 mg | 150 mg | 200 mg | 300 mg | 400 mg | Overall |
| Categories | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Baseline [1] | | | | | | | |
| Normal | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Abnormal - New Finding - NCS | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Abnormal - New Finding - NCS Abnormal - New Finding - CS | X (XX.X%) | X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Central Retinal Exam Review Not Performed | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Due to Inadequacy of Retinal Photographs | X (XX.X70) | Λ (ΛΛ.Λ/0) | Λ (ΛΛ.Λ/0) | Λ (ΛΛ.Λ/0) | Λ (ΛΛ.Λ /0) | X (XX.X70) | X (XX.X70) |
| 1 , 3 1 | | | | | | | |
| Week 13 | | | | | | | |
| Normal | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Abnormal - Unchanged from Baseline | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Abnormal - New Finding - NCS | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Abnormal - New Finding - CS | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Central Retinal Exam Review Not Performed | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Due to Inadequacy of Retinal Photographs | | | | | | | |
| Week 25 EOT | | | | | | | |
| Normal | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Abnormal - Unchanged from Baseline | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Abnormal - New Finding - NCS | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Abnormal - New Finding - CS | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Central Retinal Exam Review Not Performed | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Due to Inadequacy of Retinal Photographs | , (, 5 (, 7 (, 7 ) | , (, 5 (, , (, 6) | 7. (20.07.70) | . (, 5 (., 1, 1, 0) | 7. (2.0.7.70) | , (, 5 (, , (, 0)) | , (, 5 (, 7 (, 0) |

Abbreviations: CS = Clinically significant; NCS = Not clinically significant.
[1] Baseline is the last non-missing observation recorded before the first dose on Day 1. Baseline visit is displayed for all dose levels irrespective of whether they were receiving that dose level at baseline.

SOURCE: Listing 16.2.9.6

Programming Note: Repeat for other body systems

Table 14.3.6.4 **Summary of Concomitant Medications** Safety Population

| | Dose Levels | | | | | | |
|---|---|---|---|---|---|---|---|
| ATC Class Level 4 Preferred Term (ATC Class Level 5) | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) | Overall<br>(N=XX) |
| Patients with at least one Prior<br>Medication | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| ATC Class 1 | | | | | | | |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | x (xx.x%) | x (xx.x%) | X (XX.X%) | X (XX.X%) | x (xx.x%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| ATC Class 2 | , , | , | , , | , , | , | , | , , |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Note: Percentages are based on the number of patients in the Safety Population.

Medications coded using WHO-DD B3 version September 2020.

Concomitant medications are medications taken or ongoing after the date of the first dose of study drug.

Medications are displayed by descending frequency of Anatomic Therapeutic Chemical (ATC) Level 4 classification, by Preferred Term (PT) within ATC and then alphabetically.

Patients were counted only once for each ATC and PT,

Table 14.3.6.5.1
Summary of Use of Antibiotics, G-CSF, Immunoglobulins, and Imiquamod – Concomitant Medications Safety Population

| | Dose Levels | | | | | | |
|---|---|---|---|---|---|---|---|
| ATC Class Level 4 Preferred Term | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) | Overall<br>(N=XX) |
| Patients with at least one Infection Medication | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| ATC Class 1 | | | | | | | |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| ATC Class 2 | , , | , | , | , , | , | , | , , |
| Preferred Term 1 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 2 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Preferred Term 3 | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |

Note: Percentages are based on the number of patients in the Safety Population.

Medications coded using WHO-DD B3 version September 2020.

Concomitant medications are medications taken or ongoing after the date of the first dose of study drug.

Medications are displayed by descending frequency of Anatomic Therapeutic Chemical (ATC) Level 4 classification, by Preferred Term (PT) within ATC and then alphabetically.

Patients were counted only once for each ATC and PT.

SOURCE: Listing 16.2.9.1

Table 14.3.6.5.2 Summary of Use of Antibiotics, G-CSF, Immunoglobulins, and Imiquamod – Prior Medications Safety Population

(Same shell as Table 14.3.6.5.1: SOURCE: Listing 16.2.9.1. Update footnote to reference prior medications instead of concomitant medications: Prior medication is any medication that is started or ended prior to the first dose of the study medication)

#### Table 14.3.6.6 Summary of Actual and Change from Baseline in SF-36 QOL Scores Safety Population

(Same shell as Table 14.3.5.1.1: SOURCE: Listing 16.2.9.8)

Table 14.3.6.6
Summary of Actual and Change from Baseline in HPV Impact Profile (HIP) Questionnaire - Domain Scores
Safety Population

(Same shell as Table 14.3.5.1.1: SOURCE: Listing 16.2.9.9.2)

Table 14.4.1 Summary of Plasma X4P-001 Concentrations by Dose Level Safety Population

| | | Dose Levels | | | | |
|---|---|---|---|---|---|---|
| Time Point<br>Statistic | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) |
| Predose | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Geometric Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| %CV | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| 30 mins post dose | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Geometric Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| %CV | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| 24 hrs post dose | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Geomètric Mean | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| %CV | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

Abbreviations: CV = Coefficient of variation; NE = Not estimable; SD = Standard deviation.

Note: measurements were made predose and at 30, 60, 90 mins and 2, 3, 4, 8, 12, 16 and 24 hrs post-dose. Unit of plasma X4P-001 concentrations is ng/mL.

SOURCE: Listing 16.2.5.1

Programming Note: Repeat table for all relevant visits.

Table 14.4.2 Summary of Plasma X4P-001 Pharmacokinetic Parameters by Dose Level Safety Population

Study Week: Week 5

| - | | | Dose I | Levels | | |
|---|---|---|---|---|---|---|
| Parameter<br>Statistic | 50 mg<br>(N=XX) | 100 mg<br>(N=XX) | 150 mg<br>(N=XX) | 200 mg<br>(N=XX) | 300 mg<br>(N=XX) | 400 mg<br>(N=XX) |
| AUC Over Dosing Interval (h*ng/mL) | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Geometric Mean [95%CI] | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| %CV | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| CMax (ng/mL) | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Geomètric Mean [95%CI] | xx.x | xx.x | xx.x | XX.X | XX.X | XX.X |
| · | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| %CV | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Time of CMax (h) | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Geometric Mean [95%CI] | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] |
| Median | XX.X | XX.X | XX.X | ` XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| %CV | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

Note: As some subjects provided multiple values for the same dose level, median values were taken at the same dose level for each subject, the median values were then used in the analysis.

Abbreviations: AUC = Area under the plasma concentration; CV = Coefficient of variation; NE = Not estimable; SD = Standard deviation.

SOURCE: Listings 16.2.5.1, 16.2.5.2

Programming Note: Repeat table for all applicable visits.

#### 14.3. Planned Figure Shells

Figure 14.4.1.1 WBC over Time by Patient Safety Population

Y-axis: Leukocytes (10^9/L)

X-axis: Weeks Since First Study Treatment

\*Value obtained during infection and considered to be confounded.

SOURCE: Listing 16.2.8.2

Programming Note: If a patient has multiple values at a particular time point, use mean.

Figure 14.4.1.2a
ANC over Time by Patient
Safety Population

Header: Patient ID = XXX-XXX
Y-axis: ANC Value (10^9/L)

X-axis: Hours Since Study Treatment

Footnote:

Note: The imputation of baseline observation carried forward (BOCF) is used for missing 24 hour assessment. Patients and took the Week 5 dose at home instead of the clinic resulting in the site not getting dense PK samples for the first few hours. Therefore, samples were taken the next day and the timepoints that were missed the day before were replaced with these samples. Patient assessments on 21 and 22 February 2018 were analyzed and presented as Week 21 assessments. For patient the assessment on 20FEB2018 at 9:25 was used as time 0.

Patient , Extension Phase - Residence Visit 1 Post EOS and Extension Phase - Residence Visit 3 occurred during episodes of infection. These values were excluded from the analysis. Patient , Week 21 occurred during an episode of infection. These values were excluded from the analysis.

Dense sample data for subject will be excluded from the TAT summary tables and figures since the WBC, ANC, ALC, and AMC levels were normal at screening due to splenectomy.

\*Value obtained during infection and considered to be confounded.

SOURCE: Listing 16.2.6.1

Programming Note: If a patient has multiple values at a particular time point, use mean.

Figure 14.4.1.2b
ANC over Time by Dose Level
Safety Population

**Header:** Treatment Level (mg) = XXX **Y-axis:** ANC Value (10^9/L)

**X-axis:** Hours Since Study Treatment

Footnote:

Note: The imputation of baseline observation carried forward (BOCF) is used for missing 24 hour assessment. Patients and took the Week 5 dose at home instead of the clinic resulting in the site not getting dense PK samples for the first few hours. Therefore, samples were taken the next day and the timepoints that were missed the day before were replaced with these samples. Patient assessments on 21 and 22 February 2018 were analyzed and presented as Week 21 assessments. For patient the assessment on 20FEB2018 at 9:25 was used as time 0.

| Patient , Extension Phase - Residence Visit 1 Post EOS and Extension Phase - Residence Visit 3 occurred during episodes of infection. These values were excluded from the analysis. Patient , Week 21 occurred during an episode of infection. These values were excluded from the analysis. Dense sample data for subject will be excluded from the TAT summary tables and figures since the WBC, ANC, ALC, and AMC levels were normal at screening due to splenectomy. SOURCE: Listing 16.2.6.1 Programming Note: If a patient has multiple values at a particular time point, use mean. |
|---|
| Figure 14.4.1.3a<br>ALC over Time by Patient<br>Safety Population |
| Header: Patient ID = XXX-XXX Y-axis: ALC Value (10^9/L) X-axis: Hours Since Study Treatment Footnote: Note: The imputation of BOCF is used for missing 24 hour assessment. Patients and getting dense PK samples for the first few hours. Therefore, samples were taken the next day and the timepoints that were missed the day before were replaced with these samples. Patient assessments on 21 and 22 February 2018 were analyzed and presented as Week 21 assessments. For patient the assessment on 20FEB2018 at 9:25 was used as time 0. Patient the analysis. Patient the analysis occurred during episodes of infection. These values were excluded from the analysis. Patient the analysis occurred during an episode of infection. These values were excluded from the TAT summary tables and figures since the WBC, ANC, ALC, and AMC levels were normal at screening due to splenectomy. *Value obtained during infection and considered to be confounded. SOURCE: Listing 16.2.6.1 *Programming Note: If a patient has multiple values at a particular time point, use mean. |
| Figure 14.4.1.3b<br>ALC over Time by Dose Level<br>Safety Population |
| Header: Treatment Level (mg) = XXX Y-axis: ALC Value (10^9/L) X-axis: Hours Since Study Treatment Footnote: Note: The imputation of BOCF is used for missing 24 hour assessment. Patients and getting dense PK samples for the first few hours. Therefore, samples were taken the next day and the timepoints that were missed the day before were replaced with these samples. Patient assessments on 21 and 22 February 2018 were analyzed and presented as Week 21 assessments. For patient the assessment on 20FEB2018 at 9:25 was used as time 0. Patient personal patient person |

Figure 14.4.1.4a Monocytes over Time by Patient Safety Population Header: Patient ID = XXX-XXX Y-axis: AMC Value (10^9/L)

X-axis: Hours Since Study Treatment

Footnote:

Note: The imputation of BOCF is used for missing 24 hour assessment. Patients and getting dense PK samples for the first few hours. Therefore, samples were taken the next day and the timepoints that were missed the day before were replaced with these samples. Patient assessments on 21 and 22 February 2018 were analyzed and presented as Week 21 assessments. For patient the assessment on 20FEB2018 at 9:25 was used as time 0. Patient Examples, Extension Phase - Residence Visit 1 Post EOS and Extension Phase - Residence Visit 3 occurred during episodes of infection. These values were excluded from the analysis. Patient Week 21 occurred during an episode of infection. These values were excluded from the TAT summary tables and figures since the WBC, ANC, ALC, and AMC levels were normal at screening due to splenectomy.

\*Value obtained during infection and considered to be confounded.

SOURCE: Listing 16.2.6.2.4

Programming Note: If a patient has multiple values at a particular time point, use mean.

### Figure 14.4.1.4b Monocytes over Time by Dose Level Safety Population

**Header:** Treatment Level (mg) = XXX **Y-axis:** AMC Value (10^9/L) **X-axis:** Hours Since Study Treatment

Footnote:

Note: The imputation of BOCF is used for missing 24 hour assessment. Patients and took the Week 5 dose at home instead of the clinic resulting in the site not getting dense PK samples for the first few hours. Therefore, samples were taken the next day and the timepoints that were missed the day before were replaced with these samples. Patient assessments on 21 and 22 February 2018 were analyzed and presented as Week 21 assessments. For patient the assessment on 20FEB2018 at 9:25 was used as time 0. Patient personal pers

**Programming Note:** If a patient has multiple values at a particular time point, use mean.
Figure 14.4.1.5
Mean (+/– SE) Plasma Concentration - Time Profile of X4P-001 by Dose Level
Safety Population



**Header:** Treatment Level (mg) = XXX

Y-axis: Mean X4P-001 plasma concentrations (ng/mL)

**X-axis:** Time Point (hours postdose)

SOURCE: Table 14.4.1

Programming Note:All visits will be presented on the same figure. If a patient has multiple values at a particular time point, use median.





**Y-axis:** Mean Neutrophils (10^9/L) **X-axis:** Time Point (hours postdose)

Patient , Extension Phase - Residence Visit 1 Post EOS and Extension Phase – Residence Visit 3 occurred during episodes of infection. These values were excluded from the analysis. Patient , Week 21 occurred during an episode of infection. These values were excluded from the analysis. Dense sample data for subject will be excluded from the TAT summary tables and figures since the WBC, ANC, ALC, and AMC levels were normal at screening due to splenectomy.

The ANC threshold (500 neutrophils per microliter) is indicated by the blue line.

SOURCE: Listing 16.2.8.2

**Programming Note:** All visits will be presented on the same figure. If a patient has multiple values at a particular time point, use mean. No reference line required. All relevant visits should be used for derivation, and not limited to Weeks 5, 13 and 21.

# Figure 14.4.1.7 Mean Dose Response of ALC - Time Profile Safety Population

(Same shell as Table 14.4.1.6)

analysis. Patient with the same and extension Phase – Residence visit 3 occurred during episodes of infection. These values were excluded from the analysis. Dense sample data for subject will be excluded from the TAT summary tables and figures since the WBC, ANC, ALC, and AMC levels were normal at screening due to splenectomy.

The ALC threshold (1000 cells per microliter) is indicated by the blue line.

SOURCE: Listing 16.2.8.2

**Programming Note:** All visits will be presented on the same figure, If a patient has multiple values at a particular time point, use mean. Reference line at y=1 required. All relevant visits should be used for derivation, and not limited to Weeks 5, 13 and 21

Figure 14.4.1.8

Mean Dose Response of Monocytes - Time Profile
Safety Population

(Same shell as Table 14.4.1.6)

**Y-axis:** Mean Monocytes (10^9/L) **X-axis:** Time Point (hours postdose)

Patient , Extension Phase - Residence Visit 1 Post EOS and Extension Phase – Residence Visit 3 occurred during episodes of infection. These values were excluded from the analysis. Patient , Week 21 occurred during an episode of infection. These values were excluded from the analysis. Dense sample data for subject will be excluded from the TAT summary tables and figures since the WBC, ANC, ALC, and AMC levels were normal at screening due to splenectomy.

SOURCE: Listing 16.2.8.2

Programming Note: All visits will be presented on the same figure. If a patient has multiple values at a particular time point, use mean. No reference line required. All relevant visits should be used for derivation, and not limited to Weeks 5, 13 and 21

Figure 14.4.1.9
Box plots of WBC change from baseline ratio at 300mg and 400mg by Dose Level Safety Population



Y-axis: WBC Change from baseline (ratio)

X-axis: X4P-001 dose (mg QD)

Patient Patient Patient Patient Phase - Residence Visit 1 Post EOS and Extension Phase - Residence Visit 3 occurred during episodes of infection. These values were excluded from the analysis. Patient Week 21 occurred during an episode of infection. These values were excluded from the analysis. Dense sample data for subject will be excluded from the TAT summary tables and figures since the WBC, ANC, ALC, and AMC levels were normal at screening due to splenectomy.

SOURCE: Listing 16.2.8.2

**Programming Note:** All visits will be presented on the same figure. Use mean value across visits. The ratio is to be calculated as visit value / baseline value, same as fold-change.

Figure 14.4.1.10
Box plots of AUC for ANC by Dose Level
Safety Population



Y-axis: AUC<sub>ANC</sub> (10^9/L) X-axis: X4P-001 dose (mg QD)

Patient , Extension Phase - Residence Visit 1 Post EOS and Extension Phase - Residence Visit 3 occurred during episodes of infection. These values were excluded from the analysis. Patient , Week 21 occurred during an episode of infection. These values were excluded from the analysis. Dense sample data for subject will be excluded from the TAT summary tables and figures since the WBC, ANC, ALC, and AMC levels were normal at screening due to splenectomy.

SOURCE: Table 14.2.6.2.1

Programming Note: All visits will be presented on the same figure. If a patient has multiple values at a particular time point, use mean.

Figure 14.4.1.11
Scatter Plot of Time above Threshold values for ANC versus AUC for ANC Safety Population



Y-axis: Time Above Threshold for ANC (hours)

X-axis: X4P-001 AUC (ng\*hr/mL)

Patient , Extension Phase - Residence Visit 1 Post EOS and Extension Phase - Residence Visit 3 occurred during episodes of infection. These values were excluded from the analysis. Patient , Week 21 occurred during an episode of infection. These values were excluded from the analysis. Dense sample data for subject will be excluded from the TAT summary tables and figures since the WBC, ANC, ALC, and AMC levels were normal at screening due to splenectomy.

SOURCE: Table 14.2.9, Listing 16.2.6.2.3

Programming Note: display Pearson correlation coefficient (r) in the plot

Figure 14.4.1.12
Scatter Plot of Time above Threshold values for ALC versus AUC for ALC
Safety Population

(Same shell as Table 14.4.1.11)

Y-axis: Time Above Threshold for ALC (hours)

X-axis: X4P-001 AUC (ng\*hr/mL)

Patient Patien

SOURCE: Table 14.2.10, Listing 16.2.6.2.3

Programming Note: display Pearson correlation coefficient (r) in the plot

Figure 14.4.1.13.1
Plot of Yearly Infection Rate by Dose Level
Safety Population



Y-axis: Annualized Infection Rate (95% CI)

**X-axis:** X4P-001 dose (mg QD) SOURCE: Table 14.3.2.7.1

**Programming Note:** For Rate use ADIR.PARAMCD=OINFRATE. For number of infection events use NOINF along with appropriate DOSEA. Table 14.3.2.7 doesn't have a pre-study column.

### Add footnote:

Notes: Infections are identified as follows: for Prior 12 months, events are identified from the Medical History CRF under History of WHIM infections. While on study, infections are identified as all events with a MedDRA System Organ Class of "Infections and infestations". Rate is defined as number of infection events in a given dose level /duration of exposure on a dose level in years. 95% CI is based on normal approximation. Events at dose level are assigned based on the start date of the event occurring within start and end dates of that dose for each patient. Confidence limits below 0 are not shown.

# Figure 14.4.1.13.2 Plot of Yearly Infection Score by Dose Level Safety Population

Y-axis: Infection Score (95% CI) X-axis: X4P-001 dose (mg QD) SOURCE: Table 14.2.2.3

Programming Note: For Rate use ADIR.PARAMCD=OINFSC along with appropriate DOSEA. Pre-study infection score is not calculated.

Table 14.3.2.7 doesn't have a pre-study column.

### Add footnote:

Notes: Infections are identified as follows: for Prior 12 months, events are identified from the Medical History CRF under History of WHIM infections. While on study, infections are identified as all events with a MedDRA System Organ Class of "Infections and infestations". Infection Score is defined as number of infection events in a given dose level divided by duration of exposure on a dose level, in years. 95% CI is based on normal approximation. Events at dose level are assigned based on the start date of the event occurring within start and end dates of that dose for each patient.

Figure 14.4.1.14.1
Plot of Yearly Infection Rate for Subjects on 300mg and 400 mg Dose Levels by 6 Month Intervals
Safety Population



Y-axis: Annualized Infection Rate (95% CI)

X-axis: Time on Study SOURCE: Table 14.3.2.6.1

#### Programming Note:

For Pre-study infection rate use ADIR.PARAMCD=PINFRATE

For 0-6 months, ADIR.PARAMCD=OINFRTBP and DOSEA in (300,400) and ETINFG1=0 – 6 Months. For 6-12 months, ADIR.PARAMCD=OINFRTBP and DOSEA in (300,400) and ETINFG1=6 – 12 Months. And so on

For 0-6 months, for Number of infection events- ADIR.NOINFBP and DOSEA in (300,400) and ETINFG1=0 – 6 Months. For 6-12 months, for Number of infection events- ADIR.NOINFBP and DOSEA in (300,400) and ETINFG1=6 – 12 Months. And so on...

#### Add footnote:

Notes: Infections are identified as follows: for Prior 12 months, events are identified from the Medical History CRF under History of WHIM infections. While on study, infections are identified as all events with a MedDRA System Organ Class of "Infections and infestations". The reporting period starts on the 300 mg dose date. Rate is defined as number of infection events in a given period /duration of period in years. 95% CI is based on normal approximation. Only events with start date occurring within start and end dates of 300/400 mg dose for each patient are included. Time period assignment is based on the start date of the event. Confidence limits below 0 are not shown.

# Figure 14.4.1.14.2 Plot of Yearly Infection Score for Subjects on 300 mg and 400 mg Dose Levels by 6 Month Intervals Safety Population

Y-axis: Infection Score (95% CI)

**X-axis:** Time on Study SOURCE: Table 14.3.2.6.2

#### Programming Note:

For Pre-study infection rate use ADIR.PARAMCD=NPINF and DOSEA in (300,400).
For 0-6 months, ADIR.PARAMCD=OINFSCBP and DOSEA in (300,400) and ETINFG1=0-6 Months.
For 6-12 months, ADIR.PARAMCD=OINFSCBP and DOSEA in (300,400) and ETINFG1=6-12 Months.

• • • •

For 0-6 months, for Number of infection events- ADIR.OINFSCBP and DOSEA in (300,400) and ETINFG1=0-6 Months. For 6-12 months, for Number of infection events- ADIR.OINFSCBP and DOSEA in (300,400) and ETINFG1=6-12 Months.

. . .

Pre-study infection score is not calculated.

#### Add footnote:

Notes: Infections are identified as follows: for Prior 12 months, events are identified from the Medical History CRF under History of WHIM infections. While on study, infections are identified as all events with a MedDRA System Organ Class of "Infections and infestations". The reporting period starts on the 300 mg dose date. Rate is defined as number of infection events in a given period /duration of period in years. 95% CI is based on normal approximation. Only events with start date occurring within start and end dates of 300/400 mg dose for each patient are included. Time period assignment is based on the start date of the event.

### Figure 14.4.2.1 Scatter Plot of Plasma Drug Level and ANC Safety Population

Y-axis: Neutrophils (10^9/L)

X-axis: X4P-001 plasma concentration (ng/mL)

Patient , Extension Phase - Residence Visit 1 Post EOS and Extension Phase - Residence Visit 3 occurred during episodes of infection. These values were excluded from the analysis. Patient , Week 21 occurred during an episode of infection. These values were excluded from the analysis. Dense sample data for subject will be excluded from the TAT summary tables and figures since the WBC, ANC, ALC, and AMC levels were normal at screening due to splenectomy.

SOURCE: Table 14.4.1, Listing 16.2.6.1

Programming Note: All visits will be presented on the same figure, If a patient has multiple values at a particular time point, use mean.

Figure 14.4.2.2 Scatter Plot of Plasma Drug Level and ALC Safety Population

Y-axis: Lymphocytes (10^9/L)

X-axis: X4P-001 plasma concentration (ng/mL)

Patient , Extension Phase - Residence Visit 1 Post EOS and Extension Phase – Residence Visit 3 occurred during episodes of infection. These values were excluded from the analysis. Patient , Week 21 occurred during an episode of infection. These values were excluded from the analysis. Dense sample data for subject will be excluded from the TAT summary tables and figures since the WBC, ANC, ALC, and AMC levels were normal at screening due to splenectomy.

SOURCE: Table 14.4.1, Listing 16.2.6.1

Programming Note: All visits will be presented on the same figure. If a patient has multiple values at a particular time point, use mean.

Figure 14.4.3.1

Mean Plasma Concentrations of X4P-001 vs Nominal Time (Dense Sampling Visits) by Dose Level - Linear Scale Safety Population

**Header:** Treatment Level (mg) = XXX

**Y-axis:** Mean X4P-001 plasma concentration (ng/mL)

**X-axis:** Time Point (hours postdose)

SOURCE: Table 14.4.1

Programming Note: All visits will be presented on the same figure, If a patient has multiple values at a particular time point, use median.

Figure 14.4.3.2

Mean Plasma Concentrations of X4P-001 vs Nominal Time (Dense Sampling Visits) by Dose Level - Semi-Logarithmic Scale Safety Population

**Header:** Treatment Level (mg) = XXX

Y-axis: Mean X4P-001 plasma concentration (ng/mL)

**X-axis:** Time Point (hours postdose)

SOURCE: Table 14.4.1

Programming Note: All visits will be presented on the same figure, If a patient has multiple values at a particular time point, use median.

#### Figure 14.4.4.1

Subject Plasma Concentrations of X4P-001 vs Nominal Time (Dense Sampling Visits) by Dose Level - Linear Scale Safety Population

**Header:** Patient ID = XXX, Treatment Level (mg) = XXX **Y-axis:** X4P-001 plasma concentration (ng/mL)

**X-axis:** Time Point (hours postdose)

SOURCE: Listing 16.2.5.1

Programming Note: All visits will be presented on the same figure, If a patient has multiple values at a particular time point, use median.

### Figure 14.4.4.2

Subject Plasma Concentrations of X4P-001 vs Nominal Time (Dense Sampling Visits) by Dose Level - Semi-Logarithmic Scale Safety Population

**Header:** Patient ID = XXX, Treatment Level (mg) = XXX

Y-axis: X4P-001 plasma concentration (ng/mL)

**X-axis:** Time Point (hours postdose)

SOURCE: Listing 16.2.5.1

Programming Note: All visits will be presented on the same figure, If a patient has multiple values at a particular time point, use median.

## 14.4. Planned Listing Shells

Global programming note: for all listings, sort by subject number. Further sorting instructions will be provided if needed.

### Listing 16.2.1 Subject Disposition All Enrolled Patients

| | | | | Phase II Treat | tment Period | Extension<br>Phase | End of Study | |
|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Gender | Date of Last Dose<br>(Day) [1] | Status | Date of Completion/<br>Discontinuation<br>(Day) [1] | Reason for Discontinuation | Status | Date Extension Phase<br>Discontinued | Reason for<br>Discontinuatio<br>n |
| xxxxxx | Male | DDMMMYYYY (X) | Off | DDMMMYYYY (XX) | | Ongoing | | |
| XXXXXX | Female | DDMMMYYYY (X) | Off | DDMMMYYYY (XX) | | N/A | | |
| XXXXXX | | DDMMMYYYY (X) | Off | DDMMMYYYY (XX) | | | | |
| XXXXXX | | DDMMMYYYY (X) | Off | DDMMMYYYY (X) | XXXXXXXXXX: XXXXXXXXX | | | |
| XXXXXX | | DDMMMYYYY (X) | Off | DDMMMYYYY (XX) | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | |

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug, then data extraction date is used.

A subject that is no longer in the Phase II Treatment Period has a status of 'Off'.

Programming Note: If reason for early termination is other, concatenate the specify text as follows: "Other: XXXXXXXXX".

If reason for early termination is lost to follow-up, concatenate with date of last contact as follows: "Lost to follow-up; date of last contact: DDMMMYYYY".

If reason for discontinuation is a PI decision, concatenate PI decision reason as follows: "PI Decision: XXXXXXXXXXXX".

### Listing 16.2.2.1 Eligibility Criteria Not Met All Enrolled Patients

| | | | Date | | |
|---|---|---|---|---|---|
| Subject Number | Gender | Screening (Day)[1] | Informed Consent (Day)[1] | All Inclusion<br>Criteria Met? | Any Exclusion<br>Criteria Met? |
| XXXXXX | xxxx | DDMMMYYYY (-X) | DDMMMYYYY (-X) | Yes | No |
| xxxxx | XXXXXX | DDMMMYYYY (-X) | DDMMMYYYY (-X) | No: 02, 09 | No |
| xxxxx | XXXXXX | DDMMMYYYY (-X) | DDMMMYYYY (-X) | No: 06 | No |
| xxxxx | XXXX | DDMMMYYYY (-X) | DDMMMYYYY (-X) | Yes | Yes: 06 |
| XXXXXX | XXXXXX | DDMMMYYYY (-X) | DDMMMYYYY (-X) | Yes | No |
| XXXXXX | XXXX | DDMMMYYYY (-X) | DDMMMYYYY (-X) | Yes | No |
| XXXXXX<br>XXXXXX | XXXXXX<br>XXXX | DDMMMYYYY (-X) DDMMMYYYY (-X) DDMMMYYYY (-X) | DDMMMYYYY (-X) DDMMMYYYY (-X) DDMMMYYYY (-X) | No: 06<br>Yes<br>Yes | No<br>Yes: 06<br>No |

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

Programming note: If more than 1 inclusion or exclusion criterion number exists, concatenate with a comma. Decode any relevant criteria in the footnotes.

## Listing 16.2.2.2 Protocol Deviations Safety Population

| Subject<br>Number | Gender | Deviation Date | Deviation Category | Violation<br>Level | Description |
|---|---|---|---|---|---|
| xxxxx | XXXXXX | DDMMMYYYY | xxxxxxxxxx<br>xxxxxxxxxxxxxxxxxxxxxxxxxxx | Important (NCS)<br>Non-Important | xxxxxx<br>xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXXXX | DDMMMYYYY | xxxxxxxxxxx<br>xxxxxxxxxxxxxxxxxxxxxxxxxx | Non-Important<br>Non-Important | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | xxxxx | DDMMMYYYY | XXXXXXXXXXX | Important (CS) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

Abbreviations: CS = Clinically significant; NCS = Not clinically significant.

# Listing 16.2.3 Analysis Populations All Enrolled Patients

| Subject Number | Gender | SP<br>[1] | ITT<br>[2] |
|----------------|--------|-----------|------------|
| xxxxxx | XXXXXX | Yes | No |
| XXXXXX | xxxxx | Yes | Yes |
| XXXXXX | xxxxx | No | No |

Abbreviations: ITT = Intent to Treat Population; SP= Safety Population.
[1] The Safety Population includes all patients who receive any amount of study medication.
[2] The ITT Population is the same as the Safety Population and includes all patients who receive any amount of study medication.

Listing 16.2.4.1
Demographics and Baseline Characteristics
Safety Population

| Subject Number | Gender | Age<br>(years) | Ethnicity | Race | Weight<br>(kg) | Height<br>(cm) | BMI<br>(kg/m2) |
|---|---|---|---|---|---|---|---|
| xxxxxx | XXXXXX | XX | Not Hispanic or<br>Latino | xxxxxx | XX.X | XX.X | XX.XX |
| XXXXXX | XXXXXX | XX | Hispanic or Latino | XXXXXX | XX.X | XX.X | XX.XX |
| XXXXXX | XXXXXX | XX | | XXXXXX | XX.X | XX.X | XX.XX |
| XXXXXX | XXXX | XX | | XXXXX | XX.X | XX.X | XX.XX |
| XXXXXX | XXXXXX | XX | | XXXXXX | XX.X | XX.X | XX.XX |
| XXXXXX | XXX | XX | | XXXXXX | XX.X | XX.X | XX.XX |

Abbreviation: BMI = Body mass index

**Programming Note:** If race is other, concatenate "Other:" with specify text. If patient has multiple races, concatenate them

## Listing 16.2.4.2 Medical History Safety Population

| Subject | System Organ Class / | Start date(Day) / Currently Active? |
|---------|----------------------|-------------------------------------|
| Number | Preferred Term / | End Date(Day)[1] |
| | Verbatim Term | |
| | XXXX/ | DDMMMYYYY(XX) / |
| | XXX/ | DDMMMYYYY(XX) |
| | XXX | |
| | XXXX/ | DDMMMYYYY(XX)/ |
| | XXX/ | DDMMMYYYÝ(XX) |
| | XXX | |
| | XXXX/ | DDMMMYYYY(XX) / |
| | XXX/ | DDMMMYYYY(XX) |
| | XXX | |

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

# Listing 16.2.4.3.1 History of WHIM Syndrome - Hospitalizations Safety Population

| Subject Number | Prior Hospitalization for Infection? | Start Date (Day) /<br>End Date (Day) [1] | Reason for Hospitalization | Duration [2] |
|---|---|---|---|---|
| | Yes | DDMMMYYYY (XX) /<br>DDMMMYYYY (XX) | | |
| | No | | | |
| | No | | | |

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug. [2] Duration = End Date - Start Date + 1

## Listing 16.2.4.3.2 History of WHIM Syndrome - Infections Managed as Out-Patient Safety Population

| Subject<br>Number | Any Prior Infections Managed as Out-Patient? | Start Date (Day)/<br>End Date (Day) [1] | Antibiotic Used? | Type of Infection | Duration [2] |
|---|---|---|---|---|---|
| | Yes | DDMMMYYYY (XX)/<br>DDMMMYYYY (XX) | Yes | | |
| | | | No | | |

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

<sup>[2]</sup> Duration = End Date – Start Date + 1

# Listing 16.2.4.3.3 History of WHIM Syndrome - Prior Treatments for WHIM syndrome Safety Population

| DDMMMYYYY(XX)/ | Subject Number | Any Prior<br>Treatments of<br>WHIM? | Agent | Start Date (Day)/<br>End Date (Day) [1] | Route | AE Related to<br>Treatment | Best<br>Clinical<br>Response<br>(Specify) | Reason for discontinuation (Specify) |
|---|---|---|---|---|---|---|---|---|
| DDIVINITY Y Y (AA) | | | | DDMMMYYYY(XX)/<br>DDMMMYYYY(XX) | | | | |

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

## Listing 16.2.4.3.4 WHIM Syndrome Genotyping Safety Population

| | Was Genotyping | | | WHIM Diagnosis |
|---|---|---|---|---|
| Subject Number | Sample Collected? | Date Collected (Day) [1] | CXCR4 Genotyping Variant | Date |
| | Yes | DDMMMYYYY(XX) | Other: XXXXXX | DDMMMYYYY |
| | | DDMMMYYYY (XX) | | |
| | | DDMMMYYYY (XX) | | |

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

# Listing 16.2.4.4.1 Study Drug Administration Safety Population

| Subject<br>Number | Capsule<br>Strength<br>(mg) | Dose<br>Level<br>(mg) | Did Subject<br>Receive<br>Treatment? | Start Date (Day)/<br>Stop Date (Day) [1] | Number of<br>Days on Dose<br>Level [2] | Ongoing? | Route | Frequency | Any Doses<br>Not<br>Taken? | Reason<br>Not<br>Taken | Number Of Doses<br>Not Taken |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | 25 | 100 | Yes | DDMMMYYYY (XX)/<br>DDMMMYYYY (XX) | | Yes | Oral | QD | | | |
| | 25 | 100<br>200<br>300 | | , | | | | | | | |
| | 100 | 100<br>100<br>100<br>200 | | | | | | | | | |
| | | 200<br>200<br>300<br>400 | | | | | | | | | |

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

[2] Number of days on Dose Level = Last Date on Dose Level - Start Date on Dose Level + 1.

# Listing 16.2.4.4.2 Study Drug Exposure Safety Population

| Subject<br>Number | Capsule<br>Strength<br>(mg) | Dose Level<br>(mg) | Total number of Capsules Dispensed | Date Dispensed (Day)<br>[1] | Total number of<br>Capsules<br>Returned | Date Returned (Day)<br>[1] | Percent compliance | Treatment<br>Duration | Number of<br>Doses<br>Missed or<br>skipped |
|---|---|---|---|---|---|---|---|---|---|
| | 25<br>25 | 100<br>100<br>200<br>300 | | DDMMMYYYY (XX) | | DDMMMYYYY (XX) | | | |
| | 100 | 100<br>100<br>100<br>200<br>200<br>200<br>200<br>300 | | | | | | | |

Percent compliance = [1-(Total number of capsules returned/Total number of capsules dispensed)] x 100.
[1] Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

### Listing 16.2.4.5 Assessment of Warts Safety Population

| Subject<br>Number | Visit | Capsule<br>Strength<br>(mg) | Dose<br>Level<br>(mg) | Was<br>Assessment<br>of Warts Done? | Date Performed (Day) [1] | Area of<br>Assessment | Were any warts in area of assessment? | Number of<br>warts in the<br>area of<br>assessment | Change from baseline in the number of warts |
|---|---|---|---|---|---|---|---|---|---|
| | Screening | | | Yes | DDMMMYYYY (X) | BOTTOM LEFT FOOT | No | | |
| | | | | | | BOTTOM LEFT HAND | No | | |
| | | | | | | BOTTOM RIGHT FOOT | Yes | 2 | |
| | | | | | | BOTTOM RIGHT HAND | No | | |
| | | | | | | TOP LEFT FOOT | No | | |
| | | | | | | TOP LEFT HAND | No | | |
| | | | | | | TOP RIGHT FOOT | No | | |
| | | | | | | TOP RIGHT HAND | No | | |
| | | | | | | TOTAL NUMBER OF WARTS ACROSS<br>ALL AREAS OF ASSESSMENT | < <li>4 any of above=Yes then populate cell to the right&gt;&gt;</li> | XX | |
| | Day 1 | 25 | 50 | Yes | DDMMMYYYY (X) | BOTTOM LEFT FOOT | No | | |
| | | | | | | BOTTOM LEFT HAND | No | | |
| | | | | | | BOTTOM RIGHT FOOT | Yes | XX | |
| | | | | | | BOTTOM RIGHT HAND | No | | |
| | | | | | | TOP LEFT FOOT | No | | |
| | | | | | | TOP LEFT HAND | No | | |
| | | | | | | TOP RIGHT FOOT | No | | |
| | | | | | | TOP RIGHT HAND | No | | |
| | | | | | | TOTAL NUMBER OF WARTS ACROSS<br>ALL AREAS OF ASSESSMENT | < <li>&lt;<li>any of above=Yes<br/>then populate cell to<br/>the right&gt;&gt;</li></li> | XX | |
| | Week 5 | 25 | 50 | Yes | DDMMMYYYY (X) | BOTTOM LEFT FOOT | No | | |
| | | | | | | BOTTOM LEFT HAND | No | | |
| | | | | | | BOTTOM RIGHT FOOT | Yes | XX | XX |

[1] Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

Note: Baseline is the number of warts at Day 1.

An out of schedule assessment of warts was done at end of study visit for subject

Patient was re-enrolled into the study on DDMMMYYYY.

Patient was re-enrolled into the study on DDMMMYYYY.

Programming Note: present all data including data after re-enrollment for the 2 re-enrolled patients

## Listing 16.2.4.6 Revaccination Safety Population

| Subject<br>Number | Date of Dose<br>(Day) [1] | Capsule<br>strength<br>(mg) | Dose<br>Level<br>(mg) | Was Patient Revaccinated? | Type Of Revaccination | Date Of Revaccination (Day) [1] |
|---|---|---|---|---|---|---|
| | DDMMMYYYY (XX) | 25 | 100<br>100<br>200<br>300<br>100<br>100<br>100<br>200<br>200<br>200<br>300 | Yes | Tetanus toxoid | DDMMMYYYY (XX) |

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

## Listing 16.2.4.7 Bone Marrow Aspirate Safety Population

| Subject Number | Visit | Date Performed (Day) [1] | Was Bone Marrow aspirate Performed? | |
|---|---|---|---|---|
| | Screening | | Yes | _ |
| | Week 25 | | | |
| | Day 1 | | | |
| | Week 5 | | | |
| | Week 13 | | | |
| | Week 21 | | | |
| | Day 1 | | | |
| | Week 5 | | | |
| | Week 13 | | | |
| | Week 21 | | | |

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

# Listing 16.2.5.1 Pharmacokinetic Blood Collection and Concentrations Safety Population

| Subject<br>Number | Visit | Capsule<br>strength<br>(mg) | Dose<br>Level<br>(mg) | Was the Sample collected? | Reason Sample Not<br>Collected | Date/Time<br>Collected (Day) [1] | Time Point | X4P-001<br>Concentration<br>(ng/mL) |
|---|---|---|---|---|---|---|---|---|
| | Day 1 | 25 | 100 | Yes | xxxxx | DDMMMYYYY (X) | Predose | XXXX |
| | | | | | | | 30 mins postdose | XXXX |
| | | | | | | | 60 mins postdose | XXXX |
| | | | | | | | 90 mins postdose | XXXX |
| | | | | | | | 2 hours postdose | XXXX |
| | | | | | | | 3 hours postdose | XXXX |
| | | | | | | | 4 hours postdose | XXXX |
| | | | | | | | 8 hours postdose | XXXX |
| | | | | | | | 12 hours postdose | XXXX |
| | | | | | | | 16 hours postdose | XXXX |
| | | | | | | | 24 hours postdose | XXXX |

[1] Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

Patients and and took the Week 5 dose at home instead of the clinic resulting in the site not getting dense PK samples for the first few hours. Therefore, samples were taken the next day and the timepoints that were missed the day before were replaced with these samples. Patient and presented as Week 21 assessments.

# Listing 16.2.5.2 Calculated Pharmacokinetic Parameters Safety Population

| Subject<br>Number | Visit | Actual dose<br>of X4P-001 (mg) | AUC Over Dosing<br>Interval (h*ng/mL) | Tmax<br>(h) | Cmax<br>(ng/mL) |
|---|---|---|---|---|---|
| | Week 5 | 100 | Yes | | Yes |
| | Week 13 | 100 | | | |
| | Week 21 | 200 | | | |
| | Week 5<br>Week 13 | 100<br>200 | | | |
| | Week 21 | 100 | | | |
| | Week 5 | 200 | | | |
| | Week 13<br>Week 21 | 200<br>300 | | | |

Note: Imputed concentrations at 24 hours with predose values were used for PK parameter calculation.

Abbreviation: AUC = Area under the plasma concentration; Cmax = Maximum plasma concetration; Tmax = Time to Cmax.

Programming note: please use AUCtau to report match with tables

# Listing 16.2.6.1 ANC/ALC Sample Collection Safety Population

| Subject | | Capsule<br>Strength | Dose<br>Level | | Threshold Adjusted | | | Hours from Previous | Result | _ |
|---|---|---|---|---|---|---|---|---|---|---|
| _Number | Visit | (mg) | (mg) | Test | AUC (cell.hr/uL) [1] | Time Point | Collection Date/Time | Sample | (cell/uL) [2] | Comments |
| | Week 5 | 25 | 100 | ALC | | Time 0 | DDMMMYYYY/ HH:MM | X.XXXX | XX | |
| | | | | | | 30 Minutes | DDMMMYYYY/ HH:MM | X.XXXX | XX | |
| | | | | | | 60 Minutes | DDMMMYYYY/ HH:MM | X.XXXX | XX | |
| | | | | | | 90 Minutes | DDMMMYYYY/ HH:MM | X.XXXX | XX | |
| | | | | | | 2 Hours | DDMMMYYYY/ HH:MM | X.XXXX | XXX | |
| | | | | | | 3 Hours | DDMMMYYYY/ HH:MM | X.XXXX | XXX | |
| | | | | | | 4 Hours | DDMMMYYYY/ HH:MM | X.XXXX | XXX | |
| | | | | | | 8 Hours | DDMMMYYYY/ HH:MM | X.XXXX | XXX | |
| | | | | | | 12 Hours | DDMMMYYYY/ HH:MM | X.XXXX | XXX | |
| | | | | | | 16 Hours | DDMMMYYYY/ HH:MM | X.XXXX | XXX | |
| | | | | | | 24 Hours | DDMMMYYYY/ HH:MM | X.XXXX | XXX | |
| | | | | | | | | | (BOCF) | |
| | Week<br>13 | 25 | 100 | ALC | | Time 0 | DDMMMYYYY/ HH:MM | X.XXXX | XX | |
| | 10 | | | | | 30 Minutes | DDMMMYYYY/ HH:MM | X.XXXX | XX | |
| | | | | | | 60 Minutes | DDMMMYYYY/ HH:MM | X.XXXX | XX | |
| | | | | | | 90 Minutes | DDMMMYYYY/ HH:MM | X.XXXX | XX | |
| | | | | | | 2 Hours | DDMMMYYYY/ HH:MM | X.XXXX | XXX | |

Abbreviations: AUC = Threshold adjusted area under the plasma concentration curve, BOCF = baseline observation carried forward.

[2] The imputation of BOCF is used for missing 24 hour assessment. Imputation is not used for intermediate missing assessments. Repeat assessments are not used in AUC calculation. Patients and took the Week 5 dose at home instead of the clinic resulting in the site not getting dense PK samples for the first few hours. Therefore, samples were taken the next day and the timepoints that were missed the day before were replaced with these samples. Patient assessments on 21 and 22 February 2018 were analyzed and presented as Week 21 assessments. For patient the assessment on 20FEB2018 at 9:25 was used as time 0.

<sup>[1]</sup> Threshold adjusted AUC is calculated using the trapezoidal method with area above threshold being positive, and area below threshold negative. The threshold is defined as 600/uL for ANC and as 1000/uL for ALC.

# Listing 16.2.6.2.1 Threshold Adjusted AUC values for ANC Safety Population

| ubject Number | Visit | Capsule<br>Strength (mg) | Dose<br>Level (mg) | Threshold Adjusted AUC (cell.hr/uL) [1] |
|---|---|---|---|---|
| | Week 5 | 25 | 50 | XXXX.XXXX |
| | Week 13 | 25 | 100 | |
| | Week 21 | 25 | 200 | |
| | Week 5 | 100 | | |
| | Week 13 | 100 | | |
| | Week 21 | 100 | | |
| | Week 5 | | | |
| | Week 13 | | | |
| | Week 21 | | | |

Abbreviation: AUC = Threshold adjusted area under the plasma concentration curve.

<sup>\*</sup>Value obtained during infection and considered to be confounded, value has not been used in the analysis.

<sup>\*\*</sup>Patient had normal value at Screening, therefore values have not been used in the analysis.

[1] Threshold adjusted AUC is calculated using the trapezoidal method with area above threshold being positive, and area below threshold negative. The threshold is defined as 600/uL for ANC.

### Listing 16.2.6.2.2 Threshold Adjusted AUC values for ALC Safety Population

(Same shell as Listing 16.2.6.2.1)

### Footnote:

Abbreviation: AUC = Threshold adjusted area under the plasma concentration curve. \*Value obtained during infection and considered to be confounded, value has not been used in the analysis.

<sup>\*\*</sup>Value was normal at Screening, therefore values have not been used in the analysis.

<sup>[1]</sup> Threshold adjusted AUC is calculated using the trapezoidal method with area above threshold being positive, and area below threshold negative. The threshold is defined as 1000/uL for ALC.

# Listing 16.2.6.2.3 Time Above Threshold by Dose Level - Assessment of ANC/ALC/AMC Safety Population

| Subject Number | Test | Dose Level (mg) | Time above Threshold (Hours) [1] |
|----------------|------|-----------------|----------------------------------|
| | ALC | 50 | XX.XX |
| | | 100 | XX.XX |
| | | 150 | XX.XX |
| | | 300 | XX.XX |
| | | 400 | XX.XX |
| | | 50/100/150 | XX.XX |
| | | 300/400 | XX.XX |
| | AMC | 50 | xx.xx |
| | | 100 | XX.XX |
| | | 150 | XX.XX |
| | | 300 | XX.XX |
| | | 400 | XX.XX |
| | | 50/100/150 | XX.XX |
| | | 300/400 | XX.XX |
| | ANC | 50 | XX.XX |
| | | 100 | XX.XX |
| | | 150 | XX.XX |
| | | 300 | XX.XX |
| | | 400 | XX.XX |
| | | 50/100/150 | XX.XX |
| | | 300/400 | XX.XX |
| | ALC | 50 | XX.XX |
| | | 100 | XX.XX |
| | | 150 | XX.XX |
| | | 300 | XX.XX |
| | | 400 | XX.XX |
| | | 50/100/150 | XX.XX |
| | | 300/400 | XX.XX |

| Subject Number | Test | Dose Level (mg) | Time above Threshold (Hours) [1] |
|----------------|------|-----------------|----------------------------------|

Note: If time above threshold was >24 hours, it was rounded off to 24.

<sup>\*</sup>Value obtained during infection and considered to be confounded, value has not been used in the analysis.

<sup>\*\*</sup>Value was normal at Screening, therefore values have not been used in the analysis.

<sup>[1]</sup> The threshold is defined as 500/uL for ANC, as 1000/uL for ALC, as 190/uL for females aged 12 to 18, 180/uL for males aged 12 to 18, 250/uL for females aged >=18 and 290/Ul for males aged >=18 for AMC.

## Listing 16.2.6.2.4 Time Above Threshold - Assessment of ANC/ALC/AMC with Time Crossed Safety Population

| Subject<br>Number | Visit | Capsule<br>Strength<br>(mg) | Dose<br>Level<br>(mg) | Test | Time Point | Collection Date/Time | Result<br>(cell/uL) | Comments | Time<br>Crossed | Time<br>above<br>Threshold<br>(Hours)<br>[1] |
|---|---|---|---|---|---|---|---|---|---|---|
| | Week 5 | 25 | 50 | ALC | Time 0 | DDMMMYYYY/ HH:MM | XXXX | | HH:MM | 0 |
| | 7.55.1.5 | | | 0 | 30 Minutes | DDMMMYYYY/ HH:MM | XXXX | | HH:MM | XX.XX |
| | | | | | 60 Minutes | DDMMMYYYY/ HH:MM | XXXX | | HH:MM | XX.XX |
| | | | | | 90 Minutes | DDMMMYYYY/ HH:MM | xxxx | | HH:MM | XX.XX |
| | | | | | 2 Hours | DDMMMYYYY/ HH:MM | XXXX | | HH:MM | XX.XX |
| | | | | | 3 Hours | DDMMMYYYY/ HH:MM | XXXX | | HH:MM | XX.XX |
| | | | | | 4 Hours | DDMMMYYYY/ HH:MM | XXXX | | HH:MM | XX.XX |
| | | | | | 8 Hours | DDMMMYYYY/ HH:MM | XXXX | | HH:MM | XX.XX |
| | | | | | 12 Hours | DDMMMYYYY/ HH:MM | XXXX | | HH:MM | XX.XX |
| | | | | | 16 Hours | DDMMMYYYY/ HH:MM | XXXX | | HH:MM | XX.XX |
| | | | | | 24 Hours | DDMMMYYYY/ HH:MM | XXXX | SNS: SAMPLE NOT SUBMITTED | | XX.XX |
| | | | | AMC | Time 0 | DDMMMYYYY/ HH:MM | XXXX | | HH:MM | 0 |
| | | | | ANC | | | | | | |

Abbreviations: BOCF = baseline observation carried forward.

Note: The imputation of BOCF is used for missing 24 hour assessment. Imputation is not used for intermediate missing assessments. Repeat assessments are not used in AUC calculation. Patients and and took the Week 5 dose at home instead of the clinic resulting in the site not getting dense PK samples for the first few hours. Therefore, samples were taken the next day and the timepoints that were missed the day before were replaced with these samples. The time above threshold values are calculated based on the separate days. Patient assessments on 21 and 22 February 2018 were analyzed and presented as Week 21

assessments. For patient the assessment on 20FEB2018 at 9:25 was used as time 0. Time crossed contains the time at which the AUC value crossed the threshold in either direction. \*Value obtained during infection and considered to be confounded, value has not been used in the analysis

[1] The threshold is defined as 500/uL for ANC, as 1000/uL for ALC, as 190/uL for females aged 12 to 18, 180/uL for males aged 12 to 18, 250/uL for females aged >=18 and 290/uL for males aged >=18 for AMC.
# Listing 16.2.7.1 Treatment Emergent Adverse Events Safety Population

| | Capsule | Dose | System Organ Class/ | | | | Other | |
|---|---|---|---|---|---|---|---|---|
| Subject | strength | Level | Preferred Term/ | Start Date (Day) / | Severity [2]/ | Outcome/ | Action | |
| Number | (mg) | (mg) | Verbatim Term | End Date (Day) [1] | Relationship | Action Taken | Taken | Serious? |
| | 25 | 100 | XXXXXXXXXXXX/<br>XXXXXXXXXX/<br>XXXXXXXXXXXX | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | Grade X/<br>Unrelated | RECOVERED/RESOLVED/<br>DOSE NOT CHANGED | | No |
| | 25 | 100 | XXXXXXXXXXXX/<br>XXXXXXXXXXX/<br>XXXXXXXXXXX | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | Grade X/<br>Unrelated | RECOVERED/RESOLVED/<br>DOSE NOT CHANGED | | No |
| | 100 | 200 | XXXXXXXXXXXX/<br>XXXXXXXXXX/<br>XXXXXXXXXXXX | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | Grade X/<br>Unrelated | RECOVERED/RESOLVED/<br>DOSE NOT CHANGED | | No |
| | 100 | 300 | XXXXXXXXXXXXX/<br>XXXXXXXXXXX/<br>XXXXXXXXXX | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | Grade X/<br>Unrelated | RECOVERED/RESOLVED/<br>DOSE NOT CHANGED | | No |
| | ••• | | | | | | | |

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

Programming Note: Sort Adverse Events by Patient, Start Date, System Organ Class and Preferred Term

<sup>[2]</sup> The severity is assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (v4.03).

## Listing 16.2.7.2 Adverse Events that occur during Screening and ended before Exposure to study Drug Safety Population

| Subject<br>Number | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start date(Day) /<br>End Date(Day) [1] | Severity[2] | Outcome/<br>Action Taken | Other Action Taken | Serious?/<br>Reason for SAE |
|---|---|---|---|---|---|---|
| | | DDMMMYYYY(XX)/<br>DDMMMYYYY(XX) | Grade 4 | | | |

Abbreviation: SAE = Serious adverse event.

Programming Note: Sort Adverse Events by Patient, Start Date, System Organ Class and Preferred Term

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

<sup>[2]</sup> The severity is assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (v4.03).

## Listing 16.2.7.3 Infections Reported as Adverse Events Safety Population

| Subject<br>Number | Capsule<br>Strength<br>(mg) | Dose Level<br>(mg) | AE# | Infection | Infection<br>cause | Culture<br>identified<br>organisms | Was an antibiotic used to treat the infection? | Was G-CSF<br>used to treat<br>the<br>infection? | Was Ig used to treat the infection? | Area of<br>Infection | Did the infection require a visit to a doctor's office? |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | 100 | 100 | | | | | | | | | |
| | | 100 | | | | | | | | | |
| | 25 | 200 | | | | | | | | | |
| | | 300 | | | | | | | | | |
| | | 100 | | | | | | | | | |
| | | 100 | | | | | | | | | |
| | | 100 | | | | | | | | | |
| | | 200 | | | | | | | | | |
| | | 200 | | | | | | | | | |
| | | 200 | | | | | | | | | |
| | | 300 | | | | | | | | | |
| | | 400 | | | | | | | | | |

Abbreviations: AE = Adverse event; ER = Emergency Room.

**Programming Note:** Sort Adverse Events by Patient, Start Date, System Organ Class and Preferred Term Only include infections where SOC = Infections and infestations

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

| | | | | Infections Repo | ting 16.2.7.3<br>orted as Adve<br>ety Population | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | AE# | Number of<br>doctor's office<br>visits due to<br>infection | Did the infection require hospital admission? | Number of<br>days in<br>hospital due<br>to infection | Did the infection require a visit to the ER? | Did the infection require admission to an intensive care unit? | Number of<br>Days of<br>work/school<br>missed | Were there<br>fevers<br>associated with<br>the infection? (if<br>Y, Peak Fever<br>Temperature (C) | Fever Start Date(Day)/<br>End Date(Day) [1] |

DDMMMYYYY(XX)/ DDMMMYYYY(XX)

Abbreviation: ER = Emergency Room.

[1] Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

**Programming Note:** Sort Adverse Events by Patient, Start Date, System Organ Class and Preferred Term Only include infections where SOC = Infections and infestations

## Listing 16.2.7.4 Deaths All Enrolled Patients

| Subject Number | Capsule Strength (mg) | Dose Level (mg) | Date of<br>Death (Day) [1] |
|---|---|---|---|
| | 25 | 100 | |
| | 100 | 300 | |
| | | 200 | |

<sup>[1]</sup> Day is calculated as (assessment date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (assessment date - date of administration of first study drug) if prior to the administration of first study drug.

## Listing 16.2.7.5 Treatment Limiting Toxicities Safety Population

| Subject<br>Number | Capsule<br>Strength<br>(mg) | Dose<br>Level (mg) | Gender | Age | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date(Day)/<br>End Date(Day) [1] | Severity [2]/<br>Relationship [3] | Outcome/<br>Action Taken |
|---|---|---|---|---|---|---|---|---|
| | 25 | 100 | М | 56 | | DDMMMYYYY(XX)/<br>DDMMMYYYY(XX) | | |
| | | 100 | F | | | | | |
| | | 200 | | | | | | |

Note: A TLT event for X4P-001 is defined as an AE that meets both of the following criteria:

- 1. Is assessed by the Investigator as possibly or probably related to X4P-001.
- 2. Represents one of the following events (grading as defined by the NCI CTCAE, v4.03 or higher):
- Is a Grade 3 or Grade 4 clinical event, except grade 3 nausea, vomiting, or diarrhea lasting <48 hrs in patients who have received suboptimal medical management.
- Is a confirmed Grade 3 or Grade 4 laboratory event with the following exceptions: Grade 3 electrolyte abnormalities that persist <72 hrs and do not require hospitalization. Grade 3 AST/ALT increases that persist <5 days and with total bilirubin ≤1.5x ULN.
- Is one of the following, which are designated as critical TLT events: AST/ALT increased >3x ULN (Grade 2) with total bilirubin increased >2x ULN in the absence of cholestasis. Retinopathy confirmed treatment-emergent retinopathy. Platelets <50,000/mm3 (Grade 3) with bleeding or <25,000/mm3 (Grade 4).
- [1] Day is calculated as (exam date date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date date of administration of first study drug) if prior to the administration of first study drug.
- [2] Severity is assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (v4.03).
- [3] Related = definitely related, probably related and possibly related; Unrelated = Unlikely related, not related

Programming Note: Sort Adverse Events by System Organ Class and Preferred Term; Footne the criteria for identifying the TLT

## Listing 16.2.7.6 Infections in Subjects Treated on 300mg or 400 mg Dose by Time Period Safety Population

| Subject Number | Time Period | Number of Infections |
|---|---|---|
| | Pre-Study (12 months prior to first dose) | XX |
| | 0-6 Months | xx |
| | 6-12 Months | xx |

Notes: Infections are identified as follows: for Prior 12 months, events are identified from the Medical History CRF under History of WHIM infections. While on study, infections are identified as all events with a MedDRA System Organ Class of "Infections and infestations".. The reporting period starts on the 300 mg dose date. Only events with start date occurring within start and end dates of 300/400 mg dose for each patient are included. Time period assignment is based on the start date of the event.

Patient was re-enrolled into the study on DDMMMYYYY. Patient was re-enrolled into the study on DDMMMYYYY.

Programming Note: Complete table until maximum duration in 6 month intervals; For the two patients re-enrolled, we need add "drop out period", "6 Months after re-enrollment", ....

present all data including data after re-enrollment for the 2 re-enrolled patients

### Listing 16.2.7.7 Infections by Dose Level Safety Population

| Subject Number | Dose Level | Number of Infections | Yearly Rate |
|----------------|---------------|----------------------|-------------|
| | 50/400/450 | | |
| | 50/100/150 mg | XX | XX |
| | 200 mg | XX | XX |
| | 300 mg | XX | XX |
| | 300 mg | XX | XX |
| | 400 mg | XX | XX |
| | 300/400 mg | XX | XX |
| | · · | | |
| | ••• | | |

Notes: Infections are identified as follows: for Prior 12 months, events are identified from the Medical History CRF. While on study, infections are identified as all events with a MedDRA System Organ Class of "Infections and infestations". Events at dose level are assigned based on the start date of the event occurring within start and end dates of that dose. Rate is defined as number of infection events in a given dose level / duration of exposure on a dose level in years.

Patient was re-enrolled into the study on DDMMMYYYY.

Patient was re-enrolled into the study on DDMMMYYYY.

Programming Note: present all data including data after re-enrollment for the 2 re-enrolled patients

## Listing 16.2.7.8 Infections by Subject Safety Population

| | | | | | | | | | Infection Details [1] | |
|---|---|---|---|---|---|---|---|---|---|---|
| ıbject | Date of | Dose | Treatment | Treatment | Duration<br>(Days) | Number<br>of | AE Start | AE End | Preferred Term/ | Infection |
| mber | Consent | \ 0/ | Start Date | End Date | at Dose Level | Infections | | Date | AE Term | Severity |
| | DDMMMYYY | YPrior 12<br>months | | | | 5 | DDMMMYYYY | ´// | /Cellulitis | Grade X |
| | | | | | | | DDMMMYYYY | DDMMMYYYY | /Otitis media | Grade X |
| | | | | | | | DDMMMYYYY | DDMMMYYYY | /Pneumonia | Grade X |
| | | | | | | | DDMMMYYYY | DDMMMYYYY | /Skin abscesses | Grade X |
| | | | | | | | DDMMMYYYY | DDMMMYYYY | /URI (sinusitis, otitis, pharyngitis) | Grade X |
| | | 50 | DDMMMYYYY | DDMMMYYY | Y 37 | 4 | | | Ear infection/ear inflammation causing discomfort | Grade X |
| | | | | | | | DDMMMYYYY | DDMMMYYYY | Sinusitis/sinus inflammation causing discomfort | Grade X |
| | | | | | | | DDMMMYYYY | DDMMMYYYY | Ear infection/Ear infection | Grade X |
| | | | | | | | DDMMMYYYY | DDMMMYYYY | Sinusitis/sinus infection | Grade X |
| | | 100 | DDMMMYYYY | DDMMMYYY | Y 52 | 0 | | | | |
| | | 150 | DDMMMYYYY | DDMMMYYY | Y145 | 0 | | | | |
| | | 300 | DDMMMYYYY | DDMMMYYY | Y126 | 2 | DDMMMYYYY | DDMMMYYYY | Sinusitis/Sinus infection | Grade X |
| | | | | | | | DDMMMYYYY | DDMMMYYYY | Sinusitis/Sinusitis | Grade X |
| | | 400 | DDMMMYYYY | DDMMMYYY | Y513 | 4 | DDMMMYYYY | DDMMMYYYY | Pharyngitis/Pharyngitis | Grade X |
| | | | | | | | | | | Grade X |
| | | | | | | | DDMMMYYYY | DDMMMYYYY | Sinusitis/Sinusitis | Grade X |
| | | | | | | | DDMMMYYYY | • | Cellulitis/Cellulitis (left forearm) | Grade X |
| | | 400 (after re-<br>enrollment) | DDMMMYYYY | DDMMMYYY' | YXX | XX | | | xxxxxxxxxxx | O.a.o.z. |
| | DDMMMYYY | | | | | 5 | DDMMMYYYY | DDMMMYYYY | /Abscess, left leg/thigh | Grade X |
| | | months | | | | | DDMMMYYYY | DDMMMYYYY | /Cellulitis at skin biopsy site - left side of neck | Grade X |
| | | | | | | | DDMMMYYYY | DDMMMYYYY | /Cellulitis at skin biopsy site - right arm | Grade X |
| | | | | | | | | | /Cellulitis, left external ear | Grade X |
| | | | | | | | | | /Cellulitis, left forearm | Grade X |

| | | | | | | | | | Infection Details [1] | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Date of<br>Consent | Dose<br>Level (mg) | Treatment<br>Start Date | Treatment<br>End Date | Duration<br>(Days)<br>at Dose Level | Number<br>of<br>Infections | AE Start | AE End<br>Date | Preferred Term/<br>AE Term | Infection<br>Severity |

Abbreviation: AE = Adverse event.

[1] Infections identified as follows: for Prior 12 months, events are identified from the Medical History CRF under History of WHIM infections. While on study, infections are identified as all events with a MedDRA System Organ Class of 'Infections and infestations'; dose level is assigned based on the start date of the event occurring within start and end dates of that dose for each subject.

Patient was re-enrolled into the study on DDMMMYYYY. Patient was re-enrolled into the study on DDMMMYYYY.

Programming note: Present all dose levels with start and end dates available. If patient didn't have any infection events, then the number of infections is 0.

## Listing 16.2.8.1 Clinical Laboratory Data: Serum Chemistry Safety Population

Test Name: XXXXX (units)

| | | Dose | | | | | Change | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject | | Level | Date/Time of | Standard | Reference | Abnormal?/ | from | Calculated | Comments/ |
| Number | Visit | (mg) | Assessment (Day) [1] | Results | Range | High/Low [2] | Baseline [3] | CTC Grade | Reason not Done |
| | Day 1 | 100 | DDMMMYYYY/ | XX | XX - XX | No | | | |
| | • | | HH:MM (XX) | | | | | | |
| | Week 5 | 100 | , | | | | | | |
| | Week 13 | 200 | | | | | | | |
| | Week 21 | 300 | | | | | | | |
| | Day 1 | 100 | | | | | | | |
| | Week 5 | 100 | | | | | | | |
| | Week 13 | 100 | | | | | | | |
| | Week 21 | 200 | | | | | | | |
| | Day 1 | 200 | | | | | | | |
| | Week 5 | 200 | | | | | | | |
| | Week 13 | 300 | | | | | | | |
| | Week 21 | 400 | | | | | | | |

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

<sup>[2]</sup> L = Low, H = High.

<sup>[3]</sup> Change from baseline = value - Baseline value. Baseline is defined as the last assessment prior to the first study drug.

Listing 16.2.8.2 Clinical Laboratory Data: Hematology Safety Population

(Same shell as Listing 16.2.8.1)

Listing 16.2.8.3
Serology and Other Laboratory Test Results
Safety Population

(Same shell as Listing 16.2.8.1)

## Listing 16.2.8.4 Serum Ig and Specific Antibody Laboratory Test Results Safety Population

| Subject<br>Number | Visit | Capsule<br>strength<br>(mg) | Dose<br>Level<br>(mg) | Date/Time Collected<br>(Day) [1] | Test Name | Standard Results | Reference<br>Range | CFB<br>[2] | Fold-<br>Change | Flag<br>[3] |
|---|---|---|---|---|---|---|---|---|---|---|
| | Day 1 | 25 | 100 | DDMMMYYYY/HH:MM (XX) | Haemophilus Influenzae B Polysaccharide (mg/L) Immunoglobulin A (g/L) Immunoglobulin G (g/L) Immunoglobulin G Subclass 1 (g/L) Immunoglobulin G Subclass 2 (g/L) Immunoglobulin G Subclass 3 (g/L) Immunoglobulin G Subclass 4 (g/L) Immunoglobulin M (g/L) Rubeola IgG (Measles) Rubella IgG Antibody Index (INDEX) Tetanus Toxoid (IU/L) | Positive/Negative | - | | • | |
| | Week X | 25 | 200 | DDMMMYYYY/HH:MM (XX) | | | | | | |

Abbreviation: CFB = Change from Baseline.

Fold-Change = Value/Baseline

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

<sup>[2]</sup> Change from Baseline - value - baseline value. Baseline is defined as the last assessment prior to the first study drug.

<sup>[3]</sup> L = Low, H = High, N = Normal.

Listing 16.2.8.5 Pregnancy Test Safety Population

| Subject<br>Number | Visit | Dose Level<br>(mg) | Was Pregnancy Test Performed? | Date Performed (Day)<br>[1] | Time of<br>Assessment | Specimen Type | Result of Pregnancy<br>Test |
|---|---|---|---|---|---|---|---|
| | Screening | 100 | Yes | DDMMMYYYY(XX) | HH:MM | Serum<br>Urine | <5 (IU/L)/Negative<br>Negative |
| | Week X/ | 100 | Yes | DDMMMYYYY(XX) | HH:MM | Serum<br>Urine | <5 (IU/L)/Negative<br>Negative |
| | Screening | 100 | Yes | DDMMMYYYY(XX) | НН:ММ | Serum<br>Urine | <5 (IU/L)/Negative<br>Negative |
| | Screening | 200 | Yes | DDMMMYYYY(XX) | НН:ММ | Serum<br>Urine | <5 (IU/L)/Negative<br>Negative |

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

### Listing 16.2.8.6 Coagulation Laboratory Test Results Safety Population

Test Name: XXXXXXX (units)

| | | Dose | | | | | Change from | Fold- |
|---|---|---|---|---|---|---|---|---|
| Subject | | Level | Date/Time of | | Reference | Abnormal? | Baseline | Change |
| Number | Visit | (mg) | Assessment (Day) [1] | Test Result | Range | High/Low [2] | [3] | [4] |
| | Week 9 | XXX | DDMMMYYYY/HH:MM (XX) | XX.X | XX - XX | Yes / H | | |
| | Week 13 | XXX | , | XX.X | XX - XX | No | | |
| | Week 17 | XXX | | XX.X | XX - XX | Yes / H | | |
| | Week 21 | XXX | | XX.X | XX - XX | No | | |
| | Week 9 | XXX | | XX.X | XX - XX | No | | |
| | Week 13 | XXX | | XX.X | XX - XX | No | | |
| | Week 17 | XXX | | XX.X | XX - XX | No | | |
| | Week 21 | XXX | | XX.X | XX - XX | No | | |
| | Screening | | | | | | | |
| | Day 1 | | | XX.X | XX - XX | No | | |
| | Week 2 | XXX | | XX.X | | | | |
| | Week 3 | XXX | | XX.X | XX - XX | No | XX.X | XX.X |
| | Week 4 | XXX | | XX.X | XX - XX | No | XX.X | XX.X |
| | Week 5 | XXX | | XX.X | XX - XX | No | XX.X | XX.X |

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

<sup>[2]</sup> L = Low, H = High.

<sup>[3]</sup> Change from Baseline = value - Baseline value. Baseline is defined as the last assessment prior to the first study drug.

<sup>[4]</sup> Fold-Change = Value/Baseline.

## Listing 16.2.8.7 Urinalysis Laboratory Test Results Safety Population

Test Name: XXXXXX

| Subject | | Dose Leve | el Date/Time of | • | Reference | Abnormal? | Change from | Fold-Change |
|---|---|---|---|---|---|---|---|---|
| Number | Visit | (mg) | Assessment (Day) [1] | Test Result | Range | High/Low [2] | Baseline [3] | [4] |
| | Screening | | DDMMMYYYY/HH:MM (XX) | xxxxxx | | No | | |
| | Day 1 | | DDMMMYYYY/HH:MM (XX) | XXXXXX | | No | | |
| | Week 13 | XXX | DDMMMYYYY/HH:MM (XX) | XXXXXX | | No | | |
| | Week 21 | XXX | DDMMMYYYY/HH:MM (XX) | XXXXXX | | No | | |
| | Screening | | | xxxxxx | | No | | |
| | Day 1 | | | XXXXXX | | No | | |
| | Week 13 | XXX | | XXXXXX | | No | | |
| | Week 21 | XXX | | XXXXXX | | No | | |
| | Screening | | | XXXXXX | | No | | |
| | Day 1 | | | XXXXXX | | No | | |
| | Week 5 | XXX | | XXXXXX | | No | | |
| | Screening | | | xxxxxx | | No | | |
| | Day 1 | | | XXXXXX | | No | | |
| | Week 5 | XXX | | XXXXXX | | No | | |

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

<sup>[2]</sup> L = Low, H = High.

<sup>[3]</sup> Change from Baseline = value - Baseline value. Baseline is defined as the last assessment prior to the first study drug. [4] Fold-Change = Value/Baseline.

### Listing 16.2.8.8 CytometryTest Results Safety Population

Test Name: XXXXXX

| Subject | | Dose Level | Date/Time of | | | Change from |
|---|---|---|---|---|---|---|
| Number | Visit | (mg) | Assessment (Day) [1] | Replicate | Test Result | Baseline [2] |
| | Screening | | DDMMMYYYY/HH:MM (XX) | А | xxxxxx | XXXXXX |
| | 3 | | DDMMMYYYY/HH:MM (XX) | В | XXXXXX | XXXXXX |
| | | | DDMMMYYYY/HH:MM (XX) | С | XXXXXX | XXXXXX |
| | Day 1 | | DDMMMYYYY/HH:MM (XX) | X | XXXXXX | XXXXXX |
| | Week 13 | XXX | DDMMMYYYY/HH:MM (XX) | X | XXXXXX | XXXXXX |
| | Week 21 | XXX | DDMMMYYYY/HH:MM (XX) | X | XXXXXX | XXXXXX |
| | Screening | | | X | xxxxxx | XXXXXX |
| | Day 1 | | | X | XXXXXX | XXXXXX |
| | Week 13 | XXX | | X | XXXXXX | XXXXXX |
| | Week 21 | XXX | | X | XXXXXX | XXXXXX |
| | Screening | | | Χ | xxxxxx | XXXXXX |
| | Day 1 | | | X | XXXXXX | XXXXXX |
| | Week 5 | XXX | | X | XXXXXX | XXXXXX |
| | Screening | | | Χ | XXXXXX | XXXXXX |
| | Day 1 | | | X | XXXXXX | XXXXXX |
| | Week 5 | XXX | | X | XXXXXX | XXXXXX |

Note: Each sample was run 3 times producing triplicate results A, B, C for each laboratory test.

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

<sup>[2]</sup> Change from Baseline - value - Baseline value. Baseline is defined as the last assessment prior to the first study drug.

### Listing 16.2.9.1 Prior or Concomitant Medications Safety Population

| Subject<br>Number | Prior,<br>Concomitant<br>or Both? | ATC Class (Level 5)/<br>PT (ATC Level 4)/<br>VT | Start Date (Day)/<br>End Date (Day) [1] | Dose<br>(Unit) | Route | Frequency | Reason for Use |
|---|---|---|---|---|---|---|---|
| | Both | XXXXXXXXXXXXX/<br>XXXXXXXXXXXXX/<br>XXXXXXXXX | Ongoing | XX (mg) | ORAL | OTHER<br>(QD, PRN) | Seasonal allergies |
| | Concomitant | XXXXXXXXXXXXX/<br>XXXXXXXXXXXXXX/<br>XXXXXXXX | DDMMMYYYY (XX)/<br>DDMMMYYYY (XX) | | ORAL | QD | Seasonal allergies |
| | Prior | XXXXXXXXXXXXX/<br>XXXXXXXXXXXXX/<br>XXXXXXXXX | DDMMMYYYY (XX)/<br>DDMMMYYYY (XX) | | ORAL | QD | body aches and pains |

Abbreviations: ATC = Anatomic Therapeutic Chemical; PT = Preferred Term; VT = Verbatim Term.

Concomitant medication is any medication taken or ongoing on or after the first dose of the study medication.

**Programming Note:** Sort Concomitant Medications by ATC Class and Preferred Term

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

Prior medication is any medication that is started or ended prior to the first dose of the study medication.

# Listing 16.2.9.2 Vital Signs Measurements Safety Population

| Subject | | Capsule<br>strength | Dose<br>Level | Date of | Body<br>Temp | Pulse<br>Rate | (mi | Pressure<br>mHg) | Height | Weight | ВМІ |
|---|---|---|---|---|---|---|---|---|---|---|---|
| number | Visit | (mg) | (mg) | Assessment(Day)[1] | (C) | (bpm) | Systolic | Diastolic | (cm) | (kg) | (kg/m2) [2] |
| | Day 1 | 25 | 100 | DDMMMYYYY (XX) | XX.X | XX | XX | XX | XX | XX | XX |
| | Week 5 | | 100 | , , | XX.X | XX | XX | XX | XX | XX | XX |
| | Week 13 | | 200 | | XX.X | XX | XX | XX | XX | XX | XX |
| | Week 21 | | 300 | | XX.X | XX | XX | XX | XX | XX | XX |

Abbreviation: BMI = Body Mass Index.
[1] Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.
[2] BMI = Weight/(Height)<sup>2</sup>x10<sup>4</sup>.

## Listing 16.2.9.3 12-Lead Electrocardiograms Safety Population

| Subject Number | Visit | Date of Assessment (Day) [1] | Assessment | Investigator Interpretation/Results |
|---|---|---|---|---|
| | Day 1 | DDMMMYYYY (XX) | Summary (Mean) Heart Rate<br>Summary (Mean) PR Duration<br>Summary (Mean) QRS Duration<br>Summary (Mean) QT Duration<br>QTc Interval<br>Interpretation<br>QTc Method | XX beats/min XXX ms XXX ms XXX ms XXX ms XXX ms N Bazett's formula |
| | Week 5 | DDMMMYYYY (XX) | <br> | |

Abbreviations: CS = Clinically significant; NCS = Not clinically significant; N = Normal.

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

## Listing 16.2.9.4 Physical Examinations Safety Population

| Subject Number | Visit | Capsule<br>Strength<br>(mg) | Dose<br>Level<br>(mg) | Performed? | Date/Time of<br>Examination (Day) [1] | Body System | Result | Clinically<br>Significant? | Abnormal Findings |
|---|---|---|---|---|---|---|---|---|---|
| | Day 1 | 0.5 | 100 | | DDMMMYYYY (XX) | Cardiovascular | NORMAL | | |
| | Week 5<br>Week 13<br>Week 21 | 25 | 100<br>200<br>300 | | | Respiratory<br>Gastrointestinal<br>Neurological | ABNORMAL | Yes/No | |
| | Day 1<br>Week 5 | | 100 mg<br>100 mg | | | Musculoskeletal<br>HEENT | NOT DONE | | |
| | Week 13<br>Week 21 | | 100 mg<br>200 mg | | | Thyroid<br>Skin | | | |
| | Day 1<br>Week 5<br>Week 13<br>Week 21 | | 200 mg<br>200 mg<br>300 mg<br>400 mg | | | Extremities<br>Genitourinary<br>Other: XXXXXX | | | |

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

## Listing 16.2.9.5 Ophthalmologic Examination (Site Assessment) Safety Population

| | | | | | | Photos Collected During the Retinal Exam? | | | Centered On | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Visit | Capsule<br>Strength<br>(mg) | | Performed? | · • / | | Results | Optic<br>Nerve | Macula | Superior<br>Arcade | Inferior<br>Arcade | Temporal<br>Retina (2<br>photos) | Nasal<br>Retina |
| | Part A -<br>Screening | | | Yes | DDMMMYYYY/<br>HH:MM (XX) | Yes | Abnormal<br>- NCS | Bilateral | Bilateral | Bilateral | Bilateral | Bilateral | Bilateral |
| | Part A -<br>Week 13 | 25 | 100 | Yes | DDMMMYYYY/<br>HH:MM (XX) | Yes | Abnormal<br>- NCS | Bilateral | Bilateral | Bilateral | Bilateral | Bilateral | Bilateral |
| | Part A -<br>Week 25<br>EOT | 25 | 150 | Yes | DDMMMYYYY/<br>HH:MM (XX) | Yes | Abnormal<br>- NCS | Bilateral | Bilateral | Bilateral | Bilateral | Bilateral | Bilateral |
| | | | | No | | | | | | | | | |

Abbreviations: CS = Clinically significant; NCS = Not clinically significant.

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

## Listing 16.2.9.6 Ophthalmologic Examination (Central Readings) Safety Population

| Subject<br>Number | Visit | Date of examination (Day) [1] | Photographs<br>Reviewed? | Retinal Findings | Agree<br>with<br>Local<br>Results? | Disagreement<br>Description | Any<br>Photograph<br>Deficiencies? | Retinal<br>Photograph<br>Deficiencies | Other<br>Findings or<br>Concerns? | Non-<br>Retinal<br>Findings |
|---|---|---|---|---|---|---|---|---|---|---|
| | Day 1<br>Week 5 | DDMMYYYY<br>(XX) | Yes | Abnormal - new finding NCS | No | | No | | No | |
| | Week 13<br>Week 21 | | | | | | | | | |
| | Day 1<br>Week 5 | | | | | | | | | |
| | Week 13<br>Week 21 | | | | | | | | | |
| | Day 1<br>Week 5 | | | | | | | | | |
| | Week 13 | | | | | | | | | |
| | Week 21 | | | -£ 6:+ -+ | | | | | | |

<sup>[1]</sup> Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

Listing 16.2.9.7 Rescue Medications Safety Population

| Did subject receive rescue therapy for acute, severe bacterial infection while on study? | Medication<br>Record Number | Start date/Time (Day)/<br>End Date/Time (Day)[1] | Ongoing? | |
|---|---|---|---|---|
| Yes | | | | |
| | severe bacterial infection while on study? | severe bacterial infection while on study? Record Number | severe bacterial infection while on study? Record Number End Date/Time (Day)[1] | severe bacterial infection while on study? Record Number End Date/Time (Day)[1] Ongoing? |

[1] Day is calculated as (start/end date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (start/end date - date of administration of first study drug) if prior to the administration of first study drug.

Listing 16.2.9.8 SF-36 QOL Safety Population

| Subject<br>Number | Visit | Capsule<br>Strength<br>(mg) | Dose<br>Level<br>(mg) | Was the SF-36<br>QOL<br>Questionnaire<br>Completed? | Date of Questionnaire completion (Day) [1] | Physical<br>Functioning<br>(PF) Domain<br>Score | Role-Physical<br>(RP) Domain<br>Score | Bodily Pain<br>(BD) Domain<br>Score | General<br>Health (GH)<br>Domain Score | Vitality (VT)<br>Domain Score |
|---|---|---|---|---|---|---|---|---|---|---|
| | Day 1<br>Week 3<br>Week 5<br>Week 9<br>Week 13<br>Week 17<br>Week 21 | 25 | 50<br>50<br>100<br>100<br>150<br>150 | No<br>Yes<br>Yes<br>Yes<br>Yes<br>Yes<br>Yes | DDMMMYYYY (XX) | 90<br>90<br>95<br>90<br>90<br>90 | 75<br>81.25<br>75<br>93.75<br>100<br>100 | 74<br>74<br>62<br>84<br>84<br>84 | 25<br>30<br>35<br>35<br>30<br>30<br>45 | 43.75<br>37.5<br>37.5<br>37.5<br>50<br>62.5<br>68.75 |
| | EOT<br>Extension<br>Phase -<br>Residence<br>Visit 1<br>Post EOS | 100 | 300 | Yes | DDMMMYYYY (XX) | 100 | 100 | 84 | 30 | 62.5 |
| | Extension Phase - Residence Visit 1 | 100 | 300 | Yes | DDMMMYYYY (XX) | 100 | 100 | 100 | 37 | 62.5 |
| | Extension<br>Phase -<br>Residence<br>Visit 2 | 100 | 400 | Yes | DDMMMYYYY (XX) | 100 | 100 | 62 | 30 | 56.26 |

Abbreviation: QOL = Quality of Life.

<sup>[1]</sup> Day is calculated as (collection date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (collection date - date of administration of first study drug) if prior to the administration of first study drug.

Listing 16.2.9.8 SF-36 QOL Safety Population

| Subject<br>Number | Visit | Capsule<br>Strength<br>(mg) | Dose<br>Level<br>(mg) | Was the<br>SF-36 QOL<br>Questionnaire<br>Completed? | Date of<br>Questionnaire<br>completion (Day) [1] | Social<br>Functioning<br>(SF) Domain<br>Score | Role-<br>Emotional<br>(RE)<br>Domain<br>Score | Mental<br>Health (MH)<br>Domain<br>Score | Reported<br>Health<br>Transition<br>(HT) Item<br>Score | Physical<br>Component<br>Summary<br>(PSC)<br>Score | Mental<br>Component<br>Summary<br>(MCS)<br>Score |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day 1 | | | No | | | | | | | |
| | Week 3 | 25 | 50 | Yes | DDMMMYYYY (XX) | 90 | 75 | 74 | 25 | 43.75 | |
| | Week 5 | 25 | 50 | Yes | DDMMMYYYY (XX) | 90 | 81.25 | 74 | 30 | 37.5 | |
| | Week 9 | 25 | 100 | Yes | DDMMMYYYY (XX) | 95 | 75 | 62 | 35 | 37.5 | |
| | Week 13 | 25 | 100 | Yes | DDMMMYYYY (XX) | 90 | 93.75 | 84 | 35 | 37.5 | |
| | Week 17 | 25 | 150 | Yes | DDMMMYYYY (XX) | 90 | 100 | 84 | 30 | 50 | |
| | Week 21 | 25 | 150 | Yes | DDMMMYYYY (XX) | 90 | 100 | 84 | 30 | 62.5 | |
| | Week 25<br>EOT | 25 | 150 | Yes | DDMMMYYYY (XX) | 90 | 100 | 84 | 45 | 68.75 | |
| | Extension<br>Phase -<br>Residence<br>Visit 1<br>Post EOS | 100 | 300 | Yes | DDMMMYYYY (XX) | 100 | 100 | 84 | 30 | 62.5 | |
| | Extension<br>Phase -<br>Residence<br>Visit 1 | 100 | 300 | Yes | DDMMMYYYY (XX) | 100 | 100 | 100 | 37 | 62.5 | |
| | Extension<br>Phase -<br>Residence<br>Visit 2 | 100 | 400 | Yes | DDMMMYYYY (XX) | 100 | 100 | 62 | 30 | 56.26 | |

Abbreviation: QOL = Quality of Life.
[1] Day is calculated as (exam date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (exam date - date of administration of first study drug) if prior to the administration of first study drug.

## Listing 16.2.9.9.1 HPV Impact Profile (HIP) Questionnaire Safety Population

| Subject<br>Number | Visit | Capsule<br>Strength<br>(mg) | Dose<br>Level<br>(mg) | Collection Date<br>(Day) [1] | Does the<br>Subject<br>have<br>Genital<br>Warts? | HIP<br>Questi-<br>onnaire<br>Colle-<br>cted? | Question | Subject<br>Response | Subject<br>Response<br>Description |
|---|---|---|---|---|---|---|---|---|---|
| | xxxxxxxxx | xx | XXX | DDMMMYYYY (XX) | Yes | Yes | When I think about my recent gynecology exam or test results, I feel good about myself. | X | XXXXXX |
| | | | | | | | <ol> <li>When I think about my recent<br/>gynecology exam or test results, I feel<br/>anxious.</li> </ol> | Х | XXXXXX |
| | | | | | | | 3. I feel my recent gynecology test results were unexpected. | Х | XXXXXX |
| | | | | | | | When I think about my recent gynecology exam or test results, I feel in control of my health. | X | XXXXXX |
| | | | | | | | When I think about my recent<br>gynecology exam or test results, I feel<br>depressed. | X | XXXXXX |
| | | | | | | | After my recent gynecology exam or<br>test results, I feel I can concentrate as wel<br>as usual on everyday matters. | X | XXXXXX |
| | | | | | | | 7. When I think about my recent gynecology exam or test results, I feel something is seriously wrong with me. | X | XXXXXX |
| | | | | | | | 8. When I think about my recent gynecology exam or test results, I feel angry. | Х | XXXXXX |

<sup>[1]</sup> Day is calculated as (collection date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (collection date - date of administration of first study drug) if prior to the administration of first study drug.

## Listing 16.2.9.9.2 HPV Impact Profile (HIP) Questionnaire - Domain Scores Safety Population

| Subject<br>Number | Visit | Capsule<br>Strength<br>(mg) | Dose<br>Level<br>(mg) | Collection Date<br>(Day) [1] | Does the<br>Subject<br>have<br>Genital<br>Warts? | HIP<br>Questi-<br>onnaire<br>Colle-<br>cted? | Domain | Mean<br>Transformed<br>Score | Overall<br>Mean<br>d Transformed<br>Score |
|---|---|---|---|---|---|---|---|---|---|
| | XXXXXXXX | | | xxxxxx | Yes | Yes | Self Image Emotional Impact Control/Life Impact Worries and Concerns Partner and Transmission Sexual Impact Interactions with Doctors | XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX.X |
| | Part A - Day 1 | | | | Yes | No | | | |
| | Part A - Week 3 | xx | XXX | XXXXXX | Yes | Yes | Self Image Emotional Impact Control/Life Impact Worries and Concerns Partner and Transmission Sexual Impact Interactions with Doctors | XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX.X |

<sup>[1]</sup> Day is calculated as (collection date - date of administration of first study drug) + 1 if on or after the administration of first study drug. Day is calculated as (collection date - date of a dministration of first study drug) if prior to the administration of first study drug.